CLINICAL TRIAL: NCT00502593
Title: A Phase II, Randomized, Open, Controlled Study to Evaluate the Safety and Immunogenicity of Different Formulations of a Pandemic Influenza Vaccine Candidate (Split Virus Formulation Adjuvanted With AS03) Given Following a Two-administration Schedule (21 Days Apart) in Children Between 3 and 9 Years of Age.
Brief Title: Evaluate Safety & Immunogenicity of a Pandemic Influenza Vaccine (GSK1562902A) in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107066; 108498 (Other: GSK); 108500 (Other: GSK)
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2017-06

CONDITIONS: Influenza
Keywords: Influenza; Pandemic Influenza Vaccine (GSK1562902A)
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- GSK1562902A-A Lot 1 3-5Y Group (Experimental): Subjects aged 3-5 years received 2 doses of GSK1562902A vaccine, lot 1. These subjects were enrolled in the Phase A of this NCT00502593 study (or study 107066). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-A 3-5Y Group (Active Comparator): Subjects aged 3-5 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase A of this NCT00502593 study (or study 107066). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™
- GSK1562902A-A Lot 1 6-9Y Group (Experimental): Subjects aged 6-9 years received 2 doses of GSK1562902A vaccine, lot 1. These subjects were enrolled in the Phase A of this NCT00502593 study (or study 107066). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-A 6-9Y Group (Active Comparator): Subjects aged 6-9 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase A of this NCT00502593 study (or study 107066). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™
- GSK1562902A-B Lot 2 3-5Y Group (Experimental): Subjects aged 3-5 years received 2 doses of GSK1562902A vaccine, lot 2. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-B 3-5Y Group (Active Comparator): Subjects aged 3-5 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™
- GSK1562902A-B Lot 2 6-9Y Group (Experimental): Subjects aged 6-9 years received 2 doses of GSK1562902A vaccine, lot 2. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-B 6-9Y Group (Active Comparator): Subjects aged 6-9 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™
- GSK1562902A-C Lot 3 3-5Y Group (Experimental): Subjects aged 3-5 years received 2 doses of GSK1562902A vaccine, lot 3. These subjects were enrolled in the Phase C of this NCT00502593 study (or study 108500). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-C 3-5Y Group (Active Comparator): Subjects aged 3-5 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase C of this NCT00502593 study (or study 108500). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™
- GSK1562902A-C Lot 3 6-9Y Group (Experimental): Subjects aged 6-9 years received 2 doses of GSK1562902A vaccine, lot 3. These subjects were enrolled in the Phase C of this NCT00502593 study (or study 108500). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Pandemic Influenza Vaccine (GSK1562902A)
- Fluarix-C 6-9Y Group (Active Comparator): Subjects aged 6-9 years received 2 doses of Fluarix™ vaccine. These subjects were enrolled in the Phase C of this NCT00502593 study (or study 108500). The Fluarix™ vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Pandemic Influenza Vaccine (GSK1562902A) — 2 doses, intramuscular injection on Days 0 and 21, 3 different formulations are tested.
  Arms: GSK1562902A-A Lot 1 3-5Y Group; GSK1562902A-A Lot 1 6-9Y Group; GSK1562902A-B Lot 2 3-5Y Group; GSK1562902A-B Lot 2 6-9Y Group; GSK1562902A-C Lot 3 3-5Y Group; GSK1562902A-C Lot 3 6-9Y Group
Biological: Fluarix™ — 2 doses, intramuscular injection on Days 0 and 21.
  Arms: Fluarix-A 3-5Y Group; Fluarix-A 6-9Y Group; Fluarix-B 3-5Y Group; Fluarix-B 6-9Y Group; Fluarix-C 3-5Y Group; Fluarix-C 6-9Y Group

SUMMARY:
The present study is designed to evaluate in children (aged between 3 and 9 years) the immunogenicity and safety of different antigen doses of the candidate vaccine (GSK1562902A) administered following a two-administration schedule (21 days apart). Subjects in the control group will receive Fluarix. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This 107066 study is a participating study to the broader NCT00502593 study, which included 2 other studies, the 108498 and 108500 studies. The NCT00502593 study had a staggered design (subjects from each group being enrolled sequentially into 2 age strata, '6-9 years' 1st, and '3-5 years' next) and was run in 3 phases, phases A (Study 107066), B (Study 108498) and C (Study 108500). In each phase, the decision to vaccinate subjects aged 3-5 years and to administer a 2nd injection to subjects aged 6-9 years was made based on safety data collected on Days 0-6 after the 1st injection for the subjects aged 6-9 years. Decision to start Phase B was made on complete safety data including those collected on Day 28 of Phase A (7 days after the 2nd injection) for each age group. A similar approach was to be used to start Phase C. As safety data in Phase A did not raise any safety concerns, Phases B and C were run in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Children who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Children aged between and including 3 and 9 years of age at the time of first vaccination.
* Written informed consent obtained from the parent(s) or guardian of the subject.
* Healthy children as established by medical history and clinical examination before entering the study.
* Subjects who are likely to reside in the vicinity of the study center for the duration of the study.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the investigational vaccine within 30 days prior to the enrolment in this study, or planned use during the study period.
* Administration of licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 30 days after the second vaccination, with the exception of routine childhood inoculations which cannot be delayed, but which must not be administered on the same day as the investigational vaccine candidate.
* Administration of the interpandemic influenza vaccine 21 days prior to Day 0 or up to Day 51.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the enrolment in this study.
* Any chronic drug therapy to be continued during the study period, with the exception of inhalative treatment for seasonal allergies or asthma.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines used in this study.
* History of any neurological disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study or planned during the study.
* Any condition which, in the opinion of the investigator, renders the subject unfit for participation in the study

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2007-07-23; Primary Completion 2009-12-04 (Actual); Study Completion 2009-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Spain (5):
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, L'Eliana, Valencia
  - GSK Investigational Site, Paiporta, Valencia
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Diez-Domingo J, Baldo JM, Planelles-Catarino MV, Garces-Sanchez M, Ubeda I, Jubert-Rosich A, Mares J, Garcia-Corbeira P, Moris P, Teko M, Vanden Abeele C, Gillard P. Phase II, randomized, open, controlled study of AS03-adjuvanted H5N1 pre-pandemic influenza vaccine in children aged 3 to 9 years: follow-up of safety and immunogenicity persistence at 24 months post-vaccination. Influenza Other Respir Viruses. 2015 Mar;9(2):68-77. doi: 10.1111/irv.12295. Epub 2015 Feb 5. PMID 25652873
- [Derived] Diez-Domingo J, Garces-Sanchez M, Baldo JM, Planelles MV, Ubeda I, JuBert A, Mares J, Moris P, Garcia-Corbeira P, Drame M, Gillard P. Immunogenicity and Safety of H5N1 A/Vietnam/1194/2004 (Clade 1) AS03-adjuvanted prepandemic candidate influenza vaccines in children aged 3 to 9 years: a phase ii, randomized, open, controlled study. Pediatr Infect Dis J. 2010 Jun;29(6):e35-46. doi: 10.1097/INF.0b013e3181daf921. PMID 20375709
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study are summarised with studies 108498 (second cohort study) and 108500 (third cohort study) on the GSK Clinical Study Register.
- Available data/document: Dataset Specification: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107066 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 138 subjects were enrolled as part of the first 107066/Phase A part of this NCT00502593 study. This first part was then followed by a second and third part (Phases B [study 108498] and C [study 108500] during which 134 and 133 subjects were enrolled, respectively. Duration of the study was of 24 months for all subjects.
Pre-assignment Details: For safety reasons, subjects in each group were enrolled in a staggered manner, with enrolment taking place sequentially into 2 age strata, '6-9 years' 1st, and '3-5 years' next.
Period: Overall Study
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Started | 51 | 18 | 51 | 18 | 51 | 17 | 49 | 17 | 49 | 17 | 49 | 18
Completed | 48 | 16 | 41 | 14 | 47 | 17 | 44 | 17 | 43 | 17 | 47 | 18
Not Completed | 3 | 2 | 10 | 4 | 4 | 0 | 5 | 0 | 6 | 0 | 2 | 0
Not completed — Withdrawn unspecified reason | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 2 | 2 | 0 | 3 | 0 | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK1562902A -A Lot 1 3-5Y Group: Subjects aged 3-5 years received 2 doses of GSK1562902A vaccine, lot 1. These subjects were enrolled in the Phase A of this NCT00502593 study (or study 107066). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
- Total: Total of all reporting groups
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group | Total
Number analyzed (Participants) | 51 | 18 | 51 | 18 | 51 | 17 | 49 | 17 | 49 | 17 | 49 | 18 | 405
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.9 (0.84) | 3.6 (0.70) | 7.6 (1.06) | 7.6 (1.38) | 4.2 (0.85) | 4.4 (0.79) | 7.3 (1.28) | 7.2 (1.20) | 4.2 (0.85) | 3.9 (0.93) | 7.0 (1.06) | 7.4 (0.98) | 6.1 (0.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 24 | 7 | 25 | 10 | 19 | 3 | 22 | 11 | 18 | 9 | 182
  Male | 26 | 9 | 27 | 11 | 26 | 7 | 30 | 14 | 27 | 6 | 31 | 9 | 223

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: Titers of serum HI antibodies are presented as geometric mean titers (GMTs). The 2 influenza strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO). The cut-off of the assay was the seropositivity cut-off value of 1:10.
Time Frame: At Day 0
Population: The analysis was based on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, e.g. for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 42 | 16 | 45 | 17 | 44 | 15 | 43 | 13
Titer
  A/VIET | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.1 [4.9 to 5.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 41 | 16 | 45 | 17 | 43 | 15 | 30 | 9
Titer
  A/VIET | 8.7 [6.2 to 12.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 12.1 [8.4 to 17.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 22.7 [14.6 to 35.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 23.7 [14.3 to 39.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 25.0 [16.0 to 39.3] | 5.7 [4.3 to 7.7] | 27.3 [16.2 to 46.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | 5.2 [4.9 to 5.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.2 [4.8 to 5.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.5 [4.9 to 6.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.3 [4.9 to 5.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 7.7 [6.0 to 9.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 6.0 [5.0 to 7.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

3. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The 2 flu strains assessed were A/Vietnam/1194/2004 (A/VIET) and A/Indonesia/5/2005 (A/INDO). The cut-off of the assay was the seropositivity cut-off value of 1:10
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 42 | 16 | 45 | 17 | 44 | 15 | 43 | 13
Titer
  A/VIET | 392.7 [280.4 to 550.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 540.3 [424.5 to 687.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 678.1 [475.7 to 966.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 615.8 [429 to 884] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 956.4 [769.2 to 1189.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 883.5 [737.3 to 1058.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | 53.5 [35 to 81.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 60.8 [38.7 to 95.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 73.7 [45.2 to 120.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 64.9 [38.7 to 108.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 167.9 [121.7 to 231.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 92.5 [59.3 to 144.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

4. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: At Month 6
Population: The analysis was performed on the According-to-Protocol cohort for persistence, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component on Month 6/Day 180, Month 12 and Month 24.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 50 | 15 | 44 | 14 | 47 | 16 | 45 | 17 | 29 | 11 | 41 | 16
Titer
  A/VIET | 29.3 [19.2 to 44.6] | 5.9 [4.2 to 8.3] | 33.4 [21.2 to 52.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 46.3 [29.8 to 72.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 43.2 [27.9 to 66.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 80.0 [47.0 to 136.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 61.5 [38.9 to 97.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | 6.9 [5.6 to 8.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 6.6 [5.2 to 8.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 21.7 [14.3 to 33.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 11.9 [8.4 to 16.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 42.5 [23.7 to 76.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 36.8 [22.3 to 60.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

5. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 3
Time Frame: At Month 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 14 | 37 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
Titer
  A/VIET | 13.9 [9.7 to 20.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 12.0 [8.0 to 18.1] | 5.8 [4.2 to 8.0] | 19.8 [13.6 to 28.8] | 5.2 [4.8 to 5.7] | 22.4 [15.4 to 32.5] | 5.2 [4.8 to 5.7] | 23.9 [15.1 to 37.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 27.7 [19.1 to 40.4] | 5.4 [4.6 to 6.4]
  A/INDO | 13.0 [9.1 to 18.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 10.5 [7.0 to 15.8] | 5.5 [4.5 to 6.8] | 16.4 [11.4 to 23.5] | 5.9 [4.5 to 7.9] | 15.0 [11.1 to 20.1] | 6.5 [5.2 to 8.2] | 18.5 [11.5 to 29.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 20.4 [13.4 to 31.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

6. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 1
Time Frame: At Month 24
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 13 | 37 | 11 | 39 | 16 | 42 | 16 | 26 | 10 | 34 | 13
Titer
  A/VIET | 14.9 [10.3 to 21.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 13.2 [9.1 to 19.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 52.2 [33.6 to 81.1] | 6.8 [4.7 to 9.7] | 20.1 [13.9 to 29.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 55.8 [33.2 to 93.8] | 6.6 [3.5 to 12.4] | 36.5 [24.8 to 53.8] | 6.2 [3.9 to 9.8]
  A/INDO | 10.1 [7.7 to 13.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 7.7 [5.9 to 10.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 22.7 [15.2 to 33.7] | 5.3 [4.6 to 6.1] | 8.7 [7.0 to 10.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 27.5 [16.1 to 47] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 18.2 [12.1 to 27.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

7. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: A seroconverted subject was a subject with a pre-vaccination serum haemagglutination-inhibition (HI) antibody titer below (<) 1:10 and a post-vaccination HI antibody titer above than or equal to (≥)1:40 or a pre-vaccination HI antibody titer ≥ 1:10 and at least four-fold increase in post-vaccination HI antibody titer. The 2 strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 41 | 16 | 45 | 17 | 43 | 15 | 30 | 9
Participants
  A/VIET | 6 | 0 | 13 | 0 | 20 | 0 | 19 | 0 | 20 | 1 | 17 | 0
  A/INDO | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0

8. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: A seroconverted subject was a subject with a pre-vaccination serum haemagglutination-inhibition (HI) antibody titer < 1:10 and a post-vaccination HI antibody titer ≥1:40 or a pre-vaccination HI antibody titer ≥ 1:10 and at least four-fold increase in post-vaccination HI antibody titer. The 2 strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 42 | 16 | 45 | 17 | 44 | 15 | 43 | 13
Participants
  A/VIET | 47 | 0 | 43 | 0 | 41 | 0 | 44 | 0 | 44 | 0 | 43 | 0
  A/INDO | 35 | 0 | 32 | 0 | 32 | 0 | 31 | 0 | 42 | 0 | 34 | 0

9. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 8
Time Frame: At Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 50 | 15 | 41 | 14 | 47 | 16 | 45 | 17 | 29 | 11 | 41 | 16
Participants
  A/VIET | 28 | 1 | 25 | 0 | 32 | 0 | 31 | 0 | 24 | 0 | 32 | 0
  A/INDO | 3 | 0 | 1 | 0 | 23 | 0 | 12 | 0 | 20 | 0 | 25 | 0

10. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 8
Time Frame: At Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 14 | 37 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
Participants
  A/VIET | 18 | 0 | 8 | 1 | 17 | 0 | 20 | 0 | 13 | 0 | 22 | 0
  A/INDO | 17 | 0 | 6 | 0 | 16 | 1 | 7 | 0 | 12 | 0 | 15 | 0

11. Primary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease
Description: as for outcome 8
Time Frame: At Month 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 13 | 35 | 11 | 39 | 16 | 42 | 16 | 26 | 10 | 34 | 13
Participants
  A/VIET | 18 | 0 | 8 | 0 | 30 | 1 | 18 | 0 | 19 | 1 | 23 | 1
  A/INDO | 5 | 0 | 3 | 0 | 19 | 0 | 2 | 0 | 14 | 0 | 10 | 0

12. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 41 | 16 | 45 | 17 | 43 | 15 | 30 | 9
Fold
  A/VIET | 1.7 [1.2 to 2.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 2.4 [1.7 to 3.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 4.4 [2.9 to 6.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 4.7 [2.9 to 7.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.0 [3.2 to 7.9] | 1.1 [0.9 to 1.5] | 5.5 [3.2 to 9.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.1 [1.0 to 1.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.1 [1.0 to 1.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.5 [1.2 to 2.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.2 [1.0 to 1.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

13. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 12
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 42 | 16 | 45 | 17 | 44 | 15 | 43 | 13
Fold
  A/VIET | 78.5 [56.1 to 110.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 108.1 [84.9 to 137.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 132.3 [91.8 to 190.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 123.2 [85.8 to 176.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 191.3 [153.8 to 237.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 176.7 [147.5 to 211.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | 10.7 [7.0 to 16.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 12.2 [7.7 to 19.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 14.7 [9.0 to 24.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 13.0 [7.7 to 21.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 33.6 [24.3 to 46.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 18.5 [11.9 to 28.8] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

14. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 12
Time Frame: At Month 6
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 50 | 15 | 41 | 14 | 47 | 16 | 45 | 17 | 29 | 11 | 41 | 16
Fold
  A/VIET | 5.9 [3.8 to 8.9] | 1.2 [0.8 to 1.7] | 6.1 [3.8 to 9.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 9.1 [5.8 to 14.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 8.6 [5.6 to 13.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 16.0 [9.4 to 27.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 12.3 [7.8 to 19.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)
  A/INDO | 1.4 [1.1 to 1.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.2 [1.0 to 1.5] | 1.2 [1.0 to 1.5] | 4.3 [2.9 to 6.6] | 1.1 [0.9 to 1.4] | 2.4 [1.7 to 3.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 8.5 [4.7 to 15.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 7.4 [4.5 to 12.1] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

15. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 2 flu strains assessed were A/Vietnam/1194/2004 (A/VIET) and A/Indonesia/5/2005 (A/INDO).
Time Frame: At Month 12
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 14 | 35 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
Fold
  A/VIET | 2.8 [1.9 to 4.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 2.2 [1.5 to 3.3] | 1.2 [0.8 to 1.6] | 4.0 [2.7 to 5.8] | 1.0 [1.0 to 1.1] | 4.5 [3.1 to 6.5] | 1.0 [1.0 to 1.1] | 4.8 [3.0 to 7.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.5 [3.8 to 8.1] | 1.1 [0.9 to 1.3]
  A/INDO: number analyzed (Participants) | 47 | 14 | 34 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
  A/INDO | 2.6 [1.8 to 3.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.9 [1.3 to 2.8] | 1.1 [0.9 to 1.4] | 3.3 [2.3 to 4.7] | 1.2 [0.9 to 1.6] | 3.0 [2.2 to 4.0] | 1.3 [1.0 to 1.6] | 3.7 [2.3 to 6.0] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 4.1 [2.7 to 6.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

16. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 2 Strains of Influenza Disease
Description: as for outcome 15
Time Frame: At Month 24
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 13 | 35 | 11 | 39 | 16 | 42 | 16 | 26 | 10 | 34 | 13
Fold
  A/VIET | 3.0 [2.1 to 4.3] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 2.5 [1.7 to 3.6] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 10.4 [6.7 to 16.2] | 1.4 [0.9 to 1.9] | 4.0 [2.8 to 5.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 11.2 [6.6 to 18.8] | 1.3 [0.7 to 2.5] | 7.3 [5.0 to 10.8] | 1.2 [0.8 to 2.0]
  A/INDO | 2.0 [1.5 to 2.7] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 1.5 [1.1 to 1.9] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 4.5 [3.0 to 6.7] | 1.1 [0.9 to 1.2] | 1.7 [1.4 to 2.2] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 5.5 [3.2 to 9.4] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation) | 3.6 [2.4 to 5.5] | NA [NA to NA] — Data was not computed (titers below cut-off value for titer calculation)

17. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with a haemagglutination-inhibition (HI) antibody titer above or equal to the seroprotection threshold of 1:40. The 2 influenza strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/5/2005 (A/INDO).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 45 | 17 | 42 | 16 | 44 | 15 | 43 | 13
Participants
  A/VIET | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  A/INDO | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: as for outcome 17
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 41 | 16 | 45 | 17 | 43 | 15 | 30 | 9
Participants
  A/VIET | 6 | 0 | 13 | 0 | 20 | 0 | 19 | 0 | 20 | 1 | 17 | 0
  A/INDO | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0

19. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: as for outcome 17
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 15 | 43 | 15 | 42 | 16 | 45 | 17 | 44 | 15 | 43 | 13
Participants
  A/VIET | 47 | 0 | 43 | 0 | 41 | 0 | 44 | 0 | 44 | 0 | 43 | 0
  A/INDO | 35 | 0 | 32 | 0 | 32 | 0 | 31 | 0 | 42 | 0 | 34 | 0

20. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: as for outcome 17
Time Frame: At Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 50 | 15 | 44 | 14 | 47 | 16 | 45 | 17 | 29 | 11 | 41 | 16
Participants
  A/VIET | 28 | 1 | 28 | 0 | 33 | 0 | 31 | 0 | 24 | 0 | 32 | 0
  A/INDO | 3 | 0 | 2 | 0 | 23 | 0 | 12 | 0 | 20 | 0 | 25 | 0

21. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: as for outcome 17
Time Frame: At Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 14 | 37 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
Participants
  A/VIET | 18 | 0 | 9 | 1 | 17 | 0 | 20 | 0 | 13 | 0 | 22 | 0
  A/INDO: number analyzed (Participants) | 47 | 14 | 36 | 14 | 40 | 16 | 43 | 16 | 27 | 10 | 35 | 13
  A/INDO | 17 | 0 | 7 | 0 | 16 | 1 | 7 | 0 | 12 | 0 | 15 | 0

22. Primary Outcome: Number of Seroprotected Subjects Against the 2 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI antibody titer ≥ 1:40, a level of HI antibody that has been viewed as correlating with protection against influenza. The 2 influenza strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/5/2005 (A/INDO).
Time Frame: At Month 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 47 | 13 | 37 | 11 | 39 | 16 | 42 | 16 | 26 | 10 | 34 | 13
Participants
  A/VIET | 18 | 0 | 9 | 0 | 30 | 1 | 18 | 0 | 19 | 1 | 23 | 1
  A/INDO | 5 | 0 | 4 | 0 | 19 | 0 | 2 | 0 | 14 | 0 | 10 | 0

23. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling at the injection site. Any = occurrence of a symptom regardless of intensity. Grade 3 pain = significant pain at rest/ that prevented normal activities. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling larger than (>) 100 millimeters (mm). All solicited local symptoms were considered to be related to study vaccination. This outcome presents results from subjects participating in Phase A of the study.
Time Frame: During the 7 day follow-up period after each vaccination
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 51 | 18 | 51 | 18
Participants
  Any ecchymosis | 9 | 3 | 3 | 2
  Ecchymosis >50mm | 0 | 0 | 0 | 0
  Any induration | 7 | 1 | 12 | 6
  Induration >50mm | 1 | 0 | 0 | 1
  Any pain | 31 | 7 | 44 | 12
  Grade 3 pain | 2 | 0 | 5 | 0
  Any redness | 10 | 2 | 12 | 5
  Redness >50mm | 0 | 0 | 0 | 0
  Any swelling | 10 | 1 | 14 | 7
  Swelling >50mm | 1 | 0 | 1 | 0

24. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling at the injection site. Any = occurrence of a symptom regardless of intensity. Grade 3 pain = significant pain at rest/ that prevented normal activities. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling larger than (>) 100 millimeters (mm). All solicited local symptoms were considered to be related to study vaccination. This outcome presents results from subjects participating in Phase C of the study.
Time Frame: During the 7-day follow-up period after each vaccination
Population: The analysis was based on theTotal Vaccinated cohort, which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 49 | 17 | 49 | 18
Participants
  Any ecchymosis | 4 | 0 | 0 | 2
  Ecchymosys >50mm | 0 | 0 | 0 | 0
  Any induration | 14 | 0 | 10 | 1
  Induration >50mm | 1 | 0 | 1 | 0
  Any pain | 37 | 7 | 44 | 15
  Grade 3 pain | 5 | 0 | 3 | 0
  Any redness | 16 | 2 | 6 | 1
  Redness >50mm | 1 | 0 | 2 | 0
  Any swelling | 18 | 2 | 14 | 3
  Swelling >50mm | 2 | 0 | 2 | 0

25. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever (axillary temperature above or equal (≥) 37.5°C), irritability, loss of appetite, shivering, sweating and vomiting. Any = occurrence of a symptom regardless of intensity or relationship to vaccination. Grade 3 = general symptom that prevented normal activity. Grade 3 temperature = axillary temperature > 39.0°C. Related = symptom assessed as causally related to study vaccination. This outcome presents results for subjects aged between 3 and 5 years participating in Phases A, B and C of the study.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group
Number analyzed (Participants) | 51 | 18 | 51 | 17 | 49 | 17
Participants
  Any drowsiness | 7 | 1 | 9 | 1 | 12 | 1
  Grade 3 drowsiness | 1 | 0 | 1 | 0 | 2 | 0
  Related drowsiness | 6 | 1 | 6 | 0 | 12 | 1
  Fever (Axillary) >=37.5 deg C | 8 | 0 | 10 | 2 | 18 | 0
  Fever >39degC (Axillary) | 2 | 0 | 0 | 1 | 5 | 0
  Related fever (Axillary) | 6 | 0 | 5 | 1 | 17 | 0
  Any irritability | 9 | 1 | 13 | 2 | 18 | 0
  Grade 3 irritability | 0 | 0 | 0 | 0 | 1 | 0
  Related irritability | 7 | 1 | 9 | 1 | 15 | 0
  Any loss of appetite | 12 | 1 | 8 | 1 | 15 | 1
  Grade 3 loss of appetite | 3 | 0 | 1 | 0 | 5 | 0
  Related loss of appetite | 4 | 1 | 5 | 1 | 13 | 1
  Any shivering | 1 | 0 | 4 | 1 | 10 | 1
  Grade 3 shivering | 0 | 0 | 0 | 0 | 0 | 0
  Related shivering | 1 | 0 | 2 | 0 | 9 | 1
  Any sweating | 4 | 0 | 1 | 0 | 4 | 0
  Grade 3 sweating | 0 | 0 | 0 | 0 | 1 | 0
  Related sweating | 2 | 0 | 1 | 0 | 3 | 0
  Any vomiting | 7 | 0 | 6 | 0 | 6 | 1
  Grade 3 vomiting | 0 | 0 | 1 | 0 | 0 | 0
  Related vomiting | 3 | 0 | 2 | 0 | 3 | 1

26. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms were arthralgia, fatigue, headache, muscle aches, shivering and fever, assessed as oral temperature above or equal (≥) 37.0 degrees Celsius (°C). Any = occurrence of a symptom regardless of intensity or relationship to vaccination. Grade 3 = general symptom that prevented normal activity, everyday activities, or required intervention of a physician/healthcare provider. Grade 3 fever= oral temperature ≥ 39.0°C. Related = symptom assessed as causally related to study vaccination. This outcome presents results related to subjects aged 6 to 9 years participating in the study phases A, B and C.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 51 | 18 | 49 | 17 | 49 | 18
Participants
  Any arthralgia | 6 | 3 | 7 | 0 | 9 | 2
  Grade 3 arthralgia | 0 | 0 | 1 | 0 | 0 | 0
  Related arthralgia | 6 | 3 | 7 | 0 | 7 | 2
  Any fatigue | 7 | 1 | 6 | 1 | 11 | 2
  Grade 3 fatigue | 0 | 0 | 0 | 0 | 1 | 0
  Related fatigue | 7 | 1 | 6 | 1 | 11 | 2
  Fever >=37.5 deg C | 7 | 3 | 3 | 0 | 18 | 0
  Fever >39.0 deg C | 0 | 1 | 1 | 0 | 7 | 0
  Related fever | 6 | 2 | 1 | 0 | 17 | 0
  Any gastrointestinal symptoms | 9 | 5 | 4 | 5 | 16 | 5
  Grade 3 gastrointestinal symptoms | 1 | 0 | 1 | 0 | 0 | 1
  Related gastrointestinal symptoms | 8 | 4 | 2 | 2 | 13 | 3
  Any headache | 20 | 5 | 11 | 2 | 25 | 3
  Grade 3 headache | 2 | 0 | 2 | 0 | 3 | 0
  Related headache | 16 | 3 | 8 | 2 | 22 | 3
  Any myalgia | 10 | 3 | 11 | 2 | 13 | 2
  Grade 3 myalgia | 1 | 0 | 1 | 0 | 1 | 0
  Related myalgia | 9 | 3 | 11 | 1 | 11 | 2
  Any shivering | 3 | 1 | 7 | 0 | 13 | 3
  Grade 3 Shivering | 0 | 0 | 0 | 0 | 2 | 0
  Related Shivering | 3 | 1 | 5 | 0 | 13 | 2
  Any sweating | 3 | 2 | 3 | 2 | 6 | 1
  Grade 3 sweating | 0 | 0 | 0 | 0 | 0 | 0
  Related sweating | 3 | 2 | 1 | 1 | 6 | 1

27. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling at the injection site. Any = occurrence of a symptom regardless of intensity. Grade 3 pain = significant pain at rest/ that prevented normal activities. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling larger than (>) 100 millimeters (mm). All solicited local symptoms were considered to be related to study vaccination. This outcome presents results from subjects participating to Phase B of the study.
Time Frame: During the 7-day follow-up period after each vaccination
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 49 | 17
Participants
  Any ecchymosis | 4 | 0 | 4 | 1
  Ecchymosis >50mm | 0 | 0 | 0 | 0
  Any induration | 4 | 1 | 6 | 1
  Induration >50mm | 0 | 0 | 1 | 0
  Any pain | 27 | 3 | 36 | 9
  Grade 3 pain | 5 | 0 | 3 | 0
  Any redness | 6 | 4 | 6 | 3
  Redness >50mm | 1 | 0 | 0 | 0
  Any swelling | 9 | 2 | 10 | 2
  Swelling >50mm | 0 | 0 | 1 | 0

28. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any SAE = any SAE regardless of intensity or relationship to vaccination.
Time Frame: During the entire study (Day 0 to Month 24)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 51 | 18 | 51 | 18 | 51 | 17 | 49 | 17 | 49 | 17 | 49 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0

29. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event. Grade 3 AE = AE that prevented normal activity, everyday activities, or required intervention of a physician/healthcare provider. Related = symptom assessed as causally related to study vaccination.
Time Frame: During a 21 day follow-up period after the first vaccination, during a 30-day follow-up period after the second vaccination
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 51 | 18 | 51 | 18 | 51 | 17 | 49 | 17 | 49 | 17 | 49 | 18
Participants
  Subjects with any AE(s) | 29 | 12 | 10 | 5 | 28 | 9 | 19 | 6 | 26 | 8 | 27 | 6
  Subjects with any Grade 3 AE(s) | 4 | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 3 | 0 | 1 | 1
  Subjects with any related AE(s) | 6 | 2 | 2 | 1 | 3 | 1 | 4 | 1 | 9 | 0 | 3 | 1

30. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Alanine Aminotransferase (ALT) for Subjects in Study Phase A
Description: Changes from baseline are categorised as below, within(normal), or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for ALT for subjects participating in Phase A of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  ALT,Unknown,Day 21,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Unknown,Day 21,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 21,Normal | 1 | 0 | 0 | 1
  ALT,Unknown,Day 21,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  ALT,Unknown,Day 21,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  ALT,Normal,Day 21,Below: number analyzed (Participants) | 48 | 17 | 48 | 17
  ALT,Normal,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Normal,Day 21,Normal: number analyzed (Participants) | 48 | 17 | 48 | 17
  ALT,Normal,Day 21,Normal | 47 | 16 | 44 | 17
  ALT,Normal,Day 21,Above: number analyzed (Participants) | 48 | 17 | 48 | 17
  ALT,Normal,Day 21,Above | 0 | 0 | 0 | 0
  ALT,Normal,Day 21,Unknown: number analyzed (Participants) | 48 | 17 | 48 | 17
  ALT,Normal,Day 21,Unknown | 1 | 1 | 4 | 0
  ALT,Unknown,Day 42,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Unknown,Day 42,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 42,Normal | 1 | 0 | 0 | 1
  ALT,Unknown,Day 42,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  ALT,Unknown,Day 42,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  ALT,Normal,Day 42,Below: number analyzed (Participants) | 49 | 17 | 49 | 17
  ALT,Normal,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Normal,Day 42,Normal: number analyzed (Participants) | 49 | 17 | 49 | 17
  ALT,Normal,Day 42,Normal | 48 | 15 | 45 | 15
  ALT,Normal,Day 42,Above: number analyzed (Participants) | 49 | 17 | 49 | 17
  ALT,Normal,Day 42,Above | 0 | 1 | 0 | 0
  ALT,Normal,Day 42,Unknown: number analyzed (Participants) | 49 | 17 | 49 | 17
  ALT,Normal,Day 42,Unknown | 1 | 1 | 4 | 2
  ALT,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  ALT,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  ALT,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  ALT,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  ALT,Normal, Month 6,Below: number analyzed (Participants) | 49 | 17 | 47 | 16
  ALT,Normal, Month 6,Below | 0 | 0 | 0 | 0
  ALT,Normal, Month 6,Normal: number analyzed (Participants) | 49 | 17 | 47 | 16
  ALT,Normal, Month 6,Normal | 47 | 15 | 42 | 16
  ALT,Normal, Month 6,Above: number analyzed (Participants) | 49 | 17 | 47 | 16
  ALT,Normal, Month 6,Above | 1 | 0 | 1 | 0
  ALT,Normal, Month 6,Unknown: number analyzed (Participants) | 49 | 17 | 47 | 16
  ALT,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  ALT,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  ALT,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  ALT,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  ALT,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  ALT,Normal, Month 12,Below: number analyzed (Participants) | 49 | 17 | 44 | 16
  ALT,Normal, Month 12,Below | 0 | 0 | 0 | 0
  ALT,Normal, Month 12,Normal: number analyzed (Participants) | 49 | 17 | 44 | 16
  ALT,Normal, Month 12,Normal | 45 | 17 | 41 | 16
  ALT,Normal, Month 12,Above: number analyzed (Participants) | 49 | 17 | 44 | 16
  ALT,Normal, Month 12,Above | 1 | 0 | 1 | 0
  ALT,Normal, Month 12,Unknown: number analyzed (Participants) | 49 | 17 | 44 | 16
  ALT,Normal, Month 12,Unknown | 3 | 0 | 2 | 0
  ALT,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  ALT,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  ALT,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  ALT,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  ALT,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  ALT,Normal, Month 24,Below: number analyzed (Participants) | 46 | 16 | 42 | 13
  ALT,Normal, Month 24,Below | 0 | 0 | 0 | 0
  ALT,Normal, Month 24,Normal: number analyzed (Participants) | 46 | 16 | 42 | 13
  ALT,Normal, Month 24,Normal | 46 | 16 | 40 | 13
  ALT,Normal, Month 24,Above: number analyzed (Participants) | 46 | 16 | 42 | 13
  ALT,Normal, Month 24,Above | 0 | 0 | 0 | 0
  ALT,Normal, Month 24,Unknown: number analyzed (Participants) | 46 | 16 | 42 | 13
  ALT,Normal, Month 24,Unknown | 0 | 0 | 2 | 0

31. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Aspartate Aminotransferase (AST) in Study Phase A
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for AST for subjects participating in Phase A of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  AST,Unknown,Day 21,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  AST,Unknown,Day 21,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 21,Normal | 1 | 0 | 0 | 1
  AST,Unknown,Day 21,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  AST,Unknown,Day 21,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  AST,Normal,Day 21,Below: number analyzed (Participants) | 44 | 17 | 48 | 17
  AST,Normal,Day 21,Below | 0 | 0 | 0 | 0
  AST,Normal,Day 21,Normal: number analyzed (Participants) | 44 | 17 | 48 | 17
  AST,Normal,Day 21,Normal | 39 | 16 | 44 | 16
  AST,Normal,Day 21,Above: number analyzed (Participants) | 44 | 17 | 48 | 17
  AST,Normal,Day 21,Above | 4 | 0 | 0 | 0
  AST,Normal,Day 21,Unknown: number analyzed (Participants) | 44 | 17 | 48 | 17
  AST,Normal,Day 21,Unknown | 1 | 1 | 4 | 1
  AST,Above,Day 21,Below: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 21,Below | 0 | 0 | 0 | 0
  AST,Above,Day 21,Normal: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 21,Normal | 2 | 0 | 0 | 0
  AST,Above,Day 21,Above: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 21,Above | 2 | 0 | 0 | 0
  AST,Above,Day 21,Unknown: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 21,Unknown | 0 | 0 | 0 | 0
  AST,Unknown,Day 42,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  AST,Unknown,Day 42,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 42,Normal | 1 | 0 | 0 | 1
  AST,Unknown,Day 42,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  AST,Unknown,Day 42,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  AST,Normal,Day 42,Below: number analyzed (Participants) | 45 | 17 | 49 | 17
  AST,Normal,Day 42,Below | 0 | 0 | 0 | 0
  AST,Normal,Day 42,Normal: number analyzed (Participants) | 45 | 17 | 49 | 17
  AST,Normal,Day 42,Normal | 42 | 13 | 45 | 15
  AST,Normal,Day 42,Above: number analyzed (Participants) | 45 | 17 | 49 | 17
  AST,Normal,Day 42,Above | 2 | 2 | 0 | 0
  AST,Normal,Day 42,Unknown: number analyzed (Participants) | 45 | 17 | 49 | 17
  AST,Normal,Day 42,Unknown | 1 | 2 | 4 | 2
  AST,Above,Day 42,Below: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 42,Below | 0 | 0 | 0 | 0
  AST,Above,Day 42,Normal: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 42,Normal | 3 | 0 | 0 | 0
  AST,Above,Day 42,Above: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 42,Above | 1 | 0 | 0 | 0
  AST,Above,Day 42,Unknown: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  AST,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  AST,Normal, Month 6,Below: number analyzed (Participants) | 45 | 17 | 47 | 16
  AST,Normal, Month 6,Below | 0 | 0 | 0 | 0
  AST,Normal, Month 6,Normal: number analyzed (Participants) | 45 | 17 | 47 | 16
  AST,Normal, Month 6,Normal | 42 | 14 | 42 | 16
  AST,Normal, Month 6,Above: number analyzed (Participants) | 45 | 17 | 47 | 16
  AST,Normal, Month 6,Above | 2 | 1 | 1 | 0
  AST,Normal, Month 6,Unknown: number analyzed (Participants) | 45 | 17 | 47 | 16
  AST,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  AST,Above, Month 6,Below: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 6,Below | 0 | 0 | 0 | 0
  AST,Above,Month 6,Normal: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above,Month 6,Normal | 3 | 0 | 0 | 0
  AST,Above, Month 6,Above: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 6,Above | 1 | 0 | 0 | 0
  AST,Above, Month 6,Unknown: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  AST,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  AST,Normal, Month 12,Below: number analyzed (Participants) | 45 | 17 | 44 | 16
  AST,Normal, Month 12,Below | 0 | 0 | 0 | 0
  AST,Normal, Month 12,Normal: number analyzed (Participants) | 45 | 17 | 44 | 16
  AST,Normal, Month 12,Normal | 41 | 16 | 42 | 16
  AST,Normal, Month 12,Above: number analyzed (Participants) | 45 | 17 | 44 | 16
  AST,Normal, Month 12,Above | 2 | 1 | 0 | 0
  AST,Normal, Month 12,Unknown: number analyzed (Participants) | 45 | 17 | 44 | 16
  AST,Normal, Month 12,Unknown | 2 | 0 | 2 | 0
  AST,Above, Month 12,Below: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 12,Below | 0 | 0 | 0 | 0
  AST,Above, Month 12,Normal: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 12,Normal | 1 | 0 | 0 | 0
  AST,Above, Month 12,Above: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 12,Above | 2 | 0 | 0 | 0
  AST,Above, Month 12,Unknown: number analyzed (Participants) | 4 | 0 | 0 | 0
  AST,Above, Month 12,Unknown | 1 | 0 | 0 | 0
  AST,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  AST,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  AST,Normal,Month 24,Below: number analyzed (Participants) | 43 | 16 | 42 | 13
  AST,Normal,Month 24,Below | 0 | 0 | 0 | 0
  AST,Normal,Month 24,Normal: number analyzed (Participants) | 43 | 16 | 42 | 13
  AST,Normal,Month 24,Normal | 41 | 16 | 40 | 13
  AST,Normal,Month 24,Above: number analyzed (Participants) | 43 | 16 | 42 | 13
  AST,Normal,Month 24,Above | 2 | 0 | 0 | 0
  AST,Normal,Month 24,Unknown: number analyzed (Participants) | 43 | 16 | 42 | 13
  AST,Normal,Month 24,Unknown | 0 | 0 | 2 | 0
  AST,Above,Month 24,Below: number analyzed (Participants) | 3 | 0 | 0 | 0
  AST,Above,Month 24,Below | 0 | 0 | 0 | 0
  AST,Above,Month 24,Normal: number analyzed (Participants) | 3 | 0 | 0 | 0
  AST,Above,Month 24,Normal | 2 | 0 | 0 | 0
  AST,Above,Month 24,Above: number analyzed (Participants) | 3 | 0 | 0 | 0
  AST,Above,Month 24,Above | 1 | 0 | 0 | 0
  AST,Above,Month 24,Unknown: number analyzed (Participants) | 3 | 0 | 0 | 0
  AST,Above,Month 24,Unknown | 0 | 0 | 0 | 0

32. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Urea Nitrogen (BUN) in Study Phase A
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for BUN for subjects participating in Phase A of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  BUN,Unknown, Day 21, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 21, Below | 0 | 0 | 0 | 0
  BUN,Unknown, Day 21, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 21, Normal | 1 | 0 | 0 | 0
  BUN,Unknown, Day 21, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 21, Above | 0 | 0 | 0 | 1
  BUN,Unknown, Day 21, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 21, Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Day 21, Below: number analyzed (Participants) | 46 | 17 | 47 | 16
  BUN,Normal, Day 21, Below | 0 | 1 | 0 | 0
  BUN,Normal, Day 21, Normal: number analyzed (Participants) | 46 | 17 | 47 | 16
  BUN,Normal, Day 21, Normal | 43 | 14 | 38 | 16
  BUN,Normal, Day 21, Above: number analyzed (Participants) | 46 | 17 | 47 | 16
  BUN,Normal, Day 21, Above | 2 | 1 | 5 | 0
  BUN,Normal, Day 21, Unknown: number analyzed (Participants) | 46 | 17 | 47 | 16
  BUN,Normal, Day 21, Unknown | 1 | 1 | 4 | 0
  BUN,Above, Day 21, Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 21, Below | 0 | 0 | 0 | 0
  BUN,Above, Day 21, Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 21, Normal | 1 | 0 | 1 | 0
  BUN,Above, Day 21, Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 21, Above | 1 | 0 | 0 | 1
  BUN,Above, Day 21, Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 21, Unknown | 0 | 0 | 0 | 0
  BUN,Unknown, Day 42, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 42, Below | 0 | 0 | 0 | 0
  BUN,Unknown, Day 42, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 42, Normal | 1 | 0 | 0 | 1
  BUN,Unknown, Day 42, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 42, Above | 0 | 0 | 0 | 0
  BUN,Unknown, Day 42, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Day 42, Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Day 42, Below: number analyzed (Participants) | 47 | 17 | 48 | 16
  BUN,Normal, Day 42, Below | 0 | 0 | 0 | 0
  BUN,Normal, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 48 | 16
  BUN,Normal, Day 42, Normal | 40 | 16 | 38 | 12
  BUN,Normal, Day 42,Above: number analyzed (Participants) | 47 | 17 | 48 | 16
  BUN,Normal, Day 42,Above | 6 | 0 | 6 | 2
  BUN,Normal, Day 42, Unknown: number analyzed (Participants) | 47 | 17 | 48 | 16
  BUN,Normal, Day 42, Unknown | 1 | 1 | 4 | 2
  BUN,Above, Day 42, Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 42, Below | 0 | 0 | 0 | 0
  BUN,Above, Day 42, Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 42, Normal | 1 | 0 | 1 | 1
  BUN,Above, Day 42, Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 42, Above | 1 | 0 | 0 | 0
  BUN,Above, Day 42, Unknkwn: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Day 42, Unknkwn | 0 | 0 | 0 | 0
  BUN,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  BUN,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 6,Below: number analyzed (Participants) | 47 | 17 | 46 | 15
  BUN,Normal, Month 6,Below | 0 | 1 | 0 | 0
  BUN,Normal, Month 6,Normal: number analyzed (Participants) | 47 | 17 | 46 | 15
  BUN,Normal, Month 6,Normal | 43 | 13 | 38 | 14
  BUN,Normal, Month 6,Above: number analyzed (Participants) | 47 | 17 | 46 | 15
  BUN,Normal, Month 6,Above | 3 | 1 | 4 | 1
  BUN,Normal, Month 6,Unknown: number analyzed (Participants) | 47 | 17 | 46 | 15
  BUN,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  BUN,Above, Month 6,Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 6,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 6,Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above,Month 6,Normal | 2 | 0 | 1 | 0
  BUN,Above, Month 6,Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 6,Above | 0 | 0 | 0 | 1
  BUN,Above, Month 6,Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  BUN,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 12,Below: number analyzed (Participants) | 47 | 17 | 43 | 15
  BUN,Normal, Month 12,Below | 0 | 0 | 1 | 0
  BUN,Normal, Month 12,Normal: number analyzed (Participants) | 47 | 17 | 43 | 15
  BUN,Normal, Month 12,Normal | 41 | 16 | 40 | 13
  BUN,Normal, Month 12,Above: number analyzed (Participants) | 47 | 17 | 43 | 15
  BUN,Normal, Month 12,Above | 3 | 1 | 0 | 2
  BUN,Normal, Month 12,Unknown: number analyzed (Participants) | 47 | 17 | 43 | 15
  BUN,Normal, Month 12,Unknown | 3 | 0 | 2 | 0
  BUN,Above, Month 12,Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 12,Below | 0 | 0 | 0 | 0
  BUN,Above, Month 12,Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 12,Normal | 0 | 0 | 1 | 1
  BUN,Above, Month 12,Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 12,Above | 2 | 0 | 0 | 0
  BUN,Above, Month 12,Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  BUN,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  BUN,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 24,Below: number analyzed (Participants) | 44 | 16 | 41 | 12
  BUN,Normal, Month 24,Below | 0 | 0 | 1 | 0
  BUN,Normal, Month 24,Normal: number analyzed (Participants) | 44 | 16 | 41 | 12
  BUN,Normal, Month 24,Normal | 42 | 16 | 37 | 11
  BUN,Normal, Month 24,Above: number analyzed (Participants) | 44 | 16 | 41 | 12
  BUN,Normal, Month 24,Above | 2 | 0 | 1 | 1
  BUN,Normal, Month 24,Unknown: number analyzed (Participants) | 44 | 16 | 41 | 12
  BUN,Normal, Month 24,Unknown | 0 | 0 | 2 | 0
  BUN,Above, Month 24,Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 24,Below | 0 | 0 | 0 | 0
  BUN,Above, Month 24,Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 24,Normal | 2 | 0 | 1 | 0
  BUN,Above, Month 24,Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 24,Above | 0 | 0 | 0 | 1
  BUN,Above, Month 24,Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  BUN,Above, Month 24,Unknown | 0 | 0 | 0 | 0

33. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Creatine Phosphokinase (CPK) in Study Phase A
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CPK for subjects participating in Phase A of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  CPK,Unknown, Day 21,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 21,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Day 21,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 21,Normal | 1 | 0 | 0 | 1
  CPK,Unknown, Day 21,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 21,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Day 21,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 21,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Day 21, Below: number analyzed (Participants) | 47 | 16 | 48 | 17
  CPK,Normal, Day 21, Below | 0 | 0 | 0 | 0
  CPK,Normal, Day 21, Normal: number analyzed (Participants) | 47 | 16 | 48 | 17
  CPK,Normal, Day 21, Normal | 44 | 15 | 42 | 16
  CPK,Normal, Day 21, Above: number analyzed (Participants) | 47 | 16 | 48 | 17
  CPK,Normal, Day 21, Above | 2 | 0 | 2 | 1
  CPK,Normal, Day 21, Unknown: number analyzed (Participants) | 47 | 16 | 48 | 17
  CPK,Normal, Day 21, Unknown | 1 | 1 | 4 | 0
  CPK, Above, Day 21, Below: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK, Above, Day 21, Below | 0 | 0 | 0 | 0
  CPK, Above, Day 21, Normal: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK, Above, Day 21, Normal | 1 | 1 | 0 | 0
  CPK, Above, Day 21, Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK, Above, Day 21, Above | 0 | 0 | 0 | 0
  CPK, Above, Day 21, Unknown: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK, Above, Day 21, Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Day 42,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 42,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Day 42,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 42,Normal | 1 | 0 | 0 | 1
  CPK,Unknown, Day 42,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 42,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Day 42,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Day 42,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Day 42, Below: number analyzed (Participants) | 49 | 16 | 49 | 17
  CPK,Normal, Day 42, Below | 0 | 0 | 0 | 0
  CPK,Normal, Day 42, Normal: number analyzed (Participants) | 49 | 16 | 49 | 17
  CPK,Normal, Day 42, Normal | 46 | 14 | 42 | 14
  CPK,Normal, Day 42, Above: number analyzed (Participants) | 49 | 16 | 49 | 17
  CPK,Normal, Day 42, Above | 2 | 1 | 3 | 1
  CPK,Normal, Day 42, Unknown: number analyzed (Participants) | 49 | 16 | 49 | 17
  CPK,Normal, Day 42, Unknown | 1 | 1 | 4 | 2
  CPK, Above, Day 42, Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK, Above, Day 42, Below | 0 | 0 | 0 | 0
  CPK, Above, Day 42, Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK, Above, Day 42, Normal | 0 | 1 | 0 | 0
  CPK, Above, Day 42, Above | 0 | 0 | 1 | 0
  CPK, Above, Day 42, Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK, Above, Day 42, Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  CPK,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 6,Below: number analyzed (Participants) | 48 | 16 | 47 | 16
  CPK,Normal, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 6,Normal: number analyzed (Participants) | 48 | 16 | 47 | 16
  CPK,Normal, Month 6,Normal | 45 | 13 | 38 | 15
  CPK,Normal, Month 6,Above: number analyzed (Participants) | 48 | 16 | 47 | 16
  CPK,Normal, Month 6,Above | 2 | 1 | 5 | 1
  CPK,Normal, Month 6,Unknown: number analyzed (Participants) | 48 | 16 | 47 | 16
  CPK,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  CPK,Above, Month 6,Below: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 6,Normal: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above,Month 6,Normal | 1 | 1 | 0 | 0
  CPK,Above, Month 6,Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 6,Above | 0 | 0 | 0 | 0
  CPK,Above, Month 6,Unknown: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  CPK,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 12,Below: number analyzed (Participants) | 48 | 16 | 44 | 16
  CPK,Normal, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 12,Normal: number analyzed (Participants) | 48 | 16 | 44 | 16
  CPK,Normal, Month 12,Normal | 43 | 14 | 40 | 15
  CPK,Normal, Month 12,Above: number analyzed (Participants) | 48 | 16 | 44 | 16
  CPK,Normal, Month 12,Above | 2 | 2 | 2 | 1
  CPK,Normal, Month 12,Unknown: number analyzed (Participants) | 48 | 16 | 44 | 16
  CPK,Normal, Month 12,Unknown | 3 | 0 | 2 | 0
  CPK,Above, Month 12,Below: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Above, Month 12,Normal: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 12,Normal | 1 | 1 | 0 | 0
  CPK,Above, Month 12,Above: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 12,Above | 0 | 0 | 0 | 0
  CPK,Above, Month 12,Unknown: number analyzed (Participants) | 1 | 1 | 0 | 0
  CPK,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  CPK,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CPK,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 24,Below: number analyzed (Participants) | 45 | 15 | 41 | 13
  CPK,Normal, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 24,Normal: number analyzed (Participants) | 45 | 15 | 41 | 13
  CPK,Normal, Month 24,Normal | 45 | 14 | 36 | 12
  CPK,Normal, Month 24,Above: number analyzed (Participants) | 45 | 15 | 41 | 13
  CPK,Normal, Month 24,Above | 0 | 1 | 2 | 1
  CPK,Normal, Month 24,Unknown: number analyzed (Participants) | 45 | 15 | 41 | 13
  CPK,Normal, Month 24,Unknown | 0 | 0 | 3 | 0
  CPK,Above, Month 24,Below: number analyzed (Participants) | 1 | 1 | 1 | 0
  CPK,Above, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Above, Month 24,Normal: number analyzed (Participants) | 1 | 1 | 1 | 0
  CPK,Above, Month 24,Normal | 1 | 1 | 0 | 0
  CPK,Above, Month 24,Above: number analyzed (Participants) | 1 | 1 | 1 | 0
  CPK,Above, Month 24,Above | 0 | 0 | 1 | 0
  CPK,Above, Month 24,Unknown: number analyzed (Participants) | 1 | 1 | 1 | 0
  CPK,Above, Month 24,Unknown | 0 | 0 | 0 | 0

34. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Creatinine (CREA) in Study Phase A
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CREA for subjects participating in Phase A of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  CREA, Unknown, Day 21, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 21, Below | 0 | 0 | 0 | 0
  CREA, Unknown, Day 21, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 21, Normal | 1 | 0 | 0 | 1
  CREA, Unknown, Day 21, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 21, Above | 0 | 0 | 0 | 0
  CREA, Unknown, Day 21, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 21, Unknown | 0 | 0 | 0 | 0
  CREA, Normal, Day 21, Below: number analyzed (Participants) | 48 | 17 | 48 | 17
  CREA, Normal, Day 21, Below | 0 | 0 | 0 | 0
  CREA, Normal, Day 21, Normal: number analyzed (Participants) | 48 | 17 | 48 | 17
  CREA, Normal, Day 21, Normal | 47 | 16 | 42 | 17
  CREA, Normal, Day 21, Above: number analyzed (Participants) | 48 | 17 | 48 | 17
  CREA, Normal, Day 21, Above | 0 | 0 | 2 | 0
  CREA, Normal, Day 21, Unknown: number analyzed (Participants) | 48 | 17 | 48 | 17
  CREA, Normal, Day 21, Unknown | 1 | 1 | 4 | 0
  CREA, Unknown, Day 42, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 42, Below | 0 | 0 | 0 | 0
  CREA, Unknown, Day 42, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 42, Normal | 1 | 0 | 0 | 1
  CREA, Unknown, Day 42, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 42, Above | 0 | 0 | 0 | 0
  CREA, Unknown, Day 42, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA, Unknown, Day 42, Unknown | 0 | 0 | 0 | 0
  CREA, Normal, Day 42, Below: number analyzed (Participants) | 49 | 17 | 49 | 17
  CREA, Normal, Day 42, Below | 0 | 0 | 0 | 0
  CREA, Normal, Day 42, Normal: number analyzed (Participants) | 49 | 17 | 49 | 17
  CREA, Normal, Day 42, Normal | 48 | 16 | 43 | 15
  CREA, Normal, Day 42, Above: number analyzed (Participants) | 49 | 17 | 49 | 17
  CREA, Normal, Day 42, Above | 0 | 0 | 2 | 0
  CREA, Normal, Day 42, Unknown: number analyzed (Participants) | 49 | 17 | 49 | 17
  CREA, Normal, Day 42, Unknown | 1 | 1 | 4 | 2
  CREA,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  CREA,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 6,Below: number analyzed (Participants) | 49 | 17 | 47 | 16
  CREA,Normal, Month 6,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 6,Normal: number analyzed (Participants) | 49 | 17 | 47 | 16
  CREA,Normal, Month 6,Normal | 48 | 15 | 43 | 16
  CREA,Normal, Month 6,Above: number analyzed (Participants) | 49 | 17 | 47 | 16
  CREA,Normal, Month 6,Above | 0 | 0 | 0 | 0
  CREA,Normal, Month 6,Unknown: number analyzed (Participants) | 49 | 17 | 47 | 16
  CREA,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  CREA,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  CREA,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 12,Below: number analyzed (Participants) | 49 | 17 | 44 | 16
  CREA,Normal, Month 12,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 12,Normal: number analyzed (Participants) | 49 | 17 | 44 | 16
  CREA,Normal, Month 12,Normal | 46 | 17 | 42 | 16
  CREA,Normal, Month 12,Above: number analyzed (Participants) | 49 | 17 | 44 | 16
  CREA,Normal, Month 12,Above | 0 | 0 | 0 | 0
  CREA,Normal, Month 12,Unknown: number analyzed (Participants) | 49 | 17 | 44 | 16
  CREA,Normal, Month 12,Unknown | 3 | 0 | 2 | 0
  CREA,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  CREA,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  CREA,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 24,Below: number analyzed (Participants) | 46 | 16 | 42 | 13
  CREA,Normal, Month 24,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 24,Normal: number analyzed (Participants) | 46 | 16 | 42 | 13
  CREA,Normal, Month 24,Normal | 46 | 16 | 39 | 13
  CREA,Normal, Month 24,Above: number analyzed (Participants) | 46 | 16 | 42 | 13
  CREA,Normal, Month 24,Above | 0 | 0 | 1 | 0
  CREA,Normal, Month 24,Unknown: number analyzed (Participants) | 46 | 16 | 42 | 13
  CREA,Normal, Month 24,Unknown | 0 | 0 | 2 | 0

35. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Lactate Dehydrogenase (LDH) in Study Phase A
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for LDH for subjects participating in Phase A of the study
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 50 | 17 | 49 | 18
Participants
  LDH, Unknown, Day 21, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Unknown, Day 21, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 21, Normal | 1 | 0 | 0 | 1
  LDH, Unknown, Day 21, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 21, Above | 0 | 0 | 0 | 0
  LDH, Unknown, Day 21, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 21, Unknown | 0 | 0 | 0 | 0
  LDH, Normal, Day 21, Below: number analyzed (Participants) | 39 | 12 | 47 | 17
  LDH, Normal, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Normal, Day 21, Normal: number analyzed (Participants) | 39 | 12 | 47 | 17
  LDH, Normal, Day 21, Normal | 36 | 8 | 40 | 14
  LDH, Normal, Day 21, Above: number analyzed (Participants) | 39 | 12 | 47 | 17
  LDH, Normal, Day 21, Above | 2 | 3 | 3 | 2
  LDH, Normal, Day 21, Unknown: number analyzed (Participants) | 39 | 12 | 47 | 17
  LDH, Normal, Day 21, Unknown | 1 | 1 | 4 | 1
  LDH, Above, Day 21, Below: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Above, Day 21, Normal: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 21, Normal | 5 | 2 | 1 | 0
  LDH, Above, Day 21, Above: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 21, Above | 4 | 3 | 0 | 0
  LDH, Above, Day 21, Unknown: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 21, Unknown | 0 | 0 | 0 | 0
  LDH, Unknown, Day 42, Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 42, Below | 0 | 0 | 0 | 0
  LDH, Unknown, Day 42, Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 42, Normal | 1 | 0 | 0 | 1
  LDH, Unknown, Day 42, Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 42, Above | 0 | 0 | 0 | 0
  LDH, Unknown, Day 42, Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH, Unknown, Day 42, Unknown | 0 | 0 | 0 | 0
  LDH, Normal, Day 42, Above: number analyzed (Participants) | 40 | 12 | 48 | 17
  LDH, Normal, Day 42, Above | 7 | 4 | 4 | 1
  LDH, Normal, Day 42, Below: number analyzed (Participants) | 40 | 12 | 48 | 17
  LDH, Normal, Day 42, Below | 0 | 0 | 0 | 0
  LDH, Normal, Day 42, Normal: number analyzed (Participants) | 40 | 12 | 48 | 17
  LDH, Normal, Day 42, Normal | 32 | 6 | 41 | 14
  LDH, Normal, Day 42, Unknown: number analyzed (Participants) | 40 | 12 | 48 | 17
  LDH, Normal, Day 42, Unknown | 1 | 2 | 3 | 2
  LDH, Above, Day 42, Above: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 42, Above | 4 | 2 | 0 | 0
  LDH, Above, Day 42, Below: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 42, Below | 0 | 0 | 1 | 0
  LDH, Above, Day 42, Normal: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 42, Normal | 5 | 3 | 0 | 0
  LDH, Above, Day 42, Unknow: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH, Above, Day 42, Unknow | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 6,Normal | 1 | 0 | 0 | 1
  LDH,Unknown, Month 6,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 6,Below: number analyzed (Participants) | 40 | 12 | 46 | 16
  LDH,Normal, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 6,Normal: number analyzed (Participants) | 40 | 12 | 46 | 16
  LDH,Normal, Month 6,Normal | 31 | 7 | 38 | 13
  LDH,Normal, Month 6,Above: number analyzed (Participants) | 40 | 12 | 46 | 16
  LDH,Normal, Month 6,Above | 8 | 3 | 4 | 3
  LDH,Normal, Month 6,Unknown: number analyzed (Participants) | 40 | 12 | 46 | 16
  LDH,Normal, Month 6,Unknown | 1 | 2 | 4 | 0
  LDH,Above, Month 6,Below: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Above,Month 6,Normal: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above,Month 6,Normal | 5 | 4 | 1 | 0
  LDH,Above, Month 6,Above: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 6,Above | 4 | 1 | 0 | 0
  LDH,Above, Month 6,Unknown: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  LDH,Unknown, Month 12,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 12,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 12,Normal | 1 | 0 | 0 | 1
  LDH,Unknown, Month 12,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  LDH,Unknown, Month 12,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 12,Below: number analyzed (Participants) | 40 | 12 | 43 | 16
  LDH,Normal, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 12,Normal: number analyzed (Participants) | 40 | 12 | 43 | 16
  LDH,Normal, Month 12,Normal | 33 | 8 | 40 | 14
  LDH,Normal, Month 12,Above: number analyzed (Participants) | 40 | 12 | 43 | 16
  LDH,Normal, Month 12,Above | 4 | 4 | 1 | 2
  LDH,Normal, Month 12,Unknown: number analyzed (Participants) | 40 | 12 | 43 | 16
  LDH,Normal, Month 12,Unknown | 3 | 0 | 2 | 0
  LDH,Above, Month 12,Below: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Above, Month 12,Normal: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 12,Normal | 6 | 4 | 1 | 0
  LDH,Above, Month 12,Above: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 12,Above | 3 | 1 | 0 | 0
  LDH,Above, Month 12,Unknown: number analyzed (Participants) | 9 | 5 | 1 | 0
  LDH,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  LDH,Unknown, Month 24,Below: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 24,Normal | 1 | 0 | 0 | 1
  LDH,Unknown, Month 24,Above: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  LDH,Unknown, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 0 | 1
  LDH,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 24,Below: number analyzed (Participants) | 38 | 11 | 42 | 13
  LDH,Normal, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 24,Normal: number analyzed (Participants) | 38 | 11 | 42 | 13
  LDH,Normal, Month 24,Normal | 35 | 8 | 36 | 11
  LDH,Normal, Month 24,Above: number analyzed (Participants) | 38 | 11 | 42 | 13
  LDH,Normal, Month 24,Above | 3 | 3 | 3 | 2
  LDH,Normal, Month 24,Unknown: number analyzed (Participants) | 38 | 11 | 42 | 13
  LDH,Normal, Month 24,Unknown | 0 | 0 | 3 | 0
  LDH,Above, Month 24,Below: number analyzed (Participants) | 8 | 5 | 0 | 0
  LDH,Above, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Above, Month 24,Normal: number analyzed (Participants) | 8 | 5 | 0 | 0
  LDH,Above, Month 24,Normal | 6 | 5 | 0 | 0
  LDH,Above, Month 24,Above: number analyzed (Participants) | 8 | 5 | 0 | 0
  LDH,Above, Month 24,Above | 2 | 0 | 0 | 0
  LDH,Above, Month 24,Unknown: number analyzed (Participants) | 8 | 5 | 0 | 0
  LDH,Above, Month 24,Unknown | 0 | 0 | 0 | 0

36. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Alanine Aminotransferase (ALT) for Subjects in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for ALT for subjects participating in Phase B of the study.
Time Frame: At Days 21 and 42 and Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 49 | 16 | 46 | 16
Participants
  ALT,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 21,Normal | 0 | 0 | 1 | 0
  ALT,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 21,Above | 0 | 1 | 0 | 0
  ALT,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  ALT,Normal,Day 21,Below: number analyzed (Participants) | 48 | 16 | 45 | 16
  ALT,Normal,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Normal,Day 21,Normal: number analyzed (Participants) | 48 | 16 | 45 | 16
  ALT,Normal,Day 21,Normal | 44 | 16 | 44 | 16
  ALT,Normal,Day 21,Above: number analyzed (Participants) | 48 | 16 | 45 | 16
  ALT,Normal,Day 21,Above | 1 | 0 | 1 | 0
  ALT,Normal,Day 21,Unknown: number analyzed (Participants) | 48 | 16 | 45 | 16
  ALT,Normal,Day 21,Unknown | 3 | 0 | 0 | 0
  ALT,Above,Day 21,Below: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Above,Day 21,Normal: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 21,Normal | 0 | 0 | 0 | 1
  ALT,Above,Day 21,Above: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 21,Above | 0 | 0 | 0 | 0
  ALT,Above,Day 21,Unknown: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 21,Unknown | 0 | 0 | 0 | 0
  ALT,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 42,Normal | 0 | 1 | 1 | 0
  ALT,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  ALT,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  ALT,Normal,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Normal,Day 42,Normal | 46 | 16 | 44 | 16
  ALT,Normal,Day 42,Above | 1 | 0 | 2 | 0
  ALT,Normal,Day 42,Unknown | 2 | 0 | 0 | 0
  ALT,Above,Day 42,Below: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Above,Day 42,Normal: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 42,Normal | 0 | 0 | 0 | 0
  ALT,Above,Day 42,Above: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 42,Above | 0 | 0 | 0 | 1
  ALT,Above,Day 42,Unknown: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  ALT,Unknown,Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Month 6,Below | 0 | 0 | 0 | 0
  ALT,Unknown,Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Month 6,Normal | 0 | 1 | 1 | 0
  ALT,Unknown,Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Month 6,Above | 0 | 0 | 0 | 0
  ALT,Unknown,Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown,Month 6,Unknown | 0 | 0 | 0 | 0
  ALT,Normal,Month 6,Below: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal,Month 6,Below | 0 | 0 | 0 | 0
  ALT,Normal,Month 6,Normal: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal,Month 6,Normal | 48 | 16 | 44 | 16
  ALT,Normal,Month 6,Above: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal,Month 6,Above | 0 | 0 | 0 | 0
  ALT,Normal,Month 6,Unknown: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal,Month 6,Unknown | 1 | 0 | 0 | 0
  ALT,Above,Month 6,Below: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Month 6,Below | 0 | 0 | 0 | 0
  ALT,Above,Month 6,Normal: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Month 6,Normal | 0 | 0 | 0 | 1
  ALT,Above, Month 6,Above: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 6,Above | 0 | 0 | 0 | 0
  ALT,Above, Month 6,Unknown: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  ALT,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  ALT,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown, Month 12,Normal | 0 | 1 | 1 | 0
  ALT,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  ALT,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  ALT,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  ALT,Normal, Month 12,Below: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal, Month 12,Below | 0 | 0 | 0 | 0
  ALT,Normal, Month 12,Normal: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal, Month 12,Normal | 44 | 16 | 44 | 16
  ALT,Normal, Month 12,Above: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal, Month 12,Above | 0 | 0 | 0 | 0
  ALT,Normal, Month 12,Unknown: number analyzed (Participants) | 49 | 16 | 44 | 16
  ALT,Normal, Month 12,Unknown | 2 | 0 | 0 | 0
  ALT,Above, Month 12,Below: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 12,Below | 0 | 0 | 0 | 0
  ALT,Above,Month 12,Normal: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above,Month 12,Normal | 0 | 0 | 0 | 1
  ALT,Above, Month 12,Above: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 12,Above | 0 | 0 | 0 | 0
  ALT,Above, Month 12,Unknown: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  ALT,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  ALT,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT,Unknown, Month 24,Normal | 0 | 1 | 0 | 0
  ALT,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  ALT,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  ALT,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  ALT,Normal, Month 24,Below: number analyzed (Participants) | 45 | 16 | 44 | 16
  ALT,Normal, Month 24,Below | 0 | 0 | 0 | 0
  ALT,Normal, Month 24,Normal: number analyzed (Participants) | 45 | 16 | 44 | 16
  ALT,Normal, Month 24,Normal | 44 | 16 | 43 | 16
  ALT,Normal, Month 24,Above: number analyzed (Participants) | 45 | 16 | 44 | 16
  ALT,Normal, Month 24,Above | 1 | 0 | 1 | 0
  ALT,Normal, Month 24,Unknown: number analyzed (Participants) | 45 | 16 | 44 | 16
  ALT,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  ALT,Above, Month 24,Below: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 24,Below | 0 | 0 | 0 | 0
  ALT,Above, Month 24,Normal: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 24,Normal | 0 | 0 | 0 | 1
  ALT,Above, Month 24,Above: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 24,Above | 0 | 0 | 0 | 0
  ALT,Above, Month 24,Unknown: number analyzed (Participants) | 0 | 0 | 0 | 1
  ALT,Above, Month 24,Unknown | 0 | 0 | 0 | 0

37. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Aspartate Aminotransferase (AST) in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for AST for subjects participating in Phase B of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 47 | 15 | 43 | 16
Participants
  AST,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  AST,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 15 | 1 | 16
  AST,Unknown,Day 21,Normal | 0 | 0 | 1 | 0
  AST,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown,Day 21,Above | 0 | 1 | 0 | 0
  AST,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  AST,Normal,Day 21,Below: number analyzed (Participants) | 46 | 15 | 42 | 16
  AST,Normal,Day 21,Below | 0 | 0 | 0 | 0
  AST,Normal,Day 21,Normal: number analyzed (Participants) | 46 | 15 | 42 | 16
  AST,Normal,Day 21,Normal | 40 | 15 | 41 | 16
  AST,Normal,Day 21,Above: number analyzed (Participants) | 46 | 15 | 42 | 16
  AST,Normal,Day 21,Above | 3 | 0 | 1 | 0
  AST,Normal,Day 21,Unknown: number analyzed (Participants) | 46 | 15 | 42 | 16
  AST,Normal,Day 21,Unknown | 3 | 0 | 0 | 0
  AST,Above,Day 21,Below: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 21,Below | 0 | 0 | 0 | 0
  AST,Above,Day 21,Normal: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 21,Normal | 1 | 1 | 3 | 1
  AST,Above,Day 21,Above: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 21,Above | 0 | 0 | 0 | 0
  AST,Above,Day 21,Unknown: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 21,Unknown | 1 | 0 | 0 | 0
  AST,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  AST,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown,Day 42,Normal | 0 | 1 | 1 | 0
  AST,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  AST,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  AST,Normal,Day 42,Below | 0 | 0 | 0 | 0
  AST,Normal,Day 42,Normal | 40 | 13 | 40 | 16
  AST,Normal,Day 42,Above | 5 | 2 | 3 | 0
  AST,Normal,Day 42,Unknown | 2 | 0 | 0 | 0
  AST,Above,Day 42,Below: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 42,Below | 0 | 0 | 0 | 0
  AST,Above,Day 42,Normal: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 42,Normal | 2 | 1 | 3 | 0
  AST,Above,Day 42,Above: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 42,Above | 0 | 0 | 0 | 1
  AST,Above,Day 42,Unknown: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 6,Normal | 0 | 1 | 1 | 0
  AST,Unknown, Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  AST,Normal, Month 6,Below: number analyzed (Participants) | 47 | 15 | 41 | 16
  AST,Normal, Month 6,Below | 0 | 0 | 0 | 0
  AST,Normal, Month 6,Normal: number analyzed (Participants) | 47 | 15 | 41 | 16
  AST,Normal, Month 6,Normal | 45 | 14 | 40 | 16
  AST,Normal, Month 6,Above: number analyzed (Participants) | 47 | 15 | 41 | 16
  AST,Normal, Month 6,Above | 2 | 1 | 0 | 0
  AST,Normal, Month 6,Unknown: number analyzed (Participants) | 47 | 15 | 41 | 16
  AST,Normal, Month 6,Unknown | 0 | 0 | 1 | 0
  AST,Above, Month 6,Below: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above, Month 6,Below | 0 | 0 | 0 | 0
  AST,Above,Month 6,Normal: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above,Month 6,Normal | 2 | 1 | 3 | 1
  AST,Above, Month 6,Above: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above, Month 6,Above | 0 | 0 | 0 | 0
  AST,Above, Month 6,Unknown: number analyzed (Participants) | 2 | 1 | 3 | 1
  AST,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 12,Normal | 0 | 1 | 1 | 0
  AST,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  AST,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  AST,Normal, Month 12,Below: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 12,Below | 0 | 0 | 0 | 0
  AST,Normal, Month 12,Normal: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 12,Normal | 44 | 15 | 41 | 16
  AST,Normal, Month 12,Above: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 12,Above | 0 | 0 | 0 | 0
  AST,Normal, Month 12,Unknown: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 12,Unknown | 1 | 0 | 0 | 0
  AST,Above, Month 12,Below: number analyzed (Participants) | 1 | 1 | 3 | 1
  AST,Above, Month 12,Below | 0 | 0 | 0 | 0
  AST,Above,Month 12,Normal: number analyzed (Participants) | 1 | 1 | 3 | 1
  AST,Above,Month 12,Normal | 0 | 1 | 3 | 1
  AST,Above, Month 12,Above: number analyzed (Participants) | 1 | 1 | 3 | 1
  AST,Above, Month 12,Above | 0 | 0 | 0 | 0
  AST,Above, Month 12,Unknown: number analyzed (Participants) | 1 | 1 | 3 | 1
  AST,Above, Month 12,Unknown | 1 | 0 | 0 | 0
  AST,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  AST,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown, Month 24,Normal | 0 | 1 | 0 | 0
  AST,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  AST,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  AST,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  AST,Normal, Month 24,Below: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 24,Below | 0 | 0 | 0 | 0
  AST,Normal, Month 24,Normal: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 24,Normal | 44 | 15 | 41 | 16
  AST,Normal, Month 24,Above: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 24,Above | 1 | 0 | 0 | 0
  AST,Normal, Month 24,Unknown: number analyzed (Participants) | 45 | 15 | 41 | 16
  AST,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  AST,Above, Month 24,Below: number analyzed (Participants) | 0 | 1 | 3 | 1
  AST,Above, Month 24,Below | 0 | 0 | 0 | 0
  AST,Above, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 3 | 1
  AST,Above, Month 24,Normal | 0 | 1 | 2 | 1
  AST,Above, Month 24,Above: number analyzed (Participants) | 0 | 1 | 3 | 1
  AST,Above, Month 24,Above | 0 | 0 | 1 | 0
  AST,Above, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 3 | 1
  AST,Above, Month 24,Unknown | 0 | 0 | 0 | 0

38. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Urea Nitrogen (BUN) in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for BUN for subjects participating in Phase B of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 49 | 17 | 47 | 17
Participants
  BUN,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 21,Normal | 0 | 0 | 1 | 1
  BUN,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 21,Above | 0 | 1 | 0 | 0
  BUN,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Day 21,Below: number analyzed (Participants) | 44 | 14 | 40 | 13
  BUN,Normal,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Normal,Day 21,Normal: number analyzed (Participants) | 44 | 14 | 40 | 13
  BUN,Normal,Day 21,Normal | 35 | 13 | 37 | 12
  BUN,Normal,Day 21,Above: number analyzed (Participants) | 44 | 14 | 40 | 13
  BUN,Normal,Day 21,Above | 6 | 1 | 3 | 1
  BUN,Normal,Day 21,Unknown: number analyzed (Participants) | 44 | 14 | 40 | 13
  BUN,Normal,Day 21,Unknown | 3 | 0 | 0 | 0
  BUN,Above,Day 21,Below: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Above,Day 21,Normal: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 21,Normal | 3 | 1 | 5 | 2
  BUN,Above,Day 21,Above: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 21,Above | 1 | 1 | 0 | 1
  BUN,Above,Day 21,Unknown: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 21,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 42,Normal | 0 | 1 | 1 | 1
  BUN,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Day 42,Below: number analyzed (Participants) | 45 | 14 | 41 | 13
  BUN,Normal,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Normal,Day 42,Normal: number analyzed (Participants) | 45 | 14 | 41 | 13
  BUN,Normal,Day 42,Normal | 38 | 12 | 39 | 11
  BUN,Normal,Day 42,Above: number analyzed (Participants) | 45 | 14 | 41 | 13
  BUN,Normal,Day 42,Above | 6 | 2 | 2 | 2
  BUN,Normal,Day 42,Unknown: number analyzed (Participants) | 45 | 14 | 41 | 13
  BUN,Normal,Day 42,Unknown | 1 | 0 | 0 | 0
  BUN,Above,Day 42,Below: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Above,Day 42,Normal: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 42,Normal | 2 | 1 | 3 | 2
  BUN,Above,Day 42,Above: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 42,Above | 1 | 1 | 2 | 1
  BUN,Above,Day 42,Unknown: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Day 42,Unknown | 1 | 0 | 0 | 0
  BUN,Unknown, Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 6,Normal | 0 | 1 | 1 | 1
  BUN,Unknown, Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 6,Below: number analyzed (Participants) | 45 | 14 | 39 | 13
  BUN,Normal, Month 6,Below | 0 | 0 | 0 | 0
  BUN,Normal, Month 6,Normal: number analyzed (Participants) | 45 | 14 | 39 | 13
  BUN,Normal, Month 6,Normal | 42 | 12 | 39 | 13
  BUN,Normal, Month 6,Above: number analyzed (Participants) | 45 | 14 | 39 | 13
  BUN,Normal, Month 6,Above | 3 | 2 | 0 | 0
  BUN,Normal, Month 6,Unknown: number analyzed (Participants) | 45 | 14 | 39 | 13
  BUN,Normal, Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Above, Month 6,Below: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 6,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 6,Normal: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Month 6,Normal | 4 | 1 | 5 | 3
  BUN,Above, Month 6,Above: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 6,Above | 0 | 1 | 0 | 0
  BUN,Above, Month 6,Unknown: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 12,Normal | 0 | 1 | 1 | 1
  BUN,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 1
  BUN,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 12,Below: number analyzed (Participants) | 42 | 14 | 39 | 13
  BUN,Normal, Month 12,Below | 0 | 0 | 0 | 0
  BUN,Normal, Month 12,Normal: number analyzed (Participants) | 42 | 14 | 39 | 13
  BUN,Normal, Month 12,Normal | 36 | 12 | 38 | 11
  BUN,Normal, Month 12,Above: number analyzed (Participants) | 42 | 14 | 39 | 13
  BUN,Normal, Month 12,Above | 4 | 2 | 1 | 2
  BUN,Normal, Month 12,Unknown: number analyzed (Participants) | 42 | 14 | 39 | 13
  BUN,Normal, Month 12,Unknown | 2 | 0 | 0 | 0
  BUN,Above, Month 12,Below: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 12,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 12,Normal: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above,Month 12,Normal | 3 | 2 | 5 | 2
  BUN,Above, Month 12,Above: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 12,Above | 1 | 0 | 0 | 1
  BUN,Above, Month 12,Unknown: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 1
  BUN,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 1
  BUN,Unknown, Month 24,Normal | 0 | 1 | 0 | 1
  BUN,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 1
  BUN,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  BUN,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 1
  BUN,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  BUN,Normal, Month 24,Below: number analyzed (Participants) | 41 | 14 | 39 | 13
  BUN,Normal, Month 24,Below | 0 | 0 | 0 | 0
  BUN,Normal, Month 24,Normal: number analyzed (Participants) | 41 | 14 | 39 | 13
  BUN,Normal, Month 24,Normal | 36 | 11 | 39 | 13
  BUN,Normal, Month 24,Above: number analyzed (Participants) | 41 | 14 | 39 | 13
  BUN,Normal, Month 24,Above | 5 | 3 | 0 | 0
  BUN,Normal, Month 24,Unknown: number analyzed (Participants) | 41 | 14 | 39 | 13
  BUN,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  BUN,Above, Month 24,Below: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 24,Below | 0 | 0 | 0 | 0
  BUN,Above, Month 24,Normal: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 24,Normal | 4 | 1 | 2 | 2
  BUN,Above, Month 24,Above: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 24,Above | 0 | 1 | 3 | 1
  BUN,Above, Month 24,Unknown: number analyzed (Participants) | 4 | 2 | 5 | 3
  BUN,Above, Month 24,Unknown | 0 | 0 | 0 | 0

39. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Creatine Phosphokinase (CPK) in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CPK for subjects participating in Phase B of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 49 | 17 | 47 | 17
Participants
  CPK,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 21,Normal | 0 | 1 | 1 | 0
  CPK,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  CPK,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  CPK,Normal,Day 21,Below: number analyzed (Participants) | 46 | 16 | 43 | 16
  CPK,Normal,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Normal,Day 21,Normal: number analyzed (Participants) | 46 | 16 | 43 | 16
  CPK,Normal,Day 21,Normal | 46 | 16 | 43 | 16
  CPK,Normal,Day 21,Above: number analyzed (Participants) | 46 | 16 | 43 | 16
  CPK,Normal,Day 21,Above | 2 | 1 | 0 | 0
  CPK,Normal,Day 21,Unknown: number analyzed (Participants) | 46 | 16 | 43 | 16
  CPK,Normal,Day 21,Unknown | 2 | 0 | 0 | 0
  CPK,Above,Day 21,Below: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Above,Day 21,Normal: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 21,Normal | 0 | 0 | 1 | 0
  CPK,Above,Day 21,Above: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 21,Above | 1 | 0 | 1 | 1
  CPK,Above,Day 21,Unknown: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 21,Unknown | 1 | 0 | 0 | 1
  CPK,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 42,Normal | 0 | 1 | 1 | 0
  CPK,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  CPK,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  CPK,Normal,Day 42,Below: number analyzed (Participants) | 47 | 16 | 44 | 16
  CPK,Normal,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Normal,Day 42,Normal: number analyzed (Participants) | 47 | 16 | 44 | 16
  CPK,Normal,Day 42,Normal | 43 | 16 | 42 | 14
  CPK,Normal,Day 42,Above: number analyzed (Participants) | 47 | 16 | 44 | 16
  CPK,Normal,Day 42,Above | 2 | 2 | 2 | 0
  CPK,Normal,Day 42,Unknown: number analyzed (Participants) | 47 | 16 | 44 | 16
  CPK,Normal,Day 42,Unknown | 2 | 0 | 0 | 0
  CPK,Above,Day 42,Below: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Above,Day 42,Normal: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 42,Normal | 0 | 0 | 1 | 0
  CPK,Above,Day 42,Above: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 42,Above | 2 | 0 | 1 | 1
  CPK,Above,Day 42,Unknown: number analyzed (Participants) | 2 | 0 | 2 | 1
  CPK,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 6,Normal | 0 | 1 | 0 | 0
  CPK,Unknown, Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 6,Above | 0 | 0 | 1 | 0
  CPK,Unknown, Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 6,Below: number analyzed (Participants) | 47 | 16 | 43 | 16
  CPK,Normal, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 6,Normal: number analyzed (Participants) | 47 | 16 | 43 | 16
  CPK,Normal, Month 6,Normal | 46 | 13 | 42 | 15
  CPK,Normal, Month 6,Above: number analyzed (Participants) | 47 | 16 | 43 | 16
  CPK,Normal, Month 6,Above | 1 | 3 | 1 | 1
  CPK,Normal, Month 6,Unknown: number analyzed (Participants) | 47 | 16 | 43 | 16
  CPK,Normal, Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Above, Month 6,Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 6,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 6,Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above,Month 6,Normal | 1 | 0 | 1 | 0
  CPK,Above, Month 6,Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 6,Above | 1 | 0 | 0 | 1
  CPK,Above, Month 6,Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 12,Normal | 0 | 1 | 1 | 0
  CPK,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CPK,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 12,Below: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 12,Normal: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 12,Normal | 39 | 13 | 42 | 16
  CPK,Normal, Month 12,Above: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 12,Above | 4 | 3 | 1 | 0
  CPK,Normal, Month 12,Unknown: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 12,Unknown | 1 | 0 | 0 | 0
  CPK,Above, Month 12,Below: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 12,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 12,Normal: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above,Month 12,Normal | 0 | 0 | 1 | 1
  CPK,Above, Month 12,Above: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 12,Above | 1 | 0 | 0 | 0
  CPK,Above, Month 12,Unknown: number analyzed (Participants) | 2 | 0 | 1 | 1
  CPK,Above, Month 12,Unknown | 1 | 0 | 0 | 0
  CPK,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK,Unknown, Month 24,Normal | 0 | 1 | 0 | 0
  CPK,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  CPK,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  CPK,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  CPK,Normal, Month 24,Below: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Normal, Month 24,Normal: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 24,Normal | 43 | 14 | 41 | 16
  CPK,Normal, Month 24,Above: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 24,Above | 1 | 2 | 2 | 0
  CPK,Normal, Month 24,Unknown: number analyzed (Participants) | 44 | 16 | 43 | 16
  CPK,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  CPK,Above, Month 24,Below: number analyzed (Participants) | 1 | 0 | 1 | 1
  CPK,Above, Month 24,Below | 0 | 0 | 0 | 0
  CPK,Above, Month 24,Normal: number analyzed (Participants) | 1 | 0 | 1 | 1
  CPK,Above, Month 24,Normal | 1 | 0 | 1 | 0
  CPK,Above, Month 24,Above: number analyzed (Participants) | 1 | 0 | 1 | 1
  CPK,Above, Month 24,Above | 0 | 0 | 0 | 1
  CPK,Above, Month 24,Unknown: number analyzed (Participants) | 1 | 0 | 1 | 1
  CPK,Above, Month 24,Unknown | 0 | 0 | 0 | 0

40. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Creatinine (CREA) in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CREA for subjects participating in Phase B of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 49 | 17 | 46 | 17
Participants
  CREA,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 21,Normal | 0 | 1 | 1 | 0
  CREA,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  CREA,Normal,Day 21,Below: number analyzed (Participants) | 48 | 16 | 44 | 17
  CREA,Normal,Day 21,Below | 0 | 0 | 0 | 0
  CREA,Normal,Day 21,Normal: number analyzed (Participants) | 48 | 16 | 44 | 17
  CREA,Normal,Day 21,Normal | 44 | 16 | 43 | 17
  CREA,Normal,Day 21,Above: number analyzed (Participants) | 48 | 16 | 44 | 17
  CREA,Normal,Day 21,Above | 1 | 0 | 1 | 0
  CREA,Normal,Day 21,Unknown: number analyzed (Participants) | 48 | 16 | 44 | 17
  CREA,Normal,Day 21,Unknown | 3 | 0 | 0 | 0
  CREA,Above,Day 21,Below: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 21,Below | 0 | 0 | 0 | 0
  CREA,Above,Day 21,Normal: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 21,Normal | 0 | 0 | 1 | 0
  CREA,Above,Day 21,Above: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 21,Above | 0 | 0 | 0 | 0
  CREA,Above,Day 21,Unknow: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 21,Unknow | 0 | 0 | 0 | 0
  CREA,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 42,Normal | 0 | 1 | 1 | 0
  CREA,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  CREA,Normal,Day 42,Below: number analyzed (Participants) | 49 | 16 | 45 | 17
  CREA,Normal,Day 42,Below | 0 | 0 | 0 | 0
  CREA,Normal,Day 42,Normal: number analyzed (Participants) | 49 | 16 | 45 | 17
  CREA,Normal,Day 42,Normal | 46 | 16 | 45 | 17
  CREA,Normal,Day 42,Above: number analyzed (Participants) | 49 | 16 | 45 | 17
  CREA,Normal,Day 42,Above | 1 | 0 | 0 | 0
  CREA,Normal,Day 42,Unknown: number analyzed (Participants) | 49 | 16 | 45 | 17
  CREA,Normal,Day 42,Unknown | 2 | 0 | 0 | 0
  CREA,Above,Day 42,Below: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 42,Below | 0 | 0 | 0 | 0
  CREA,Above,Day 42,Normal: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 42,Normal | 0 | 0 | 1 | 0
  CREA,Above,Day 42,Above: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 42,Above | 0 | 0 | 0 | 0
  CREA,Above,Day 42,Unknown: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  CREA,Unknown, Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 6,Normal | 0 | 1 | 1 | 0
  CREA,Unknown, Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 6,Below: number analyzed (Participants) | 49 | 16 | 43 | 17
  CREA,Normal, Month 6,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 6,Normal: number analyzed (Participants) | 49 | 16 | 43 | 17
  CREA,Normal, Month 6,Normal | 49 | 16 | 42 | 17
  CREA,Normal, Month 6,Above: number analyzed (Participants) | 49 | 16 | 43 | 17
  CREA,Normal, Month 6,Above | 0 | 0 | 1 | 0
  CREA,Normal, Month 6,Unknown: number analyzed (Participants) | 49 | 16 | 43 | 17
  CREA,Normal, Month 6,Unknown | 0 | 0 | 0 | 0
  CREA,Above, Month 6,Below: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 6,Below | 0 | 0 | 0 | 0
  CREA,Above, Month 6,Normal: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 6,Normal | 0 | 0 | 0 | 0
  CREA,Above, Month 6,Above: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 6,Above | 0 | 0 | 1 | 0
  CREA,Above, Month 6,Unknown: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  CREA,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 12,Normal | 0 | 1 | 1 | 0
  CREA,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 12,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  CREA,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 12,Below: number analyzed (Participants) | 46 | 16 | 43 | 17
  CREA,Normal, Month 12,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 12,Normal: number analyzed (Participants) | 46 | 16 | 43 | 17
  CREA,Normal, Month 12,Normal | 44 | 16 | 42 | 17
  CREA,Normal, Month 12,Above: number analyzed (Participants) | 44 | 16 | 43 | 17
  CREA,Normal, Month 12,Above | 0 | 0 | 1 | 0
  CREA,Normal, Month 12,Unknown: number analyzed (Participants) | 44 | 16 | 43 | 17
  CREA,Normal, Month 12,Unknown | 2 | 0 | 0 | 0
  CREA,Above, Month 12,Below: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 12,Below | 0 | 0 | 0 | 0
  CREA,Above,Month 12,Normal: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above,Month 12,Normal | 0 | 0 | 1 | 0
  CREA,Above, Month 12,Above: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 12,Above | 0 | 0 | 0 | 0
  CREA,Above, Month 12,Unknown: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 12,Unknown | 0 | 0 | 0 | 0
  CREA,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  CREA,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  CREA,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  CREA,Unknown, Month 24,Normal | 0 | 1 | 0 | 0
  CREA,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  CREA,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  CREA,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  CREA,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  CREA,Normal, Month 24,Below: number analyzed (Participants) | 45 | 16 | 43 | 17
  CREA,Normal, Month 24,Below | 0 | 0 | 0 | 0
  CREA,Normal, Month 24,Normal: number analyzed (Participants) | 45 | 16 | 43 | 17
  CREA,Normal, Month 24,Normal | 45 | 16 | 43 | 17
  CREA,Normal, Month 24,Above: number analyzed (Participants) | 45 | 16 | 43 | 17
  CREA,Normal, Month 24,Above | 0 | 0 | 0 | 0
  CREA,Normal, Month 24,Unknown: number analyzed (Participants) | 45 | 16 | 43 | 17
  CREA,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  CREA,Above, Month 24,Below: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 24,Below | 0 | 0 | 0 | 0
  CREA,Above, Month 24,Normal: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 24,Normal | 0 | 0 | 1 | 0
  CREA,Above, Month 24,Above: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 24,Above | 0 | 0 | 0 | 0
  CREA,Above, Month 24,Unknown: number analyzed (Participants) | 0 | 0 | 1 | 0
  CREA,Above, Month 24,Unknown | 0 | 0 | 0 | 0

41. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Lactate Dehydrogenase (LDH) in Study Phase B
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for LDH for subjects participating in Phase B of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 49 | 17 | 47 | 17
Participants
  LDH,Unknown,Day 21,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Unknown,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 21,Normal | 0 | 0 | 1 | 0
  LDH,Unknown,Day 21,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 21,Above | 0 | 1 | 0 | 0
  LDH,Unknown,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 21,Unknown | 0 | 0 | 0 | 0
  LDH,Normal,Day 21,Below: number analyzed (Participants) | 43 | 14 | 38 | 15
  LDH,Normal,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Normal,Day 21,Normal: number analyzed (Participants) | 43 | 14 | 38 | 15
  LDH,Normal,Day 21,Normal | 33 | 13 | 38 | 15
  LDH,Normal,Day 21,Above: number analyzed (Participants) | 43 | 14 | 38 | 15
  LDH,Normal,Day 21,Above | 7 | 1 | 0 | 0
  LDH,Normal,Day 21,Unknown: number analyzed (Participants) | 43 | 14 | 38 | 15
  LDH,Normal,Day 21,Unknown | 3 | 0 | 0 | 0
  LDH,Above,Day 21,Below: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Above,Day 21,Normal: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 21,Normal | 2 | 1 | 3 | 1
  LDH,Above,Day 21,Above: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 21,Above | 2 | 1 | 4 | 1
  LDH,Above,Day 21,Unknown: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 21,Unknown | 1 | 0 | 0 | 0
  LDH,Unknown,Day 42,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Unknown,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 42,Normal | 0 | 0 | 1 | 0
  LDH,Unknown,Day 42,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 42,Above | 0 | 1 | 0 | 0
  LDH,Unknown,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  LDH,Normal,Day 42,Below: number analyzed (Participants) | 44 | 14 | 39 | 15
  LDH,Normal,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Normal,Day 42,Normal: number analyzed (Participants) | 44 | 14 | 39 | 15
  LDH,Normal,Day 42,Normal | 33 | 9 | 37 | 14
  LDH,Normal,Day 42,Above: number analyzed (Participants) | 44 | 14 | 39 | 15
  LDH,Normal,Day 42,Above | 9 | 5 | 2 | 1
  LDH,Normal,Day 42,Unknown: number analyzed (Participants) | 44 | 14 | 39 | 15
  LDH,Normal,Day 42,Unknown | 2 | 0 | 0 | 0
  LDH,Above,Day 42,Below: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Above,Day 42,Normal: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 42,Normal | 2 | 1 | 3 | 0
  LDH,Above,Day 42,Above: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 42,Above | 3 | 1 | 4 | 2
  LDH,Above,Day 42,Unknown: number analyzed (Participants) | 5 | 2 | 7 | 2
  LDH,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 6,Normal | 0 | 1 | 1 | 0
  LDH,Unknown, Month 6,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 6,Above | 0 | 0 | 0 | 0
  LDH,Unknown, Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 6,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 6,Below: number analyzed (Participants) | 44 | 14 | 38 | 15
  LDH,Normal, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 6,Normal: number analyzed (Participants) | 44 | 14 | 38 | 15
  LDH,Normal, Month 6,Normal | 37 | 9 | 34 | 14
  LDH,Normal, Month 6,Above: number analyzed (Participants) | 44 | 14 | 38 | 15
  LDH,Normal, Month 6,Above | 6 | 5 | 3 | 1
  LDH,Normal, Month 6,Unknown: number analyzed (Participants) | 44 | 14 | 38 | 15
  LDH,Normal, Month 6,Unknown | 1 | 0 | 1 | 0
  LDH,Above, Month 6,Below: number analyzed (Participants) | 5 | 2 | 6 | 2
  LDH,Above, Month 6,Below | 0 | 0 | 0 | 0
  LDH,Above,Month 6,Normal: number analyzed (Participants) | 5 | 2 | 6 | 2
  LDH,Above,Month 6,Normal | 3 | 2 | 2 | 1
  LDH,Above, Month 6,Above: number analyzed (Participants) | 5 | 2 | 6 | 2
  LDH,Above, Month 6,Above | 2 | 0 | 4 | 1
  LDH,Above, Month 6,Unknown: number analyzed (Participants) | 5 | 2 | 6 | 2
  LDH,Above, Month 6,Unknown | 0 | 0 | 0 | 0
  LDH,Unknown, Month 12,Below: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 12,Normal: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 12,Normal | 0 | 0 | 1 | 0
  LDH,Unknown, Month 12,Above: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 12,Above | 0 | 1 | 0 | 0
  LDH,Unknown, Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 1 | 0
  LDH,Unknown, Month 12,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 12,Below: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 12,Normal: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 12,Normal | 32 | 10 | 36 | 15
  LDH,Normal, Month 12,Above: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 12,Above | 9 | 4 | 2 | 0
  LDH,Normal, Month 12,Unknown: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 12,Unknown | 1 | 0 | 0 | 0
  LDH,Above, Month 12,Below: number analyzed (Participants) | 4 | 2 | 6 | 2
  LDH,Above, Month 12,Below | 0 | 0 | 0 | 0
  LDH,Above,Month 12,Normal: number analyzed (Participants) | 4 | 2 | 6 | 2
  LDH,Above,Month 12,Normal | 3 | 2 | 5 | 1
  LDH,Above, Month 12,Above: number analyzed (Participants) | 4 | 2 | 6 | 2
  LDH,Above, Month 12,Above | 0 | 0 | 1 | 1
  LDH,Above, Month 12,Unknown: number analyzed (Participants) | 4 | 2 | 6 | 2
  LDH,Above, Month 12,Unknown | 1 | 0 | 0 | 0
  LDH,Unknown, Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  LDH,Unknown, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Unknown, Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  LDH,Unknown, Month 24,Normal | 0 | 1 | 0 | 0
  LDH,Unknown, Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  LDH,Unknown, Month 24,Above | 0 | 0 | 0 | 0
  LDH,Unknown, Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  LDH,Unknown, Month 24,Unknown | 0 | 0 | 0 | 0
  LDH,Normal, Month 24,Below: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Normal, Month 24,Normal: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 24,Normal | 40 | 13 | 37 | 15
  LDH,Normal, Month 24,Above: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 24,Above | 2 | 1 | 1 | 0
  LDH,Normal, Month 24,Unknown: number analyzed (Participants) | 42 | 14 | 38 | 15
  LDH,Normal, Month 24,Unknown | 0 | 0 | 0 | 0
  LDH,Above, Month 24,Below: number analyzed (Participants) | 3 | 2 | 6 | 2
  LDH,Above, Month 24,Below | 0 | 0 | 0 | 0
  LDH,Above, Month 24,Normal: number analyzed (Participants) | 3 | 2 | 6 | 2
  LDH,Above, Month 24,Normal | 3 | 2 | 4 | 0
  LDH,Above, Month 24,Above: number analyzed (Participants) | 3 | 2 | 6 | 2
  LDH,Above, Month 24,Above | 0 | 0 | 2 | 2
  LDH,Above, Month 24,Unknown: number analyzed (Participants) | 3 | 2 | 6 | 2
  LDH,Above, Month 24,Unknown | 0 | 0 | 0 | 0

42. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Alanine Aminotransferase (ALT) for Subjects in Study Phase C
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for ALT for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  ALT, Unknown, Day 21, Below: number analyzed (Participants) | 5 | 1 | 2 | 1
  ALT, Unknown, Day 21, Below | 0 | 0 | 0 | 0
  ALT, Unknown, Day 21, Normal: number analyzed (Participants) | 5 | 1 | 2 | 1
  ALT, Unknown, Day 21, Normal | 3 | 0 | 1 | 1
  ALT, Unknown, Day 21, Above: number analyzed (Participants) | 5 | 1 | 2 | 1
  ALT, Unknown, Day 21, Above | 0 | 0 | 0 | 0
  ALT, Unknown, Day 21, Unknown: number analyzed (Participants) | 5 | 1 | 2 | 1
  ALT, Unknown, Day 21, Unknown | 2 | 1 | 1 | 0
  ALT, Normal, Day 21, Below: number analyzed (Participants) | 42 | 15 | 44 | 17
  ALT, Normal, Day 21, Below | 0 | 0 | 0 | 0
  ALT, Normal, Day 21, Normal: number analyzed (Participants) | 42 | 15 | 44 | 17
  ALT, Normal, Day 21, Normal | 41 | 12 | 40 | 17
  ALT, Normal, Day 21, Above: number analyzed (Participants) | 42 | 15 | 44 | 17
  ALT, Normal, Day 21, Above | 0 | 0 | 0 | 0
  ALT, Normal, Day 21, Unknown: number analyzed (Participants) | 42 | 15 | 44 | 17
  ALT, Normal, Day 21, Unknown | 1 | 3 | 4 | 0
  ALT, Above, Day 21, Below: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 21, Below | 0 | 0 | 0 | 0
  ALT, Above, Day 21, Normal: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 21, Normal | 0 | 0 | 1 | 0
  ALT, Above, Day 21, Above: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 21, Above | 1 | 0 | 0 | 0
  ALT, Above, Day 21, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 21, Unknown | 0 | 0 | 0 | 0
  ALT, Unknown, Day 42, Below: number analyzed (Participants) | 5 | 2 | 2 | 1
  ALT, Unknown, Day 42, Below | 0 | 0 | 0 | 0
  ALT, Unknown, Day 42, Normal: number analyzed (Participants) | 5 | 2 | 2 | 1
  ALT, Unknown, Day 42, Normal | 5 | 2 | 2 | 1
  ALT, Unknown, Day 42, Above: number analyzed (Participants) | 5 | 2 | 2 | 1
  ALT, Unknown, Day 42, Above | 0 | 0 | 0 | 0
  ALT, Unknown, Day 42, Unknown: number analyzed (Participants) | 5 | 2 | 2 | 1
  ALT, Unknown, Day 42, Unknown | 0 | 0 | 0 | 0
  ALT, Normal, Day 42, Below: number analyzed (Participants) | 42 | 15 | 45 | 17
  ALT, Normal, Day 42, Below | 0 | 0 | 0 | 0
  ALT, Normal, Day 42, Normal: number analyzed (Participants) | 42 | 15 | 45 | 17
  ALT, Normal, Day 42, Normal | 40 | 14 | 43 | 17
  ALT, Normal, Day 42, Above: number analyzed (Participants) | 42 | 15 | 45 | 17
  ALT, Normal, Day 42, Above | 0 | 0 | 0 | 0
  ALT, Normal, Day 42, Unknown: number analyzed (Participants) | 42 | 15 | 45 | 17
  ALT, Normal, Day 42, Unknown | 2 | 1 | 2 | 0
  ALT, Above, Day 42, Below: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 42, Below | 0 | 0 | 0 | 0
  ALT, Above, Day 42, Normal: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 42, Normal | 1 | 0 | 1 | 0
  ALT, Above, Day 42, Above: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 42, Above | 0 | 0 | 0 | 0
  ALT, Above, Day 42, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Day 42, Unknown | 0 | 0 | 0 | 0
  ALT, Unknown, Month 6, Below: number analyzed (Participants) | 4 | 2 | 2 | 1
  ALT, Unknown, Month 6, Below | 0 | 0 | 0 | 0
  ALT, Unknown, Month 6, Normal: number analyzed (Participants) | 4 | 2 | 2 | 1
  ALT, Unknown, Month 6, Normal | 4 | 2 | 2 | 1
  ALT, Unknown, Month 6, Above: number analyzed (Participants) | 4 | 2 | 2 | 1
  ALT, Unknown, Month 6, Above | 0 | 0 | 0 | 0
  ALT, Unknown, Month 6, Unknown: number analyzed (Participants) | 4 | 2 | 2 | 1
  ALT, Unknown, Month 6, Unknown | 0 | 0 | 0 | 0
  ALT, Normal , Month 6, Below: number analyzed (Participants) | 40 | 15 | 43 | 17
  ALT, Normal , Month 6, Below | 0 | 0 | 0 | 0
  ALT, Normal , Month 6, Normal: number analyzed (Participants) | 40 | 15 | 43 | 17
  ALT, Normal , Month 6, Normal | 36 | 13 | 41 | 17
  ALT, Normal , Month 6, Above: number analyzed (Participants) | 40 | 15 | 43 | 17
  ALT, Normal , Month 6, Above | 0 | 1 | 0 | 0
  ALT, Normal , Month 6, Unknown: number analyzed (Participants) | 40 | 15 | 43 | 17
  ALT, Normal , Month 6, Unknown | 4 | 1 | 2 | 0
  ALT, Above, Month 6, Below: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 6, Below | 0 | 0 | 0 | 0
  ALT, Above, Month 6, Normal: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 6, Normal | 1 | 0 | 1 | 0
  ALT, Above, Month 6, Above: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 6, Above | 0 | 0 | 0 | 0
  ALT, Above, Month 6, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 6, Unknown | 0 | 0 | 0 | 0
  ALT, Unknown, Month 12, Below: number analyzed (Participants) | 3 | 2 | 3 | 1
  ALT, Unknown, Month 12, Below | 0 | 0 | 0 | 0
  ALT, Unknown, Month 12, Normal: number analyzed (Participants) | 3 | 2 | 3 | 1
  ALT, Unknown, Month 12, Normal | 3 | 2 | 2 | 1
  ALT, Unknown, Month 12, Above: number analyzed (Participants) | 3 | 2 | 3 | 1
  ALT, Unknown, Month 12, Above | 0 | 0 | 1 | 0
  ALT, Unknown, Month 12, Unknown: number analyzed (Participants) | 3 | 2 | 3 | 1
  ALT, Unknown, Month 12, Unknown | 0 | 0 | 0 | 0
  ALT, Normal , Month 12, Below: number analyzed (Participants) | 40 | 15 | 44 | 17
  ALT, Normal , Month 12, Below | 0 | 0 | 0 | 0
  ALT, Normal , Month 12, Normal: number analyzed (Participants) | 40 | 15 | 44 | 17
  ALT, Normal , Month 12, Normal | 38 | 15 | 41 | 16
  ALT, Normal , Month 12, Above: number analyzed (Participants) | 40 | 15 | 44 | 17
  ALT, Normal , Month 12, Above | 0 | 0 | 1 | 0
  ALT, Normal , Month 12, Unknown: number analyzed (Participants) | 40 | 15 | 44 | 17
  ALT, Normal , Month 12, Unknown | 2 | 0 | 2 | 1
  ALT, Above, Month 12, Below: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 12, Below | 0 | 0 | 0 | 0
  ALT, Above, Month 12, Normal: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 12, Normal | 1 | 0 | 1 | 0
  ALT, Above, Month 12, Above: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 12, Above | 0 | 0 | 0 | 0
  ALT, Above, Month 12, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 12, Unknown | 0 | 0 | 0 | 0
  ALT, Unknown, Month 24, Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  ALT, Unknown, Month 24, Below | 0 | 0 | 0 | 0
  ALT, Unknown, Month 24, Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  ALT, Unknown, Month 24, Normal | 2 | 2 | 2 | 1
  ALT, Unknown, Month 24, Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  ALT, Unknown, Month 24, Above | 0 | 0 | 0 | 0
  ALT, Unknown, Month 24, Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  ALT, Unknown, Month 24, Unknown | 1 | 0 | 0 | 0
  ALT, Normal , Month 24, Below: number analyzed (Participants) | 38 | 15 | 43 | 17
  ALT, Normal , Month 24, Below | 0 | 0 | 0 | 0
  ALT, Normal , Month 24, Normal: number analyzed (Participants) | 38 | 15 | 43 | 17
  ALT, Normal , Month 24, Normal | 36 | 15 | 41 | 17
  ALT, Normal , Month 24, Above: number analyzed (Participants) | 38 | 15 | 43 | 17
  ALT, Normal , Month 24, Above | 2 | 0 | 2 | 0
  ALT, Normal , Month 24, Unknown: number analyzed (Participants) | 38 | 15 | 43 | 17
  ALT, Normal , Month 24, Unknown | 0 | 0 | 0 | 0
  ALT, Above, Month 24, Below: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 24, Below | 0 | 0 | 0 | 0
  ALT, Above, Month 24, Normal: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 24, Normal | 1 | 0 | 1 | 0
  ALT, Above, Month 24, Above: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 24, Above | 0 | 0 | 0 | 0
  ALT, Above, Month 24, Unknown: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT, Above, Month 24, Unknown | 0 | 0 | 0 | 0

43. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Aspartate Aminotransferase (AST) in Study Phase C
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for AST for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  AST, Unknown, Day 21, Below: number analyzed (Participants) | 5 | 1 | 2 | 1
  AST, Unknown, Day 21, Below | 0 | 0 | 0 | 0
  AST, Unknown, Day 21, Normal: number analyzed (Participants) | 5 | 1 | 2 | 1
  AST, Unknown, Day 21, Normal | 3 | 0 | 1 | 1
  AST, Unknown, Day 21, Above: number analyzed (Participants) | 5 | 1 | 2 | 1
  AST, Unknown, Day 21, Above | 0 | 0 | 0 | 0
  AST, Unknown, Day 21, Unknown: number analyzed (Participants) | 5 | 1 | 2 | 1
  AST, Unknown, Day 21, Unknown | 2 | 1 | 1 | 0
  AST, Normal, Day 21, Below: number analyzed (Participants) | 40 | 12 | 44 | 17
  AST, Normal, Day 21, Below | 0 | 0 | 0 | 0
  AST, Normal, Day 21, Normal: number analyzed (Participants) | 40 | 12 | 44 | 17
  AST, Normal, Day 21, Normal | 39 | 10 | 40 | 17
  AST, Normal, Day 21, Above: number analyzed (Participants) | 40 | 12 | 44 | 17
  AST, Normal, Day 21, Above | 0 | 0 | 0 | 0
  AST, Normal, Day 21, Unknown: number analyzed (Participants) | 40 | 12 | 44 | 17
  AST, Normal, Day 21, Unknown | 1 | 2 | 4 | 0
  AST, Above, Day 21, Below: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 21, Below | 0 | 0 | 0 | 0
  AST, Above, Day 21, Normal: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 21, Normal | 2 | 2 | 1 | 0
  AST, Above, Day 21, Above: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 21, Above | 1 | 0 | 0 | 0
  AST, Above, Day 21, Unknown: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 21, Unknown | 0 | 1 | 0 | 0
  AST, Unknown, Day 42, Below: number analyzed (Participants) | 5 | 2 | 2 | 1
  AST, Unknown, Day 42, Below | 0 | 0 | 0 | 0
  AST, Unknown, Day 42, Normal: number analyzed (Participants) | 5 | 2 | 2 | 1
  AST, Unknown, Day 42, Normal | 5 | 2 | 1 | 1
  AST, Unknown, Day 42, Above: number analyzed (Participants) | 5 | 2 | 2 | 1
  AST, Unknown, Day 42, Above | 0 | 0 | 1 | 0
  AST, Unknown, Day 42, Unknown: number analyzed (Participants) | 5 | 2 | 2 | 1
  AST, Unknown, Day 42, Unknown | 0 | 0 | 0 | 0
  AST, Normal, Day 42, Below: number analyzed (Participants) | 40 | 12 | 45 | 17
  AST, Normal, Day 42, Below | 0 | 0 | 0 | 0
  AST, Normal, Day 42, Normal: number analyzed (Participants) | 40 | 12 | 45 | 17
  AST, Normal, Day 42, Normal | 36 | 11 | 41 | 17
  AST, Normal, Day 42, Above: number analyzed (Participants) | 40 | 12 | 45 | 17
  AST, Normal, Day 42, Above | 2 | 0 | 2 | 0
  AST, Normal, Day 42, Unknown: number analyzed (Participants) | 40 | 12 | 45 | 17
  AST, Normal, Day 42, Unknown | 2 | 1 | 2 | 0
  AST, Above, Day 42, Below: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 42, Below | 0 | 0 | 0 | 0
  AST, Above, Day 42, Normal: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 42, Normal | 3 | 1 | 1 | 0
  AST, Above, Day 42, Above: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 42, Above | 0 | 2 | 0 | 0
  AST, Above, Day 42, Unknown: number analyzed (Participants) | 3 | 3 | 1 | 0
  AST, Above, Day 42, Unknown | 0 | 0 | 0 | 0
  AST, Unknown, Month 6, Below: number analyzed (Participants) | 4 | 2 | 2 | 1
  AST, Unknown, Month 6, Below | 0 | 0 | 0 | 0
  AST, Unknown, Month 6, Normal: number analyzed (Participants) | 4 | 2 | 2 | 1
  AST, Unknown, Month 6, Normal | 3 | 2 | 2 | 1
  AST, Unknown, Month 6, Above: number analyzed (Participants) | 4 | 2 | 2 | 1
  AST, Unknown, Month 6, Above | 0 | 0 | 0 | 0
  AST, Unknown, Month 6, Unknown: number analyzed (Participants) | 4 | 2 | 2 | 1
  AST, Unknown, Month 6, Unknown | 1 | 0 | 0 | 0
  AST, Normal, Month 6, Below: number analyzed (Participants) | 39 | 12 | 43 | 17
  AST, Normal, Month 6, Below | 0 | 0 | 0 | 0
  AST, Normal, Month 6, Normal: number analyzed (Participants) | 39 | 12 | 43 | 17
  AST, Normal, Month 6, Normal | 34 | 9 | 40 | 17
  AST, Normal, Month 6, Above: number analyzed (Participants) | 39 | 12 | 43 | 17
  AST, Normal, Month 6, Above | 1 | 2 | 1 | 0
  AST, Normal, Month 6, Unknown: number analyzed (Participants) | 39 | 12 | 43 | 17
  AST, Normal, Month 6, Unknown | 4 | 1 | 2 | 0
  AST, Above, Month 6, Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 6, Below | 0 | 0 | 0 | 0
  AST, Above, Month 6, Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 6, Normal | 2 | 3 | 1 | 0
  AST, Above, Month 6, Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 6, Above | 0 | 0 | 0 | 0
  AST, Above, Month 6, Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 6, Unknown | 0 | 0 | 0 | 0
  AST, Unknown, Month 12, Below: number analyzed (Participants) | 3 | 2 | 3 | 1
  AST, Unknown, Month 12, Below | 0 | 0 | 0 | 0
  AST, Unknown, Month 12, Normal: number analyzed (Participants) | 3 | 2 | 3 | 1
  AST, Unknown, Month 12, Normal | 3 | 2 | 2 | 1
  AST, Unknown, Month 12, Above: number analyzed (Participants) | 3 | 2 | 3 | 1
  AST, Unknown, Month 12, Above | 0 | 0 | 1 | 0
  AST, Unknown, Month 12, Unknown: number analyzed (Participants) | 3 | 2 | 3 | 1
  AST, Unknown, Month 12, Unknown | 0 | 0 | 0 | 0
  AST, Normal, Month 12, Below: number analyzed (Participants) | 39 | 12 | 44 | 17
  AST, Normal, Month 12, Below | 0 | 0 | 0 | 0
  AST, Normal, Month 12, Normal: number analyzed (Participants) | 39 | 12 | 44 | 17
  AST, Normal, Month 12, Normal | 36 | 12 | 37 | 16
  AST, Normal, Month 12, Above: number analyzed (Participants) | 39 | 12 | 44 | 17
  AST, Normal, Month 12, Above | 0 | 0 | 4 | 0
  AST, Normal, Month 12, Unknown: number analyzed (Participants) | 39 | 12 | 44 | 17
  AST, Normal, Month 12, Unknown | 3 | 0 | 3 | 1
  AST, Above, Month 12, Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 12, Below | 0 | 0 | 0 | 0
  AST, Above, Month 12, Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 12, Normal | 2 | 3 | 1 | 0
  AST, Above, Month 12, Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 12, Above | 0 | 0 | 0 | 0
  AST, Above, Month 12, Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 12, Unknown | 0 | 0 | 0 | 0
  AST, Unknown, Month 24, Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  AST, Unknown, Month 24, Below | 0 | 0 | 0 | 0
  AST, Unknown, Month 24, Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  AST, Unknown, Month 24, Normal | 2 | 2 | 2 | 1
  AST, Unknown, Month 24, Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  AST, Unknown, Month 24, Above | 0 | 0 | 0 | 0
  AST, Unknown, Month 24, Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  AST, Unknown, Month 24, Unknown | 1 | 0 | 0 | 0
  AST, Normal, Month 24, Below: number analyzed (Participants) | 37 | 12 | 43 | 17
  AST, Normal, Month 24, Below | 0 | 0 | 0 | 0
  AST, Normal, Month 24, Normal: number analyzed (Participants) | 37 | 12 | 43 | 17
  AST, Normal, Month 24, Normal | 34 | 12 | 42 | 17
  AST, Normal, Month 24, Above: number analyzed (Participants) | 37 | 12 | 43 | 17
  AST, Normal, Month 24, Above | 3 | 0 | 1 | 0
  AST, Normal, Month 24, Unknown: number analyzed (Participants) | 37 | 12 | 43 | 17
  AST, Normal, Month 24, Unknown | 0 | 0 | 0 | 0
  AST, Above, Month 24, Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 24, Below | 0 | 0 | 0 | 0
  AST, Above, Month 24, Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 24, Normal | 2 | 3 | 1 | 0
  AST, Above, Month 24, Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 24, Above | 0 | 0 | 0 | 0
  AST, Above, Month 24, Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  AST, Above, Month 24, Unknown | 0 | 0 | 0 | 0

44. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Urea Nitrogen (BUN) in Study Phase C
Description: Changes from baseline are categorised as below, within(normal), or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for BUN for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  BUN,Unknown,Day 21,Below: number analyzed (Participants) | 5 | 1 | 1 | 1
  BUN,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Day 21,Normal: number analyzed (Participants) | 5 | 1 | 1 | 1
  BUN,Unknown,Day 21,Normal | 3 | 0 | 0 | 1
  BUN,Unknown,Day 21,Above: number analyzed (Participants) | 5 | 1 | 1 | 1
  BUN,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  BUN,Unknown,Day 21,Unknown: number analyzed (Participants) | 5 | 1 | 1 | 1
  BUN,Unknown,Day 21,Unknown | 2 | 1 | 1 | 0
  BUN,Below,Day 21,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Below,Day 21,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 21,Normal | 0 | 0 | 0 | 0
  BUN,Below,Day 21,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 21,Above | 0 | 0 | 0 | 0
  BUN,Below,Day 21,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 21,Unknown | 0 | 1 | 0 | 0
  BUN,Normal,Day 21,Below: number analyzed (Participants) | 41 | 11 | 45 | 17
  BUN,Normal,Day 21,Below | 1 | 0 | 0 | 0
  BUN,Normal,Day 21,Normal: number analyzed (Participants) | 41 | 11 | 45 | 17
  BUN,Normal,Day 21,Normal | 37 | 9 | 41 | 16
  BUN,Normal,Day 21,Above: number analyzed (Participants) | 41 | 11 | 45 | 17
  BUN,Normal,Day 21,Above | 2 | 0 | 0 | 1
  BUN,Normal,Day 21,Unknown: number analyzed (Participants) | 41 | 11 | 45 | 17
  BUN,Normal,Day 21,Unknown | 1 | 2 | 4 | 0
  BUN,Above,Day 21,Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 21,Below | 0 | 0 | 0 | 0
  BUN,Above,Day 21,Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 21,Normal | 2 | 3 | 1 | 0
  BUN,Above,Day 21,Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 21,Above | 0 | 0 | 0 | 0
  BUN,Above,Day 21,Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 21,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Below: number analyzed (Participants) | 5 | 2 | 1 | 1
  BUN,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Normal: number analyzed (Participants) | 5 | 2 | 1 | 1
  BUN,Unknown,Day 42,Normal | 5 | 2 | 1 | 1
  BUN,Unknown,Day 42,Above: number analyzed (Participants) | 5 | 2 | 1 | 1
  BUN,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  BUN,Unknown,Day 42,Unknown: number analyzed (Participants) | 5 | 2 | 1 | 1
  BUN,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  BUN,Below,Day 42,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Below,Day 42,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 42,Normal | 0 | 1 | 0 | 0
  BUN,Below,Day 42,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 42,Above | 0 | 0 | 0 | 0
  BUN,Below,Day 42,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Day 42,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Day 42,Below: number analyzed (Participants) | 41 | 11 | 46 | 17
  BUN,Normal,Day 42,Below | 0 | 0 | 3 | 0
  BUN,Normal,Day 42,Normal: number analyzed (Participants) | 41 | 11 | 46 | 17
  BUN,Normal,Day 42,Normal | 37 | 11 | 38 | 16
  BUN,Normal,Day 42, Above: number analyzed (Participants) | 41 | 11 | 46 | 17
  BUN,Normal,Day 42, Above | 2 | 0 | 3 | 1
  BUN,Normal,Day 42,Unknown: number analyzed (Participants) | 41 | 11 | 46 | 17
  BUN,Normal,Day 42,Unknown | 2 | 0 | 2 | 0
  BUN,Above,Day 42,Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 42,Below | 0 | 0 | 0 | 0
  BUN,Above,Day 42,Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 42,Normal | 1 | 2 | 1 | 0
  BUN,Above,Day 42,Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 42,Above | 1 | 0 | 0 | 0
  BUN,Above,Day 42,Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Day 42,Unknown | 0 | 1 | 0 | 0
  BUN,Unknown,Month 6,Below: number analyzed (Participants) | 4 | 2 | 1 | 1
  BUN,Unknown,Month 6,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Month 6,Normal: number analyzed (Participants) | 4 | 2 | 1 | 1
  BUN,Unknown,Month 6,Normal | 4 | 2 | 1 | 1
  BUN,Unknown,Month 6,Above: number analyzed (Participants) | 4 | 2 | 1 | 1
  BUN,Unknown,Month 6,Above | 0 | 0 | 0 | 0
  BUN,Unknown,Month 6,Unknown: number analyzed (Participants) | 4 | 2 | 1 | 1
  BUN,Unknown,Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Below,Month 6,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 6,Below | 0 | 0 | 0 | 0
  BUN,Below,Month 6,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 6,Normal | 0 | 1 | 0 | 0
  BUN,Below,Month 6,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 6,Above | 0 | 0 | 0 | 0
  BUN,Below,Month 6,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Month 6,Below: number analyzed (Participants) | 39 | 11 | 44 | 17
  BUN,Normal,Month 6,Below | 0 | 0 | 2 | 0
  BUN,Normal,Month 6,Normal: number analyzed (Participants) | 39 | 11 | 44 | 17
  BUN,Normal,Month 6,Normal | 34 | 10 | 35 | 17
  BUN,Normal,Month 6,Above: number analyzed (Participants) | 39 | 11 | 44 | 17
  BUN,Normal,Month 6,Above | 1 | 0 | 5 | 0
  BUN,Normal,Month 6,Unknown: number analyzed (Participants) | 39 | 11 | 44 | 17
  BUN,Normal,Month 6,Unknown | 4 | 1 | 2 | 0
  BUN,Above,Month 6,Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 6,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 6,Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 6,Normal | 2 | 2 | 0 | 0
  BUN,Above,Month 6,Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 6,Above | 0 | 1 | 1 | 0
  BUN,Above,Month 6,Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 6,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown,Month 12,Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  BUN,Unknown,Month 12,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Month 12,Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  BUN,Unknown,Month 12,Normal | 3 | 2 | 1 | 1
  BUN,Unknown,Month 12,Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  BUN,Unknown,Month 12,Above | 0 | 0 | 1 | 0
  BUN,Unknown,Month 12,Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  BUN,Unknown,Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Below,Month 12,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 12,Below | 0 | 0 | 0 | 0
  BUN,Below,Month 12,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 12,Normal | 0 | 1 | 0 | 0
  BUN,Below,Month 12,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 12,Above | 0 | 0 | 0 | 0
  BUN,Below,Month 12,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Month12,Below: number analyzed (Participants) | 39 | 11 | 45 | 17
  BUN,Normal,Month12,Below | 0 | 0 | 0 | 0
  BUN,Normal,Month12,Normal: number analyzed (Participants) | 39 | 11 | 45 | 17
  BUN,Normal,Month12,Normal | 36 | 10 | 41 | 16
  BUN,Normal,Month12,Above: number analyzed (Participants) | 39 | 11 | 45 | 17
  BUN,Normal,Month12,Above | 1 | 1 | 2 | 0
  BUN,Normal,Month12,Unknown: number analyzed (Participants) | 39 | 11 | 45 | 17
  BUN,Normal,Month12,Unknown | 2 | 0 | 2 | 1
  BUN,Above,Month 12,Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 12,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 12,Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 12,Normal | 2 | 2 | 1 | 0
  BUN,Above,Month 12,Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 12,Above | 0 | 1 | 0 | 0
  BUN,Above,Month 12,Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 12,Unknown | 0 | 0 | 0 | 0
  BUN,Unknown,Month 24,Below: number analyzed (Participants) | 3 | 2 | 1 | 1
  BUN,Unknown,Month 24,Below | 0 | 0 | 0 | 0
  BUN,Unknown,Month 24,Normal: number analyzed (Participants) | 3 | 2 | 1 | 1
  BUN,Unknown,Month 24,Normal | 2 | 2 | 1 | 1
  BUN,Unknown,Month 24,Above: number analyzed (Participants) | 3 | 2 | 1 | 1
  BUN,Unknown,Month 24,Above | 0 | 0 | 0 | 0
  BUN,Unknown,Month 24,Unknown: number analyzed (Participants) | 3 | 2 | 1 | 1
  BUN,Unknown,Month 24,Unknown | 1 | 0 | 0 | 0
  BUN,Below,Month 24,Below: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 24,Below | 0 | 0 | 0 | 0
  BUN,Below,Month 24,Normal: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 24,Normal | 0 | 1 | 0 | 0
  BUN,Below,Month 24,Above: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 24,Above | 0 | 0 | 0 | 0
  BUN,Below,Month 24,Unknown: number analyzed (Participants) | 0 | 1 | 0 | 0
  BUN,Below,Month 24,Unknown | 0 | 0 | 0 | 0
  BUN,Normal,Month 24,Below: number analyzed (Participants) | 37 | 11 | 44 | 17
  BUN,Normal,Month 24,Below | 0 | 0 | 1 | 0
  BUN,Normal,Month 24,Normal: number analyzed (Participants) | 37 | 11 | 44 | 17
  BUN,Normal,Month 24,Normal | 35 | 9 | 39 | 16
  BUN,Normal,Month 24,Above: number analyzed (Participants) | 37 | 11 | 44 | 17
  BUN,Normal,Month 24,Above | 2 | 2 | 4 | 1
  BUN,Normal,Month 24,Unknown: number analyzed (Participants) | 37 | 11 | 44 | 17
  BUN,Normal,Month 24,Unknown | 0 | 0 | 0 | 0
  BUN,Above,Month 24,Below: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 24,Below | 0 | 0 | 0 | 0
  BUN,Above,Month 24,Normal: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 24,Normal | 2 | 3 | 0 | 0
  BUN,Above,Month 24,Above: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 24,Above | 0 | 0 | 1 | 0
  BUN,Above,Month 24,Unknown: number analyzed (Participants) | 2 | 3 | 1 | 0
  BUN,Above,Month 24,Unknown | 0 | 0 | 0 | 0

45. Primary Outcome: Number of Subjects With Changed Status as Regards to the Biochemical Parameter Blood Creatinine (CREA) in Study Phase C
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CREA for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  CREA,Unknown,Day 21,Below: number analyzed (Participants) | 5 | 1 | 2 | 1
  CREA,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Day 21,Normal: number analyzed (Participants) | 5 | 1 | 2 | 1
  CREA,Unknown,Day 21,Normal | 3 | 0 | 1 | 1
  CREA,Unknown,Day 21,Above: number analyzed (Participants) | 5 | 1 | 2 | 1
  CREA,Unknown,Day 21,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Day 21,Unknown: number analyzed (Participants) | 5 | 1 | 2 | 1
  CREA,Unknown,Day 21,Unknown | 2 | 1 | 1 | 0
  CREA,Normal,Day 21,Below: number analyzed (Participants) | 43 | 15 | 45 | 17
  CREA,Normal,Day 21,Below | 0 | 0 | 0 | 0
  CREA,Normal,Day 21,Normal: number analyzed (Participants) | 43 | 15 | 45 | 17
  CREA,Normal,Day 21,Normal | 42 | 12 | 41 | 17
  CREA,Normal,Day 21,Above: number analyzed (Participants) | 43 | 15 | 45 | 17
  CREA,Normal,Day 21,Above | 0 | 0 | 0 | 0
  CREA,Normal,Day 21,Unknown: number analyzed (Participants) | 43 | 15 | 45 | 17
  CREA,Normal,Day 21,Unknown | 1 | 3 | 4 | 0
  CREA,Unknown,Day 42,Below: number analyzed (Participants) | 5 | 2 | 2 | 1
  CREA,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Day 42,Normal: number analyzed (Participants) | 5 | 2 | 2 | 1
  CREA,Unknown,Day 42,Normal | 5 | 2 | 2 | 1
  CREA,Unknown,Day 42,Above: number analyzed (Participants) | 5 | 2 | 2 | 1
  CREA,Unknown,Day 42,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Day 42,Unknown: number analyzed (Participants) | 5 | 2 | 2 | 1
  CREA,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  CREA,Normal,Day 42,Below: number analyzed (Participants) | 43 | 15 | 46 | 17
  CREA,Normal,Day 42,Below | 0 | 0 | 0 | 0
  CREA,Normal,Day 42,Normal: number analyzed (Participants) | 43 | 15 | 46 | 17
  CREA,Normal,Day 42,Normal | 41 | 14 | 44 | 17
  CREA,Normal,Day 42,Above: number analyzed (Participants) | 43 | 15 | 46 | 17
  CREA,Normal,Day 42,Above | 0 | 0 | 0 | 0
  CREA,Normal,Day 42,Unknown: number analyzed (Participants) | 43 | 15 | 46 | 17
  CREA,Normal,Day 42,Unknown | 2 | 1 | 2 | 0
  CREA,Unknown,Month 6,Below: number analyzed (Participants) | 4 | 2 | 2 | 1
  CREA,Unknown,Month 6,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Month 6,Normal: number analyzed (Participants) | 4 | 2 | 2 | 1
  CREA,Unknown,Month 6,Normal | 4 | 2 | 2 | 1
  CREA,Unknown,Month 6,Above: number analyzed (Participants) | 4 | 2 | 2 | 1
  CREA,Unknown,Month 6,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Month 6,Unknown: number analyzed (Participants) | 4 | 2 | 2 | 1
  CREA,Unknown,Month 6,Unknown | 0 | 0 | 0 | 0
  CREA,Normal,Month 6,Below: number analyzed (Participants) | 41 | 15 | 44 | 17
  CREA,Normal,Month 6,Below | 0 | 0 | 0 | 0
  CREA,Normal,Month 6,Normal: number analyzed (Participants) | 41 | 15 | 44 | 17
  CREA,Normal,Month 6,Normal | 37 | 14 | 42 | 17
  CREA,Normal,Month 6,Above: number analyzed (Participants) | 41 | 15 | 44 | 17
  CREA,Normal,Month 6,Above | 0 | 0 | 0 | 0
  CREA,Normal,Month 6,Unknown: number analyzed (Participants) | 41 | 15 | 44 | 17
  CREA,Normal,Month 6,Unknown | 4 | 1 | 2 | 0
  CREA,Unknown,Month 12,Below: number analyzed (Participants) | 3 | 2 | 3 | 1
  CREA,Unknown,Month 12,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Month 12,Normal: number analyzed (Participants) | 3 | 2 | 3 | 1
  CREA,Unknown,Month 12,Normal | 3 | 2 | 3 | 1
  CREA,Unknown,Month 12,Above: number analyzed (Participants) | 3 | 2 | 3 | 1
  CREA,Unknown,Month 12,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Month 12,Unknown: number analyzed (Participants) | 3 | 2 | 3 | 1
  CREA,Unknown,Month 12,Unknown | 0 | 0 | 0 | 0
  CREA,Normal,Month 12,Below: number analyzed (Participants) | 41 | 15 | 45 | 17
  CREA,Normal,Month 12,Below | 0 | 0 | 0 | 0
  CREA,Normal,Month 12,Normal: number analyzed (Participants) | 41 | 15 | 45 | 17
  CREA,Normal,Month 12,Normal | 39 | 15 | 43 | 16
  CREA,Normal,Month 12,Above: number analyzed (Participants) | 41 | 15 | 45 | 17
  CREA,Normal,Month 12,Above | 0 | 0 | 0 | 0
  CREA,Normal,Month 12,Unknown: number analyzed (Participants) | 41 | 15 | 45 | 17
  CREA,Normal,Month 12,Unknown | 2 | 0 | 2 | 1
  CREA,Unknown,Month 24,Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  CREA,Unknown,Month 24,Below | 0 | 0 | 0 | 0
  CREA,Unknown,Month 24,Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  CREA,Unknown,Month 24,Normal | 2 | 2 | 2 | 1
  CREA,Unknown,Month 24,Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  CREA,Unknown,Month 24,Above | 0 | 0 | 0 | 0
  CREA,Unknown,Month 24,Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  CREA,Unknown,Month 24,Unknown | 1 | 0 | 0 | 0
  CREA,Normal,Month 24,Below: number analyzed (Participants) | 39 | 15 | 44 | 17
  CREA,Normal,Month 24,Below | 0 | 0 | 0 | 0
  CREA,Normal,Month 24,Normal: number analyzed (Participants) | 39 | 15 | 44 | 17
  CREA,Normal,Month 24,Normal | 39 | 15 | 44 | 17
  CREA,Normal,Month 24,Above: number analyzed (Participants) | 39 | 15 | 44 | 17
  CREA,Normal,Month 24,Above | 0 | 0 | 0 | 0
  CREA,Normal,Month 24,Unknown: number analyzed (Participants) | 39 | 15 | 44 | 17
  CREA,Normal,Month 24,Unknown | 0 | 0 | 0 | 0

46. Primary Outcome: Number of Subjects With Changed Status With Regards to Creatine Phosphokinase (CPK) in Study Phase C
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for CPK for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  CPK,Unknown,Day 21,Below: number analyzed (Participants) | 5 | 1 | 2 | 1
  CPK,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Day 21,Normal: number analyzed (Participants) | 5 | 1 | 2 | 1
  CPK,Unknown,Day 21,Normal | 3 | 0 | 0 | 1
  CPK,Unknown,Day 21,Above: number analyzed (Participants) | 5 | 1 | 2 | 1
  CPK,Unknown,Day 21,Above | 0 | 0 | 1 | 0
  CPK,Unknown,Day 21,Unknown: number analyzed (Participants) | 5 | 1 | 2 | 1
  CPK,Unknown,Day 21,Unknown | 2 | 1 | 1 | 0
  CPK,Normal,Day 21,Below: number analyzed (Participants) | 42 | 13 | 41 | 16
  CPK,Normal,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Normal,Day 21,Normal: number analyzed (Participants) | 42 | 13 | 41 | 16
  CPK,Normal,Day 21,Normal | 39 | 10 | 37 | 14
  CPK,Normal,Day 21,Above: number analyzed (Participants) | 42 | 13 | 41 | 16
  CPK,Normal,Day 21,Above | 2 | 0 | 0 | 2
  CPK,Normal,Day 21,Unknown: number analyzed (Participants) | 42 | 13 | 41 | 16
  CPK,Normal,Day 21,Unknown | 1 | 3 | 4 | 0
  CPK,Above,Day 21,Below: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 21,Below | 0 | 0 | 0 | 0
  CPK,Above,Day 21,Normal: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 21,Normal | 1 | 1 | 4 | 1
  CPK,Above,Day 21,Above: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 21,Above | 0 | 1 | 0 | 0
  CPK,Above,Day 21,Unknown: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 21,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown,Day 42,Below: number analyzed (Participants) | 5 | 2 | 2 | 1
  CPK,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Day 42,Normal: number analyzed (Participants) | 5 | 2 | 2 | 1
  CPK,Unknown,Day 42,Normal | 5 | 1 | 2 | 1
  CPK,Unknown,Day 42,Above: number analyzed (Participants) | 5 | 2 | 2 | 1
  CPK,Unknown,Day 42,Above | 0 | 1 | 0 | 0
  CPK,Unknown,Day 42,Unknown: number analyzed (Participants) | 5 | 2 | 2 | 1
  CPK,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  CPK,Normal,Day 42,Below: number analyzed (Participants) | 42 | 13 | 42 | 16
  CPK,Normal,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Normal,Day 42,Normal: number analyzed (Participants) | 42 | 13 | 42 | 16
  CPK,Normal,Day 42,Normal | 39 | 11 | 40 | 15
  CPK,Normal,Day 42,Above: number analyzed (Participants) | 42 | 13 | 42 | 16
  CPK,Normal,Day 42,Above | 1 | 1 | 0 | 1
  CPK,Normal,Day 42,Unknown: number analyzed (Participants) | 42 | 13 | 42 | 16
  CPK,Normal,Day 42,Unknown | 2 | 1 | 2 | 0
  CPK,Above,Day 42,Below: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 42,Below | 0 | 0 | 0 | 0
  CPK,Above,Day 42,Normal: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 42,Normal | 0 | 1 | 4 | 1
  CPK,Above,Day 42,Above: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 42,Above | 1 | 1 | 0 | 0
  CPK,Above,Day 42,Unknown: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown,Month 6,Below: number analyzed (Participants) | 4 | 2 | 2 | 1
  CPK,Unknown,Month 6,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Month 6,Normal: number analyzed (Participants) | 4 | 2 | 2 | 1
  CPK,Unknown,Month 6,Normal | 3 | 2 | 2 | 1
  CPK,Unknown,Month 6,Above: number analyzed (Participants) | 4 | 2 | 2 | 1
  CPK,Unknown,Month 6,Above | 1 | 0 | 0 | 0
  CPK,Unknown,Month 6,Unknown: number analyzed (Participants) | 4 | 2 | 2 | 1
  CPK,Unknown,Month 6,Unknown | 0 | 0 | 0 | 0
  CPK,Normal,Month 6,Below: number analyzed (Participants) | 40 | 13 | 40 | 16
  CPK,Normal,Month 6,Below | 0 | 0 | 0 | 0
  CPK,Normal,Month 6,Normal: number analyzed (Participants) | 40 | 13 | 40 | 16
  CPK,Normal,Month 6,Normal | 34 | 12 | 36 | 16
  CPK,Normal,Month 6,Above: number analyzed (Participants) | 40 | 13 | 40 | 16
  CPK,Normal,Month 6,Above | 2 | 0 | 3 | 0
  CPK,Normal,Month 6,Unknown: number analyzed (Participants) | 40 | 13 | 40 | 16
  CPK,Normal,Month 6,Unknown | 4 | 1 | 1 | 0
  CPK,Above,Month 6,Below: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 6,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 6,Normal: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 6,Normal | 0 | 1 | 3 | 1
  CPK,Above,Month 6,Above: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 6,Above | 1 | 1 | 0 | 0
  CPK,Above,Month 6,Unknown: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 6,Unknown | 0 | 0 | 1 | 0
  CPK,Unknown,Month 12,Below: number analyzed (Participants) | 3 | 2 | 3 | 1
  CPK,Unknown,Month 12,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Month 12,Normal: number analyzed (Participants) | 3 | 2 | 3 | 1
  CPK,Unknown,Month 12,Normal | 2 | 2 | 2 | 1
  CPK,Unknown,Month 12,Above: number analyzed (Participants) | 3 | 2 | 3 | 1
  CPK,Unknown,Month 12,Above | 1 | 0 | 1 | 0
  CPK,Unknown,Month 12,Unknown: number analyzed (Participants) | 3 | 2 | 3 | 1
  CPK,Unknown,Month 12,Unknown | 0 | 0 | 0 | 0
  CPK,Normal,Month 12,Below: number analyzed (Participants) | 40 | 13 | 41 | 16
  CPK,Normal,Month 12,Below | 0 | 0 | 0 | 0
  CPK,Normal,Month 12,Normal: number analyzed (Participants) | 40 | 13 | 41 | 16
  CPK,Normal,Month 12,Normal | 35 | 12 | 36 | 14
  CPK,Normal,Month 12,Above: number analyzed (Participants) | 40 | 13 | 41 | 16
  CPK,Normal,Month 12,Above | 3 | 1 | 3 | 1
  CPK,Normal,Month 12,Unknown: number analyzed (Participants) | 40 | 13 | 41 | 16
  CPK,Normal,Month 12,Unknown | 2 | 0 | 2 | 1
  CPK,Above,Month 12,Below: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 12,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 12,Normal: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 12,Normal | 1 | 1 | 4 | 1
  CPK,Above,Month 12,Above: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 12,Above | 0 | 1 | 0 | 0
  CPK,Above,Month 12,Unknown: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 12,Unknown | 0 | 0 | 0 | 0
  CPK,Unknown,Month 24,Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  CPK,Unknown,Month 24,Below | 0 | 0 | 0 | 0
  CPK,Unknown,Month 24,Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  CPK,Unknown,Month 24,Normal | 2 | 2 | 2 | 1
  CPK,Unknown,Month 24,Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  CPK,Unknown,Month 24,Above | 0 | 0 | 0 | 0
  CPK,Unknown,Month 24,Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  CPK,Unknown,Month 24,Unknown | 1 | 0 | 0 | 0
  CPK,Normal,Month 24,Below: number analyzed (Participants) | 38 | 13 | 40 | 16
  CPK,Normal,Month 24,Below | 0 | 0 | 0 | 0
  CPK,Normal,Month 24,Normal: number analyzed (Participants) | 38 | 13 | 40 | 16
  CPK,Normal,Month 24,Normal | 36 | 12 | 38 | 14
  CPK,Normal,Month 24,Above: number analyzed (Participants) | 38 | 13 | 40 | 16
  CPK,Normal,Month 24,Above | 2 | 1 | 2 | 2
  CPK,Normal,Month 24,Unknown: number analyzed (Participants) | 38 | 13 | 40 | 16
  CPK,Normal,Month 24,Unknown | 0 | 0 | 0 | 0
  CPK,Above,Month 24,Below: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 24,Below | 0 | 0 | 0 | 0
  CPK,Above,Month 24,Normal: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 24,Normal | 1 | 1 | 3 | 1
  CPK,Above,Month 24,Above: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 24,Above | 0 | 1 | 1 | 0
  CPK,Above,Month 24,Unknown: number analyzed (Participants) | 1 | 2 | 4 | 1
  CPK,Above,Month 24,Unknown | 0 | 0 | 0 | 0

47. Primary Outcome: Number of Subjects With Changed Status With Regards to Lactate Dehydrogenase (LDH) in Study Phase C
Description: Changes from baseline are categorised as below, within, or above the normal ranges at each scheduled post-vaccination time point versus the category of the laboratory values at baseline. Assessed parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK) Per parameter and range, it was assessed according to baseline values whether laboratory values of the subjects were below normal, normal or above the normal range. This outcome presents results for LDH for subjects participating in Phase C of the study.
Time Frame: At Days 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 48 | 17 | 48 | 18
Participants
  LDH,Unknown,Day 21,Below: number analyzed (Participants) | 5 | 1 | 1 | 1
  LDH,Unknown,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Unknown,Day 21,Normal: number analyzed (Participants) | 5 | 1 | 1 | 1
  LDH,Unknown,Day 21,Normal | 2 | 0 | 0 | 1
  LDH,Unknown,Day 21,Above: number analyzed (Participants) | 5 | 1 | 1 | 1
  LDH,Unknown,Day 21,Above | 1 | 0 | 0 | 0
  LDH,Unknown,Day 21,Unknown: number analyzed (Participants) | 5 | 1 | 1 | 1
  LDH,Unknown,Day 21,Unknown | 2 | 1 | 1 | 0
  LDH,Normal,Day 21,Below: number analyzed (Participants) | 35 | 12 | 43 | 17
  LDH,Normal,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Normal,Day 21,Normal: number analyzed (Participants) | 35 | 12 | 43 | 17
  LDH,Normal,Day 21,Normal | 31 | 9 | 37 | 16
  LDH,Normal,Day 21,Above: number analyzed (Participants) | 35 | 12 | 43 | 17
  LDH,Normal,Day 21,Above | 4 | 1 | 2 | 1
  LDH,Normal,Day 21,Unknown: number analyzed (Participants) | 35 | 12 | 43 | 17
  LDH,Normal,Day 21,Unknown | 0 | 2 | 4 | 0
  LDH,Above,Day 21,Below: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 21,Below | 0 | 0 | 0 | 0
  LDH,Above,Day 21,Normal: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 21,Normal | 5 | 2 | 2 | 0
  LDH,Above,Day 21,Above: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 21,Above | 2 | 0 | 1 | 0
  LDH,Above,Day 21,Unknown: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 21,Unknown | 1 | 1 | 0 | 0
  LDH,Unknown,Day 42,Below: number analyzed (Participants) | 5 | 2 | 1 | 1
  LDH,Unknown,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Unknown,Day 42,Normal: number analyzed (Participants) | 5 | 2 | 1 | 1
  LDH,Unknown,Day 42,Normal | 4 | 0 | 1 | 1
  LDH,Unknown,Day 42,Above: number analyzed (Participants) | 5 | 2 | 1 | 1
  LDH,Unknown,Day 42,Above | 1 | 2 | 0 | 0
  LDH,Unknown,Day 42,Unknown: number analyzed (Participants) | 5 | 2 | 1 | 1
  LDH,Unknown,Day 42,Unknown | 0 | 0 | 0 | 0
  LDH,Normal,Day 42,Below: number analyzed (Participants) | 35 | 12 | 44 | 17
  LDH,Normal,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Normal,Day 42,Normal: number analyzed (Participants) | 35 | 12 | 44 | 17
  LDH,Normal,Day 42,Normal | 29 | 7 | 39 | 16
  LDH,Normal,Day 42,Above: number analyzed (Participants) | 35 | 12 | 44 | 17
  LDH,Normal,Day 42,Above | 4 | 4 | 3 | 1
  LDH,Normal,Day 42,Unknown: number analyzed (Participants) | 35 | 12 | 44 | 17
  LDH,Normal,Day 42,Unknown | 2 | 1 | 2 | 0
  LDH,Above,Day 42,Below: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 42,Below | 0 | 0 | 0 | 0
  LDH,Above,Day 42,Normal: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 42,Normal | 2 | 1 | 2 | 0
  LDH,Above,Day 42,Above: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 42,Above | 6 | 2 | 1 | 0
  LDH,Above,Day 42,Unknown: number analyzed (Participants) | 8 | 3 | 3 | 0
  LDH,Above,Day 42,Unknown | 0 | 0 | 0 | 0
  LDH, Unknown, Month 6, Below: number analyzed (Participants) | 4 | 2 | 1 | 1
  LDH, Unknown, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Unknown, Month 6, Normal: number analyzed (Participants) | 4 | 2 | 1 | 1
  LDH, Unknown, Month 6, Normal | 2 | 0 | 1 | 1
  LDH,Unknown, Month 6, Above: number analyzed (Participants) | 4 | 2 | 1 | 1
  LDH,Unknown, Month 6, Above | 1 | 2 | 0 | 0
  LDH, Unknown, Month 6, Unknown: number analyzed (Participants) | 4 | 2 | 1 | 1
  LDH, Unknown, Month 6, Unknown | 1 | 0 | 0 | 0
  LDH, Normal, Month 6, Below: number analyzed (Participants) | 34 | 12 | 42 | 17
  LDH, Normal, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Normal, Month 6, Normal: number analyzed (Participants) | 34 | 12 | 42 | 17
  LDH, Normal, Month 6, Normal | 28 | 8 | 37 | 17
  LDH, Normal, Month 6, Above: number analyzed (Participants) | 34 | 12 | 42 | 17
  LDH, Normal, Month 6, Above | 2 | 3 | 3 | 0
  LDH, Normal, Month 6, Unknown: number analyzed (Participants) | 34 | 12 | 42 | 17
  LDH, Normal, Month 6, Unknown | 4 | 1 | 2 | 0
  LDH, Above, Month 6, Below: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Above, Month 6, Normal: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 6, Normal | 2 | 2 | 2 | 0
  LDH, Above, Month 6, Above: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 6, Above | 5 | 1 | 1 | 0
  LDH, Above, Month 6, Unknown: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 6, Unknown | 0 | 0 | 0 | 0
  LDH, Unknown, Month 12, Below: number analyzed (Participants) | 3 | 2 | 2 | 1
  LDH, Unknown, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Unknown, Month 12, Normal: number analyzed (Participants) | 3 | 2 | 2 | 1
  LDH, Unknown, Month 12, Normal | 3 | 2 | 0 | 1
  LDH, Unknown, Month 12, Above: number analyzed (Participants) | 3 | 2 | 2 | 1
  LDH, Unknown, Month 12, Above | 0 | 0 | 2 | 0
  LDH, Unknown, Month 12, Unknown: number analyzed (Participants) | 3 | 2 | 2 | 1
  LDH, Unknown, Month 12, Unknown | 0 | 0 | 0 | 0
  LDH, Normal, Month 12, Below: number analyzed (Participants) | 34 | 12 | 43 | 17
  LDH, Normal, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Normal, Month 12, Normal: number analyzed (Participants) | 34 | 12 | 43 | 17
  LDH, Normal, Month 12, Normal | 26 | 9 | 34 | 14
  LDH, Normal, Month 12, Above: number analyzed (Participants) | 34 | 12 | 43 | 17
  LDH, Normal, Month 12, Above | 6 | 3 | 6 | 2
  LDH, Normal, Month 12, Unknwon: number analyzed (Participants) | 34 | 12 | 43 | 17
  LDH, Normal, Month 12, Unknwon | 2 | 0 | 3 | 1
  LDH, Above, Month 12, Below: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Above, Month 12, Normal: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 12, Normal | 1 | 1 | 2 | 0
  LDH, Above, Month 12, Above: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 12, Above | 5 | 2 | 1 | 0
  LDH, Above, Month 12, Unknown: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 12, Unknown | 1 | 0 | 0 | 0
  LDH, Unknown, Month 24, Below: number analyzed (Participants) | 3 | 2 | 1 | 1
  LDH, Unknown, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Unknown, Month 24, Normal: number analyzed (Participants) | 3 | 2 | 1 | 1
  LDH, Unknown, Month 24, Normal | 2 | 2 | 1 | 1
  LDH, Unknown, Month 24, Above: number analyzed (Participants) | 3 | 2 | 1 | 1
  LDH, Unknown, Month 24, Above | 0 | 0 | 0 | 0
  LDH, Unknown, Month 24, Unknown: number analyzed (Participants) | 3 | 2 | 1 | 1
  LDH, Unknown, Month 24, Unknown | 1 | 0 | 0 | 0
  LDH, Normal, Month 24, Below: number analyzed (Participants) | 32 | 12 | 42 | 17
  LDH, Normal, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Normal, Month 24, Normal: number analyzed (Participants) | 32 | 12 | 42 | 17
  LDH, Normal, Month 24, Normal | 24 | 10 | 40 | 16
  LDH, Normal, Month 24, Above: number analyzed (Participants) | 32 | 12 | 42 | 17
  LDH, Normal, Month 24, Above | 8 | 2 | 2 | 1
  LDH, Normal, Month 24, Unknown: number analyzed (Participants) | 32 | 12 | 42 | 17
  LDH, Normal, Month 24, Unknown | 0 | 0 | 0 | 0
  LDH, Above, Month 24, Below: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Above, Month 24, Normal: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 24, Normal | 2 | 2 | 2 | 0
  LDH, Above, Month 24, Above: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 24, Above | 5 | 1 | 1 | 0
  LDH, Above, Month 24, Unknown: number analyzed (Participants) | 7 | 3 | 3 | 0
  LDH, Above, Month 24, Unknown | 0 | 0 | 0 | 0

48. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Alanine Aminotransferase (ALT) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents ALT results for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 52 | 18 | 53 | 18
Participants
  ALT, Day 0, Below: number analyzed (Participants) | 52 | 18 | 53 | 17
  ALT, Day 0, Below | 0 | 0 | 0 | 0
  ALT, Day 0, Normal: number analyzed (Participants) | 52 | 18 | 53 | 17
  ALT, Day 0, Normal | 50 | 18 | 51 | 17
  ALT, Day 0, Above: number analyzed (Participants) | 52 | 18 | 53 | 17
  ALT, Day 0, Above | 2 | 0 | 2 | 0
  ALT, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 18
  ALT, Day 21, Below | 0 | 0 | 0 | 0
  ALT, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 18
  ALT, Day 21, Normal | 48 | 16 | 44 | 18
  ALT, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 18
  ALT, Day 21, Above | 0 | 0 | 0 | 0
  ALT, Day 42, Below: number analyzed (Participants) | 49 | 16 | 45 | 16
  ALT, Day 42, Below | 0 | 0 | 0 | 0
  ALT, Day 42, Normal: number analyzed (Participants) | 49 | 16 | 45 | 16
  ALT, Day 42, Normal | 49 | 15 | 45 | 16
  ALT, Day 42, Above: number analyzed (Participants) | 49 | 16 | 45 | 16
  ALT, Day 42, Above | 0 | 1 | 0 | 0
  ALT, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  ALT, Month 6, Below | 0 | 0 | 0 | 0
  ALT, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  ALT, Month 6, Normal | 48 | 15 | 42 | 17
  ALT, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  ALT, Month 6, Above | 1 | 0 | 1 | 0
  ALT, Month 12, Below: number analyzed (Participants) | 47 | 17 | 42 | 17
  ALT, Month 12, Below | 0 | 0 | 0 | 0
  ALT, Month 12, Normal: number analyzed (Participants) | 47 | 17 | 42 | 17
  ALT, Month 12, Normal | 46 | 17 | 41 | 17
  ALT, Month 12, Above: number analyzed (Participants) | 47 | 17 | 42 | 17
  ALT, Month 12, Above | 1 | 0 | 1 | 0
  ALT, Month 24, Below: number analyzed (Participants) | 47 | 16 | 40 | 14
  ALT, Month 24, Below | 0 | 0 | 0 | 0
  ALT, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 40 | 14
  ALT, Month 24, Normal | 47 | 16 | 40 | 14
  ALT, Month 24, Above: number analyzed (Participants) | 47 | 16 | 40 | 14
  ALT, Month 24, Above | 0 | 0 | 0 | 0

49. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Aspartate Aminotransferase (AST) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents AST results for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 52 | 18 | 53 | 18
Participants
  AST, Day 0, Below: number analyzed (Participants) | 52 | 18 | 53 | 17
  AST, Day 0, Below | 0 | 0 | 0 | 0
  AST, Day 0, Normal: number analyzed (Participants) | 52 | 18 | 53 | 17
  AST, Day 0, Normal | 46 | 18 | 51 | 17
  AST, Day 0, Above: number analyzed (Participants) | 52 | 18 | 53 | 17
  AST, Day 0, Above | 6 | 0 | 2 | 0
  AST, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 17
  AST, Day 21, Below | 0 | 0 | 0 | 0
  AST, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 17
  AST, Day 21, Normal | 42 | 16 | 44 | 17
  AST, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 17
  AST, Day 21, Above | 6 | 0 | 0 | 0
  AST, Day 42, Below: number analyzed (Participants) | 49 | 15 | 45 | 16
  AST, Day 42, Below | 0 | 0 | 0 | 0
  AST, Day 42, Normal: number analyzed (Participants) | 49 | 15 | 45 | 16
  AST, Day 42, Normal | 46 | 13 | 45 | 16
  AST, Day 42, Above: number analyzed (Participants) | 49 | 15 | 45 | 16
  AST, Day 42, Above | 3 | 2 | 0 | 0
  AST, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  AST, Month 6, Below | 0 | 0 | 0 | 0
  AST, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  AST, Month 6, Normal | 46 | 14 | 42 | 17
  AST, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  AST, Month 6, Above | 3 | 1 | 1 | 0
  AST, Month 12, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  AST, Month 12, Below | 0 | 0 | 0 | 0
  AST, Month 12, Normal: number analyzed (Participants) | 49 | 18 | 43 | 17
  AST, Month 12, Normal | 43 | 16 | 42 | 17
  AST, Month 12, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  AST, Month 12, Above | 4 | 1 | 0 | 0
  AST, Month 24, Below: number analyzed (Participants) | 47 | 16 | 40 | 14
  AST, Month 24, Below | 0 | 0 | 0 | 0
  AST, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 40 | 14
  AST, Month 24, Normal | 44 | 16 | 40 | 14
  AST, Month 24, Above: number analyzed (Participants) | 47 | 16 | 40 | 14
  AST, Month 24, Above | 3 | 0 | 0 | 0

50. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Blood Urea Nitrogen (BUN) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents BUN results for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 53 | 18 | 53 | 18
Participants
  BUN, Day 0, Below: number analyzed (Participants) | 52 | 18 | 53 | 17
  BUN, Day 0, Below | 0 | 0 | 0 | 0
  BUN, Day 0, Normal: number analyzed (Participants) | 52 | 18 | 53 | 17
  BUN, Day 0, Normal | 50 | 18 | 52 | 16
  BUN, Day 0, Above: number analyzed (Participants) | 52 | 18 | 53 | 17
  BUN, Day 0, Above | 2 | 0 | 1 | 1
  BUN, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 18
  BUN, Day 21, Below | 0 | 1 | 0 | 0
  BUN, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 18
  BUN, Day 21, Normal | 45 | 14 | 39 | 16
  BUN, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 18
  BUN, Day 21, Above | 3 | 1 | 5 | 2
  BUN, Day 42, Below: number analyzed (Participants) | 49 | 16 | 45 | 16
  BUN, Day 42, Below | 0 | 0 | 0 | 0
  BUN, Day 42, Normal: number analyzed (Participants) | 49 | 16 | 45 | 16
  BUN, Day 42, Normal | 42 | 16 | 39 | 14
  BUN, Day 42, Above: number analyzed (Participants) | 49 | 16 | 45 | 16
  BUN, Day 42, Above | 7 | 0 | 6 | 2
  BUN, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  BUN, Month 6, Below | 0 | 1 | 0 | 0
  BUN, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  BUN, Month 6, Normal | 46 | 13 | 39 | 15
  BUN, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  BUN, Month 6, Above | 3 | 1 | 4 | 2
  BUN, Month 12, Below: number analyzed (Participants) | 47 | 17 | 42 | 17
  BUN, Month 12, Below | 0 | 0 | 1 | 0
  BUN, Month 12, Normal: number analyzed (Participants) | 47 | 17 | 42 | 17
  BUN, Month 12, Normal | 42 | 16 | 41 | 15
  BUN, Month 12, Above: number analyzed (Participants) | 47 | 17 | 42 | 17
  BUN, Month 12, Above | 5 | 1 | 0 | 2
  BUN, Month 24, Below: number analyzed (Participants) | 47 | 16 | 40 | 14
  BUN, Month 24, Below | 0 | 0 | 1 | 0
  BUN, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 40 | 14
  BUN, Month 24, Normal | 45 | 16 | 38 | 12
  BUN, Month 24, Above: number analyzed (Participants) | 47 | 16 | 40 | 14
  BUN, Month 24, Above | 2 | 0 | 1 | 2

51. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatinine (CREA) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CREA results, for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 52 | 18 | 53 | 18
Participants
  CREA, Day 0, Below | 0 | 0 | 0 | 0
  CREA, Day 0, Normal | 52 | 18 | 53 | 17
  CREA, Day 0, Above | 0 | 0 | 0 | 0
  CREA, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 18
  CREA, Day 21, Below | 0 | 0 | 0 | 0
  CREA, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 18
  CREA, Day 21, Normal | 48 | 16 | 42 | 18
  CREA, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 18
  CREA, Day 21, Above | 0 | 0 | 2 | 0
  CREA, Day 42, Below: number analyzed (Participants) | 49 | 16 | 45 | 16
  CREA, Day 42, Below | 0 | 0 | 0 | 0
  CREA, Day 42, Normal: number analyzed (Participants) | 49 | 16 | 45 | 16
  CREA, Day 42, Normal | 49 | 16 | 43 | 16
  CREA, Day 42, Above: number analyzed (Participants) | 49 | 16 | 45 | 16
  CREA, Day 42, Above | 0 | 0 | 2 | 0
  CREA, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  CREA, Month 6, Below | 0 | 0 | 0 | 0
  CREA, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  CREA, Month 6, Normal | 49 | 15 | 43 | 17
  CREA, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  CREA, Month 6, Above | 0 | 0 | 0 | 0
  CREA, Month 12, Below: number analyzed (Participants) | 47 | 17 | 42 | 17
  CREA, Month 12, Below | 0 | 0 | 0 | 0
  CREA, Month 12, Normal: number analyzed (Participants) | 47 | 17 | 42 | 17
  CREA, Month 12, Normal | 47 | 17 | 42 | 17
  CREA, Month 12, Above: number analyzed (Participants) | 47 | 17 | 42 | 17
  CREA, Month 12, Above | 0 | 0 | 0 | 0
  CREA, Month 24, Below: number analyzed (Participants) | 47 | 16 | 40 | 14
  CREA, Month 24, Below | 0 | 0 | 0 | 0
  CREA, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 40 | 14
  CREA, Month 24, Normal | 47 | 16 | 39 | 14
  CREA, Month 24, Above: number analyzed (Participants) | 47 | 16 | 40 | 14
  CREA, Month 24, Above | 0 | 0 | 1 | 0

52. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatine Phosphokinase (CPK) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CPK results for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Groups:
- Fluarix-A 3-5Y Group: Fluarix-A 3-5Y Group
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 52 | 18 | 53 | 18
Participants
  CPK, Day 0, Below | 0 | 0 | 0 | 0
  CPK, Day 0, Normal | 51 | 17 | 51 | 17
  CPK, Day 0, Above | 1 | 1 | 2 | 0
  CPK, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 18
  CPK, Day 21, Below | 0 | 0 | 0 | 0
  CPK, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 18
  CPK, Day 21, Normal | 46 | 16 | 42 | 17
  CPK, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 18
  CPK, Day 21, Above | 2 | 0 | 2 | 1
  CPK, Day 42, Below: number analyzed (Participants) | 49 | 16 | 45 | 16
  CPK, Day 42, Below | 0 | 0 | 0 | 0
  CPK, Day 42, Normal: number analyzed (Participants) | 49 | 16 | 45 | 16
  CPK, Day 42, Normal | 47 | 14 | 42 | 15
  CPK, Day 42, Above: number analyzed (Participants) | 49 | 16 | 45 | 16
  CPK, Day 42, Above | 2 | 2 | 3 | 1
  CPK, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  CPK, Month 6, Below | 0 | 0 | 0 | 0
  CPK, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  CPK, Month 6, Normal | 47 | 14 | 38 | 16
  CPK, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  CPK, Month 6, Above | 2 | 1 | 5 | 1
  CPK, Month 12, Below: number analyzed (Participants) | 47 | 17 | 42 | 17
  CPK, Month 12, Below | 0 | 0 | 0 | 0
  CPK, Month 12, Normal: number analyzed (Participants) | 47 | 17 | 42 | 17
  CPK, Month 12, Normal | 45 | 15 | 40 | 16
  CPK, Month 12, Above: number analyzed (Participants) | 47 | 17 | 42 | 17
  CPK, Month 12, Above | 2 | 2 | 2 | 1
  CPK, Month 24, Below: number analyzed (Participants) | 47 | 16 | 39 | 14
  CPK, Month 24, Below | 0 | 0 | 0 | 0
  CPK, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 39 | 14
  CPK, Month 24, Normal | 47 | 15 | 36 | 13
  CPK, Month 24, Above: number analyzed (Participants) | 47 | 16 | 39 | 14
  CPK, Month 24, Above | 0 | 1 | 3 | 1

53. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Lactate Dehydrogenase (LDH) in Study Phase A
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents LDH results for subjects participating in Phase A of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 52 | 18 | 53 | 17
Participants
  LDH, Day 0, Below | 0 | 0 | 0 | 0
  LDH, Day 0, Normal | 41 | 12 | 52 | 17
  LDH, Day 0, Above | 11 | 6 | 1 | 0
  LDH, Day 21, Below: number analyzed (Participants) | 48 | 16 | 44 | 17
  LDH, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Day 21, Normal: number analyzed (Participants) | 48 | 16 | 44 | 17
  LDH, Day 21, Normal | 42 | 10 | 41 | 15
  LDH, Day 21, Above: number analyzed (Participants) | 48 | 16 | 44 | 17
  LDH, Day 21, Above | 6 | 6 | 3 | 2
  LDH, Day 42, Below: number analyzed (Participants) | 49 | 15 | 45 | 16
  LDH, Day 42, Below | 0 | 0 | 0 | 0
  LDH, Day 42, Normal: number analyzed (Participants) | 49 | 15 | 45 | 16
  LDH, Day 42, Normal | 38 | 9 | 42 | 15
  LDH, Day 42, Above: number analyzed (Participants) | 49 | 15 | 45 | 16
  LDH, Day 42, Above | 11 | 6 | 4 | 1
  LDH, Month 6, Below: number analyzed (Participants) | 49 | 15 | 43 | 17
  LDH, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Month 6, Normal: number analyzed (Participants) | 49 | 15 | 43 | 17
  LDH, Month 6, Normal | 37 | 11 | 39 | 14
  LDH, Month 6, Above: number analyzed (Participants) | 49 | 15 | 43 | 17
  LDH, Month 6, Above | 12 | 4 | 4 | 3
  LDH, Month 12, Below: number analyzed (Participants) | 47 | 17 | 42 | 17
  LDH, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Month 12, Normal: number analyzed (Participants) | 47 | 17 | 42 | 17
  LDH, Month 12, Normal | 40 | 12 | 41 | 15
  LDH, Month 12, Above: number analyzed (Participants) | 47 | 17 | 42 | 17
  LDH, Month 12, Above | 7 | 5 | 1 | 2
  LDH, Month 24, Below: number analyzed (Participants) | 42 | 16 | 49 | 14
  LDH, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Month 24, Normal: number analyzed (Participants) | 47 | 16 | 39 | 14
  LDH, Month 24, Normal | 42 | 13 | 36 | 12
  LDH, Month 24, Above: number analyzed (Participants) | 47 | 16 | 39 | 14
  LDH, Month 24, Above | 5 | 3 | 3 | 2

54. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Alanine Aminotransferase (ALT) in Study Phase B
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents AST results, for subjects participating to Phase B of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  ALT, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 17
  ALT, Day 0, Below | 0 | 0 | 0 | 0
  ALT, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 17
  ALT, Day 0, Normal | 50 | 16 | 48 | 16
  ALT, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 17
  ALT, Day 0, Above | 1 | 0 | 0 | 1
  ALT, Day 21, Below: number analyzed (Participants) | 45 | 17 | 46 | 17
  ALT, Day 21, Below | 0 | 0 | 0 | 0
  ALT, Day 21, Normal: number analyzed (Participants) | 45 | 17 | 46 | 17
  ALT, Day 21, Normal | 44 | 16 | 45 | 17
  ALT, Day 21, Above: number analyzed (Participants) | 45 | 17 | 46 | 17
  ALT, Day 21, Above | 1 | 1 | 1 | 0
  ALT, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  ALT, Day 42, Below | 0 | 0 | 0 | 0
  ALT, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  ALT, Day 42, Normal | 46 | 17 | 45 | 16
  ALT, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  ALT, Day 42, Above | 1 | 0 | 2 | 1
  ALT, Month 6, Below: number analyzed (Participants) | 41 | 16 | 43 | 17
  ALT, Month 6, Below | 0 | 0 | 0 | 0
  ALT, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 43 | 17
  ALT, Month 6, Normal | 41 | 16 | 43 | 17
  ALT, Month 6, Above: number analyzed (Participants) | 41 | 16 | 43 | 17
  ALT, Month 6, Above | 0 | 0 | 0 | 0
  ALT, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  ALT, Month 12, Below | 0 | 0 | 0 | 0
  ALT, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  ALT, Month 12, Normal | 44 | 17 | 45 | 17
  ALT, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  ALT, Month 12, Above | 0 | 0 | 0 | 0
  ALT, Month 24, Below: number analyzed (Participants) | 45 | 17 | 44 | 17
  ALT, Month 24, Below | 0 | 0 | 0 | 0
  ALT, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 44 | 17
  ALT, Month 24, Normal | 44 | 17 | 43 | 17
  ALT, Month 24, Above: number analyzed (Participants) | 45 | 17 | 44 | 17
  ALT, Month 24, Above | 1 | 0 | 1 | 0

55. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Aspartate Aminotransferase (AST) in Study Phase B
Description: as for outcome 54
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Groups:
- GSK1562902A -B Lot 1 3-5Y Group: Subjects aged 3-5 years received 2 doses of GSK1562902A vaccine, lot 1. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
- GSK1562902A-B Lot 1 6-9Y Group: Subjects aged 6-9 years received 2 doses of GSK1562902A vaccine, lot 1. These subjects were enrolled in the Phase B of this NCT00502593 study (or study 108498). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
Arm/Group | GSK1562902A -B Lot 1 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 1 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  AST, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 17
  AST, Day 0, Below | 0 | 0 | 0 | 0
  AST, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 17
  AST, Day 0, Normal | 48 | 15 | 45 | 16
  AST, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 17
  AST, Day 0, Above | 3 | 1 | 3 | 1
  AST, Day 21, Below: number analyzed (Participants) | 44 | 17 | 46 | 17
  AST, Day 21, Below | 0 | 0 | 0 | 0
  AST, Day 21, Normal: number analyzed (Participants) | 44 | 17 | 46 | 17
  AST, Day 21, Normal | 41 | 16 | 45 | 17
  AST, Day 21, Above: number analyzed (Participants) | 44 | 17 | 46 | 17
  AST, Day 21, Above | 3 | 1 | 1 | 0
  AST, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  AST, Day 42, Below | 0 | 0 | 0 | 0
  AST, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  AST, Day 42, Normal | 42 | 15 | 44 | 16
  AST, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  AST, Day 42, Above | 5 | 2 | 3 | 1
  AST, Month 6, Below: number analyzed (Participants) | 42 | 16 | 42 | 17
  AST, Month 6, Below | 0 | 0 | 0 | 0
  AST, Month 6, Normal: number analyzed (Participants) | 42 | 16 | 42 | 17
  AST, Month 6, Normal | 40 | 15 | 42 | 17
  AST, Month 6, Above: number analyzed (Participants) | 42 | 16 | 42 | 17
  AST, Month 6, Above | 2 | 1 | 0 | 0
  AST, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  AST, Month 12, Below | 0 | 0 | 0 | 0
  AST, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  AST, Month 12, Normal | 44 | 17 | 45 | 17
  AST, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  AST, Month 12, Above | 0 | 0 | 0 | 0
  AST, Month 24, Below: number analyzed (Participants) | 45 | 17 | 44 | 17
  AST, Month 24, Below | 0 | 0 | 0 | 0
  AST, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 44 | 17
  AST, Month 24, Normal | 44 | 17 | 43 | 17
  AST, Month 24, Above: number analyzed (Participants) | 45 | 17 | 44 | 17
  AST, Month 24, Above | 1 | 0 | 1 | 0

56. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatinine (CREA) in Study Phase B
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CREA results, for subjects participating in Phase B of the study.
Time Frame: At Days 0, 21 and 42 and at Month 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  CREA, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 17
  CREA, Day 0, Below | 0 | 0 | 0 | 0
  CREA, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 17
  CREA, Day 0, Normal | 51 | 16 | 47 | 17
  CREA, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 17
  CREA, Day 0, Above | 0 | 0 | 1 | 0
  CREA, Day 21, Below: number analyzed (Participants) | 45 | 17 | 46 | 17
  CREA, Day 21, Below | 0 | 0 | 0 | 0
  CREA, Day 21, Normal: number analyzed (Participants) | 45 | 17 | 46 | 17
  CREA, Day 21, Normal | 44 | 17 | 45 | 17
  CREA, Day 21, Above: number analyzed (Participants) | 45 | 17 | 46 | 17
  CREA, Day 21, Above | 1 | 0 | 1 | 0
  CREA, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  CREA, Day 42, Below | 0 | 0 | 0 | 0
  CREA, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  CREA, Day 42, Normal | 46 | 17 | 47 | 17
  CREA, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  CREA, Day 42, Above | 1 | 0 | 0 | 0
  CREA, Month 6, Below: number analyzed (Participants) | 42 | 16 | 43 | 17
  CREA, Month 6, Below | 0 | 0 | 0 | 0
  CREA, Month 6, Normal: number analyzed (Participants) | 42 | 16 | 43 | 17
  CREA, Month 6, Normal | 42 | 16 | 41 | 17
  CREA, Month 6, Above: number analyzed (Participants) | 42 | 16 | 43 | 17
  CREA, Month 6, Above | 0 | 0 | 2 | 0
  CREA, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  CREA, Month 12, Below | 0 | 0 | 0 | 0
  CREA, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  CREA, Month 12, Normal | 44 | 17 | 44 | 17
  CREA, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  CREA, Month 12, Above | 0 | 0 | 1 | 0
  CREA, Month 24, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  CREA, Month 24, Below | 0 | 0 | 0 | 0
  CREA, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 45 | 17
  CREA, Month 24, Normal | 45 | 17 | 44 | 17
  CREA, Month 24, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  CREA, Month 24, Above | 0 | 0 | 0 | 0

57. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Lactate Dehydrogenase (LDH) in Study Phase B
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents LDH results, for subjects participating to Phase B of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  LDH, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 17
  LDH, Day 0, Below | 0 | 0 | 0 | 0
  LDH, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 17
  LDH, Day 0, Normal | 46 | 14 | 41 | 15
  LDH, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 17
  LDH, Day 0, Above | 5 | 2 | 7 | 2
  LDH, Day 21, Below: number analyzed (Participants) | 44 | 17 | 46 | 17
  LDH, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Day 21, Normal: number analyzed (Participants) | 44 | 17 | 46 | 17
  LDH, Day 21, Normal | 35 | 14 | 42 | 16
  LDH, Day 21, Above: number analyzed (Participants) | 44 | 17 | 46 | 17
  LDH, Day 21, Above | 9 | 3 | 4 | 1
  LDH, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  LDH, Day 42, Below | 0 | 0 | 0 | 0
  LDH, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  LDH, Day 42, Normal | 35 | 10 | 41 | 14
  LDH, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  LDH, Day 42, Above | 12 | 7 | 6 | 3
  LDH, Month 6, Below: number analyzed (Participants) | 41 | 16 | 42 | 17
  LDH, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 42 | 17
  LDH, Month 6, Normal | 35 | 11 | 36 | 15
  LDH, Month 6, Above: number analyzed (Participants) | 41 | 16 | 42 | 17
  LDH, Month 6, Above | 6 | 5 | 6 | 2
  LDH, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  LDH, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  LDH, Month 12, Normal | 35 | 12 | 42 | 16
  LDH, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  LDH, Month 12, Above | 9 | 5 | 3 | 1
  LDH, Month 24, Below: number analyzed (Participants) | 45 | 17 | 44 | 17
  LDH, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 44 | 17
  LDH, Month 24, Normal | 43 | 16 | 41 | 15
  LDH, Month 24, Above: number analyzed (Participants) | 45 | 17 | 44 | 17
  LDH, Month 24, Above | 2 | 1 | 3 | 2

58. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Blood Urea Nitrogen (BUN) in Study Phase B
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents BUN results, for subjects participating to Phase B of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  BUN, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 16
  BUN, Day 0, Below | 0 | 0 | 0 | 0
  BUN, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 16
  BUN, Day 0, Normal | 47 | 14 | 43 | 13
  BUN, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 16
  BUN, Day 0, Above | 4 | 2 | 5 | 3
  BUN, Day 21, Below: number analyzed (Participants) | 45 | 17 | 46 | 17
  BUN, Day 21, Below | 0 | 0 | 0 | 0
  BUN, Day 21, Normal: number analyzed (Participants) | 45 | 17 | 46 | 17
  BUN, Day 21, Normal | 38 | 14 | 43 | 15
  BUN, Day 21, Above: number analyzed (Participants) | 45 | 17 | 46 | 17
  BUN, Day 21, Above | 7 | 3 | 3 | 2
  BUN, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  BUN, Day 42, Below | 0 | 0 | 0 | 0
  BUN, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  BUN, Day 42, Normal | 40 | 14 | 43 | 14
  BUN, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  BUN, Day 42, Above | 7 | 3 | 4 | 3
  BUN, Month 6, Below: number analyzed (Participants) | 42 | 16 | 43 | 17
  BUN, Month 6, Below | 0 | 0 | 0 | 0
  BUN, Month 6, Normal: number analyzed (Participants) | 42 | 16 | 43 | 17
  BUN, Month 6, Normal | 42 | 13 | 43 | 17
  BUN, Month 6, Above: number analyzed (Participants) | 42 | 16 | 43 | 17
  BUN, Month 6, Above | 0 | 3 | 0 | 0
  BUN, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  BUN, Month 12, Below | 0 | 0 | 0 | 0
  BUN, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  BUN, Month 12, Normal | 39 | 15 | 44 | 14
  BUN, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  BUN, Month 12, Above | 5 | 2 | 1 | 3
  BUN, Month 24, Below: number analyzed (Participants) | 45 | 17 | 44 | 17
  BUN, Month 24, Below | 0 | 0 | 0 | 0
  BUN, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 44 | 17
  BUN, Month 24, Normal | 40 | 13 | 41 | 16
  BUN, Month 24, Above: number analyzed (Participants) | 45 | 17 | 44 | 17
  BUN, Month 24, Above | 5 | 4 | 3 | 1

59. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Blood Urea Nitrogen (BUN) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents BUN results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21 and 42 and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 47 | 18
Participants
  BUN, Day 0, Below: number analyzed (Participants) | 44 | 15 | 47 | 17
  BUN, Day 0, Below | 0 | 1 | 0 | 0
  BUN, Day 0, Normal: number analyzed (Participants) | 44 | 15 | 47 | 17
  BUN, Day 0, Normal | 42 | 11 | 46 | 17
  BUN, Day 0, Above: number analyzed (Participants) | 44 | 15 | 47 | 17
  BUN, Day 0, Above | 2 | 3 | 1 | 0
  BUN, Day 21, Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  BUN, Day 21, Below | 1 | 0 | 0 | 0
  BUN, Day 21, Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  BUN, Day 21, Normal | 42 | 12 | 42 | 17
  BUN, Day 21, Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  BUN, Day 21, Above | 2 | 0 | 0 | 1
  BUN, Day 42, Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  BUN, Day 42, Below | 0 | 0 | 3 | 0
  BUN, Day 42, Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  BUN, Day 42, Normal | 43 | 16 | 40 | 17
  BUN, Day 42, Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  BUN, Day 42, Above | 3 | 0 | 3 | 1
  BUN, Month 6, Below: number analyzed (Participants) | 41 | 16 | 44 | 18
  BUN, Month 6, Below | 0 | 0 | 2 | 0
  BUN, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 44 | 18
  BUN, Month 6, Normal | 40 | 15 | 36 | 18
  BUN, Month 6, Above: number analyzed (Participants) | 41 | 16 | 44 | 18
  BUN, Month 6, Above | 1 | 1 | 6 | 0
  BUN, Month 12, Below: number analyzed (Participants) | 42 | 12 | 46 | 17
  BUN, Month 12, Below | 0 | 0 | 0 | 0
  BUN, Month 12, Normal: number analyzed (Participants) | 42 | 17 | 46 | 17
  BUN, Month 12, Normal | 41 | 15 | 43 | 17
  BUN, Month 12, Above: number analyzed (Participants) | 42 | 12 | 46 | 17
  BUN, Month 12, Above | 1 | 2 | 3 | 0
  BUN, Month 24, Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  BUN, Month 24, Below | 0 | 0 | 1 | 0
  BUN, Month 24, Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  BUN, Month 24, Normal | 39 | 15 | 40 | 17
  BUN, Month 24, Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  BUN, Month 24, Above | 2 | 2 | 5 | 1

60. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Alanine Aminotransferase (ALT) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents ALT results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 46 | 18
Participants
  ALT,Day 0,Below: number analyzed (Participants) | 44 | 15 | 46 | 17
  ALT,Day 0,Below | 0 | 0 | 0 | 0
  ALT, Day 0,Normal: number analyzed (Participants) | 44 | 15 | 46 | 17
  ALT, Day 0,Normal | 43 | 15 | 45 | 17
  ALT,Day 0,Above: number analyzed (Participants) | 44 | 15 | 46 | 17
  ALT,Day 0,Above | 1 | 0 | 1 | 0
  ALT,Day 21,Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  ALT,Day 21,Below | 0 | 0 | 0 | 0
  ALT,Day 21,Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  ALT,Day 21,Normal | 44 | 12 | 42 | 18
  ALT,Day 21,Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  ALT,Day 21,Above | 1 | 0 | 0 | 0
  ALT,Day 42,Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  ALT,Day 42,Below | 0 | 0 | 0 | 0
  ALT,Day 42,Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  ALT,Day 42,Normal | 46 | 16 | 46 | 18
  ALT,Day 42,Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  ALT,Day 42,Above | 0 | 0 | 0 | 0
  ALT, Month 6, Below: number analyzed (Participants) | 41 | 16 | 44 | 18
  ALT, Month 6, Below | 0 | 0 | 0 | 0
  ALT, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 44 | 18
  ALT, Month 6, Normal | 41 | 15 | 44 | 18
  ALT, Month 6, Above: number analyzed (Participants) | 41 | 16 | 44 | 18
  ALT, Month 6, Above | 0 | 1 | 0 | 0
  ALT,Month12,Below: number analyzed (Participants) | 42 | 17 | 46 | 17
  ALT,Month12,Below | 0 | 0 | 0 | 0
  ALT,Month 12,Normal: number analyzed (Participants) | 42 | 17 | 46 | 17
  ALT,Month 12,Normal | 42 | 17 | 44 | 17
  ALT,Month 12,Above: number analyzed (Participants) | 42 | 17 | 46 | 17
  ALT,Month 12,Above | 0 | 0 | 2 | 0
  ALT,Month 24,Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  ALT,Month 24,Below | 0 | 0 | 0 | 0
  ALT,Month 24,Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  ALT,Month 24,Normal | 39 | 17 | 44 | 18
  ALT,Month 24,Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  ALT,Month 24,Above | 2 | 0 | 2 | 0

61. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatine Phosphokinase (CPK) in Study Phase B
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CPK results, for subjects participating to Phase B of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 51 | 17 | 48 | 17
Participants
  CPK, Day 0, Below: number analyzed (Participants) | 51 | 16 | 48 | 17
  CPK, Day 0, Below | 0 | 0 | 0 | 0
  CPK, Day 0, Normal: number analyzed (Participants) | 51 | 16 | 48 | 17
  CPK, Day 0, Normal | 49 | 16 | 46 | 16
  CPK, Day 0, Above: number analyzed (Participants) | 51 | 16 | 48 | 17
  CPK, Day 0, Above | 2 | 0 | 2 | 1
  CPK, Day 21, Below: number analyzed (Participants) | 45 | 17 | 46 | 17
  CPK, Day 21, Below | 0 | 0 | 0 | 0
  CPK, Day 21, Normal: number analyzed (Participants) | 45 | 17 | 46 | 17
  CPK, Day 21, Normal | 42 | 16 | 45 | 16
  CPK, Day 21, Above: number analyzed (Participants) | 45 | 17 | 46 | 17
  CPK, Day 21, Above | 3 | 1 | 1 | 1
  CPK, Day 42, Below: number analyzed (Participants) | 47 | 17 | 47 | 17
  CPK, Day 42, Below | 0 | 0 | 0 | 0
  CPK, Day 42, Normal: number analyzed (Participants) | 47 | 17 | 47 | 17
  CPK, Day 42, Normal | 43 | 15 | 44 | 16
  CPK, Day 42, Above: number analyzed (Participants) | 47 | 17 | 47 | 17
  CPK, Day 42, Above | 4 | 2 | 3 | 1
  CPK, Month 6, Below: number analyzed (Participants) | 42 | 16 | 43 | 17
  CPK, Month 6, Below | 0 | 0 | 0 | 0
  CPK, Month 6, Normal: number analyzed (Participants) | 42 | 16 | 43 | 17
  CPK, Month 6, Normal | 40 | 13 | 41 | 15
  CPK, Month 6, Above: number analyzed (Participants) | 42 | 16 | 43 | 17
  CPK, Month 6, Above | 2 | 3 | 2 | 2
  CPK, Month 12, Below: number analyzed (Participants) | 44 | 17 | 45 | 17
  CPK, Month 12, Below | 0 | 0 | 0 | 0
  CPK, Month 12, Normal: number analyzed (Participants) | 44 | 17 | 45 | 17
  CPK, Month 12, Normal | 39 | 14 | 44 | 17
  CPK, Month 12, Above: number analyzed (Participants) | 44 | 17 | 45 | 17
  CPK, Month 12, Above | 5 | 3 | 1 | 0
  CPK, Month 24, Below: number analyzed (Participants) | 45 | 17 | 44 | 17
  CPK, Month 24, Below | 0 | 0 | 0 | 0
  CPK, Month 24, Normal: number analyzed (Participants) | 45 | 17 | 44 | 17
  CPK, Month 24, Normal | 44 | 15 | 42 | 16
  CPK, Month 24, Above: number analyzed (Participants) | 45 | 17 | 44 | 17
  CPK, Month 24, Above | 1 | 2 | 2 | 1

62. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Aspartate Aminotransferase (AST) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents AST results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 46 | 18
Participants
  AST,Day 0,Below: number analyzed (Participants) | 44 | 15 | 46 | 17
  AST,Day 0,Below | 0 | 0 | 0 | 0
  AST,Day 0,Normal: number analyzed (Participants) | 44 | 15 | 46 | 17
  AST,Day 0,Normal | 41 | 12 | 45 | 17
  AST,Day 0,Above: number analyzed (Participants) | 44 | 15 | 46 | 17
  AST,Day 0,Above | 3 | 3 | 1 | 0
  AST, Day 21,Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  AST, Day 21,Below | 0 | 0 | 0 | 0
  AST,Day 21,Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  AST,Day 21,Normal | 44 | 12 | 42 | 18
  AST,Day 21,Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  AST,Day 21,Above | 1 | 0 | 0 | 0
  AST,Day 42,Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  AST,Day 42,Below | 0 | 0 | 0 | 0
  AST,Day 42,Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  AST,Day 42,Normal | 44 | 14 | 43 | 18
  AST,Day 42,Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  AST,Day 42,Above | 2 | 2 | 3 | 0
  AST,Month 6,Below: number analyzed (Participants) | 40 | 16 | 44 | 18
  AST,Month 6,Below | 0 | 0 | 0 | 0
  AST, Month 6, Normal: number analyzed (Participants) | 40 | 16 | 44 | 18
  AST, Month 6, Normal | 39 | 14 | 43 | 18
  AST, Month 6, Above: number analyzed (Participants) | 40 | 16 | 44 | 18
  AST, Month 6, Above | 1 | 2 | 1 | 0
  AST,Month 12,Below: number analyzed (Participants) | 41 | 17 | 45 | 17
  AST,Month 12,Below | 0 | 0 | 0 | 0
  AST,Month 12,Normal: number analyzed (Participants) | 41 | 17 | 45 | 17
  AST,Month 12,Normal | 41 | 17 | 40 | 17
  AST,Month 12,Above: number analyzed (Participants) | 41 | 17 | 45 | 17
  AST,Month 12,Above | 0 | 0 | 5 | 0
  AST,Month 24,Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  AST,Month 24,Below | 0 | 0 | 0 | 0
  AST,Month 24,Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  AST,Month 24,Normal | 38 | 17 | 45 | 18
  AST,Month 24,Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  AST,Month 24,Above | 3 | 0 | 1 | 0

63. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatine Phosphokinase (CPK) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CPK results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21, and 42, and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 46 | 18
Participants
  CPK, Day 0, Below: number analyzed (Participants) | 44 | 15 | 46 | 17
  CPK, Day 0, Below | 0 | 0 | 0 | 0
  CPK, Day 0, Normal: number analyzed (Participants) | 44 | 15 | 46 | 17
  CPK, Day 0, Normal | 43 | 13 | 42 | 16
  CPK, Day 0, Above: number analyzed (Participants) | 44 | 15 | 46 | 17
  CPK, Day 0, Above | 1 | 2 | 4 | 1
  CPK, Day 21, Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  CPK, Day 21, Below | 0 | 0 | 0 | 0
  CPK, Day 21, Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  CPK, Day 21, Normal | 43 | 11 | 41 | 16
  CPK, Day 21, Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  CPK, Day 21, Above | 2 | 1 | 1 | 2
  CPK, Day 42, Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  CPK, Day 42, Below | 0 | 0 | 0 | 0
  CPK, Day 42, Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  CPK, Day 42, Normal | 44 | 13 | 46 | 17
  CPK, Day 42, Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  CPK, Day 42, Above | 2 | 3 | 0 | 1
  CPK, Month 6, Below: number analyzed (Participants) | 41 | 16 | 44 | 18
  CPK, Month 6, Below | 0 | 0 | 0 | 0
  CPK, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 44 | 18
  CPK, Month 6, Normal | 37 | 15 | 41 | 18
  CPK, Month 6, Above: number analyzed (Participants) | 41 | 16 | 44 | 18
  CPK, Month 6, Above | 4 | 1 | 3 | 0
  CPK, Month 12, Below: number analyzed (Participants) | 42 | 17 | 46 | 17
  CPK, Month 12, Below | 0 | 0 | 0 | 0
  CPK, Month 12, Normal: number analyzed (Participants) | 42 | 17 | 46 | 17
  CPK, Month 12, Normal | 38 | 15 | 42 | 16
  CPK, Month 12, Above: number analyzed (Participants) | 42 | 17 | 46 | 17
  CPK, Month 12, Above | 4 | 2 | 4 | 1
  CPK, Month 24, Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  CPK, Month 24, Below | 0 | 0 | 0 | 0
  CPK, Month 24, Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  CPK, Month 24, Normal | 39 | 15 | 43 | 16
  CPK, Month 24, Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  CPK, Month 24, Above | 2 | 2 | 3 | 2

64. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Creatinine (CREA) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents CREA results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21 and 42 and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 46 | 18
Participants
  CREA, Day 0, Below: number analyzed (Participants) | 44 | 15 | 46 | 17
  CREA, Day 0, Below | 0 | 0 | 0 | 0
  CREA, Day 0, Normal: number analyzed (Participants) | 44 | 15 | 46 | 17
  CREA, Day 0, Normal | 44 | 15 | 46 | 17
  CREA, Day 0, Above: number analyzed (Participants) | 44 | 15 | 46 | 17
  CREA, Day 0, Above | 0 | 0 | 0 | 0
  CREA, Day 21, Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  CREA, Day 21, Below | 0 | 0 | 0 | 0
  CREA, Day 21, Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  CREA, Day 21, Normal | 45 | 12 | 42 | 18
  CREA, Day 21, Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  CREA, Day 21, Above | 0 | 0 | 0 | 0
  CREA, Day 42, Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  CREA, Day 42, Below | 0 | 0 | 0 | 0
  CREA, Day 42, Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  CREA, Day 42, Normal | 46 | 16 | 46 | 18
  CREA, Day 42, Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  CREA, Day 42, Above | 0 | 0 | 0 | 0
  CREA, Month 6, Below: number analyzed (Participants) | 41 | 16 | 44 | 18
  CREA, Month 6, Below | 0 | 0 | 0 | 0
  CREA, Month 6, Normal: number analyzed (Participants) | 41 | 16 | 44 | 18
  CREA, Month 6, Normal | 41 | 16 | 44 | 18
  CREA, Month 6, Above: number analyzed (Participants) | 41 | 16 | 44 | 18
  CREA, Month 6, Above | 0 | 0 | 0 | 0
  CREA, Month 12, Below: number analyzed (Participants) | 42 | 17 | 46 | 17
  CREA, Month 12, Below | 0 | 0 | 0 | 0
  CREA, Month 12, Normal: number analyzed (Participants) | 42 | 17 | 46 | 17
  CREA, Month 12, Normal | 42 | 17 | 46 | 17
  CREA, Month 12, Above: number analyzed (Participants) | 42 | 17 | 46 | 17
  CREA, Month 12, Above | 0 | 0 | 0 | 0
  CREA, Month 24, Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  CREA, Month 24, Below | 0 | 0 | 0 | 0
  CREA, Month 24, Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  CREA, Month 24, Normal | 41 | 17 | 46 | 18
  CREA, Month 24, Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  CREA, Month 24, Above | 0 | 0 | 0 | 0

65. Primary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Regards to Lactate Dehydrogenase (LDH) in Study Phase C
Description: Assessed biochemical parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine (CREA), blood urea nitrogen (BUN), lactate dehydrogenase (LDH), and creatine phosphokinase (CPK). Per parameter , it was assessed whether subjects had laboratory values below normal, normal, or above normal range. This outcome presents LDH results, for subjects participating to Phase C of the study.
Time Frame: At Days 0, 21 and 42 and at Months 6, 12 and 24
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Groups:
- GSK1562902A-C Lot 3 6-9Y Group Subjects Aged 6-9 Years Receive: Subjects aged 6-9 years received 2 doses of GSK1562902A vaccine, lot 3. These subjects were enrolled in the Phase C of this NCT00502593 study (or study 108500). The GSK1562902A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm on Days 0 and 21.
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group Subjects Aged 6-9 Years Receive | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 46 | 17 | 47 | 18
Participants
  LDH, Day 0, Below: number analyzed (Participants) | 44 | 15 | 47 | 17
  LDH, Day 0, Below | 0 | 0 | 0 | 0
  LDH, Day 0, Normal: number analyzed (Participants) | 44 | 15 | 47 | 17
  LDH, Day 0, Normal | 36 | 12 | 44 | 17
  LDH, Day 0, Above: number analyzed (Participants) | 44 | 15 | 47 | 17
  LDH, Day 0, Above | 8 | 3 | 3 | 0
  LDH, Day 21, Below: number analyzed (Participants) | 45 | 12 | 42 | 18
  LDH, Day 21, Below | 0 | 0 | 0 | 0
  LDH, Day 21, Normal: number analyzed (Participants) | 45 | 12 | 42 | 18
  LDH, Day 21, Normal | 38 | 11 | 39 | 17
  LDH, Day 21, Above: number analyzed (Participants) | 45 | 12 | 42 | 18
  LDH, Day 21, Above | 7 | 1 | 3 | 1
  LDH, Day 42, Below: number analyzed (Participants) | 46 | 16 | 46 | 18
  LDH, Day 42, Below | 0 | 0 | 0 | 0
  LDH, Day 42, Normal: number analyzed (Participants) | 46 | 16 | 46 | 18
  LDH, Day 42, Normal | 35 | 8 | 42 | 17
  LDH, Day 42, Above: number analyzed (Participants) | 46 | 16 | 46 | 18
  LDH, Day 42, Above | 11 | 8 | 4 | 1
  LDH, Month 6, Below: number analyzed (Participants) | 40 | 16 | 44 | 18
  LDH, Month 6, Below | 0 | 0 | 0 | 0
  LDH, Month 6, Normal: number analyzed (Participants) | 40 | 16 | 44 | 18
  LDH, Month 6, Normal | 32 | 10 | 40 | 18
  LDH, Month 6, Above: number analyzed (Participants) | 40 | 16 | 44 | 18
  LDH, Month 6, Above | 8 | 6 | 4 | 0
  LDH, Month 12, Below: number analyzed (Participants) | 41 | 17 | 45 | 17
  LDH, Month 12, Below | 0 | 0 | 0 | 0
  LDH, Month 12, Normal: number analyzed (Participants) | 41 | 17 | 45 | 17
  LDH, Month 12, Normal | 30 | 12 | 36 | 15
  LDH, Month 12, Above: number analyzed (Participants) | 41 | 17 | 45 | 17
  LDH, Month 12, Above | 11 | 5 | 9 | 2
  LDH, Month 24, Below: number analyzed (Participants) | 41 | 17 | 46 | 18
  LDH, Month 24, Below | 0 | 0 | 0 | 0
  LDH, Month 24, Normal: number analyzed (Participants) | 41 | 17 | 46 | 18
  LDH, Month 24, Normal | 28 | 14 | 43 | 17
  LDH, Month 24, Above: number analyzed (Participants) | 41 | 17 | 46 | 18
  LDH, Month 24, Above | 13 | 3 | 3 | 1

66. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against 1 Strain of Influenza Disease
Description: Titers of serum neutralizing antibodies are presented as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off value of 1:28. The influenza strain assessed was A/Vietnam/1194/04 (A/VIET).Results presented are for subjects participating in Phase A of the study
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 48 | 15 | 43 | 15
Titer
  A/VIET, Day 0: number analyzed (Participants) | 47 | 14 | 43 | 15
  A/VIET, Day 0 | 31.0 [21.8 to 44.0] | 29.0 [15.2 to 55.2] | 32.2 [23.1 to 44.9] | 18.2 [12.2 to 27.3]
  A/VIET, Day 21: number analyzed (Participants) | 48 | 15 | 43 | 14
  A/VIET, Day 21 | 173.5 [123.3 to 244.0] | 98.2 [52.4 to 184.1] | 177.5 [127.0 to 248.0] | 97.2 [46.3 to 204.0]
  A/VIET, Day 42: number analyzed (Participants) | 47 | 15 | 42 | 15
  A/VIET, Day 42 | 1044.4 [845.4 to 1290.3] | 158.4 [76.5 to 327.8] | 1155.1 [920.9 to 1448.7] | 104.5 [51.2 to 213.3]

67. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against 1 Strain of Influenza Disease
Description: Titers of serum neutralizing antibodies are presented as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off value of 1:28. The influenza strain assessed was A/Vietnam/1194/04 (A/VIET). Results presented are for subjects participating in Phase B of the study.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 42 | 16 | 45 | 17
Titer
  A/VIET, Day 0 | 65.5 [47.3 to 90.7] | 48.8 [29.7 to 80.2] | 46.2 [33.2 to 64.2] | 25.6 [17.3 to 37.8]
  A/VIET, Day 21: number analyzed (Participants) | 39 | 16 | 45 | 17
  A/VIET, Day 21 | 344.7 [260.9 to 455.3] | 124.9 [60.7 to 257.2] | 461.7 [376.2 to 566.5] | 148.3 [81.2 to 271.1]
  A/VIET, Day 42 | 1553.2 [1105.9 to 2181.5] | 86.9 [42.5 to 177.6] | 1519.4 [1229.9 to 1877.0] | 154.6 [97.9 to 244.0]

68. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against 1 Strain of Influenza Disease
Description: Titers of serum neutralizing antibodies are presented as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off value of 1:28. The influenza strain assessed was A/Vietnam/1194/04 (A/VIET). Results presented are for subjects participating in Phase C of the study.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 42 | 15 | 43 | 13
Titer
  A/VIET, Day 0: number analyzed (Participants) | 40 | 15 | 43 | 13
  A/VIET, Day 0 | 37.3 [23.9 to 58.1] | 35.5 [17.3 to 72.8] | 25.6 [18.6 to 35.3] | 27.1 [13.3 to 55.4]
  A/VIET, Day 21: number analyzed (Participants) | 40 | 15 | 29 | 8
  A/VIET, Day 21 | 473.8 [351.2 to 639.3] | 111.3 [52.7 to 234.9] | 313.5 [193.3 to 508.4] | 190.1 [57.6 to 628.2]
  A/VIET, Day 42: number analyzed (Participants) | 42 | 14 | 42 | 13
  A/VIET, Day 42 | 4578.3 [3786.6 to 5535.6] | 102.3 [45.9 to 228.2] | 3032.5 [2431.8 to 3781.6] | 77.6 [31.3 to 192.7]

69. Secondary Outcome: Number of Seroconverted Subjects Against One Strain of Influenza Disease With Respect to Serum Neutralizing Antibodies
Description: A seroconverted subject as regards to serum neutralizing antibodies against influenza disease was a subject with a minimum 4-fold increase in serum neutralizing antibody titer at post-vaccination. The flu strain assessed was A/Vietnam/1194/2004 (A/VIET). This outcome presents results for subjects participating to Phase A of the study.
Time Frame: At Days 21 and 42
Population: The analysis was based on the According to protocol (ATP) cohort for immunogenicity, which included all subjects meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria and no major deviation from protocol, for whom immunogenicity data for at least one antigen were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 46 | 14 | 43 | 15
Participants
  A/VIET, Day 21: number analyzed (Participants) | 46 | 14 | 43 | 14
  A/VIET, Day 21 | 31 | 6 | 28 | 10
  A/VIET, Day 42: number analyzed (Participants) | 45 | 14 | 42 | 15
  A/VIET, Day 42 | 43 | 8 | 42 | 10

70. Secondary Outcome: Number of Seroconverted Subjects Against One Strain of Influenza Disease With Respect to Serum Neutralizing Antibodies
Description: A seroconverted subject as regards to serum neutralizing antibodies against influenza disease was a subject with a minimum 4-fold increase in serum neutralizing antibody titer at post-vaccination. The flu strain assessed was A/Vietnam/1194/2004 (A/VIET). This outcome presents results for subjects participating to Phase B of the study.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group
Number analyzed (Participants) | 42 | 16 | 45 | 17
Participants
  A/VIET, Day 21: number analyzed (Participants) | 39 | 16 | 45 | 17
  A/VIET, Day 21 | 25 | 6 | 35 | 11
  A/VIET, Day 42 | 40 | 2 | 42 | 11

71. Secondary Outcome: Number of Seroconverted Subjects Against One Strain of Influenza Disease With Respect to Serum Neutralizing Antibodies
Description: A seroconverted subject as regards to serum neutralizing antibodies against influenza disease was a subject with a minimum 4-fold increase in serum neutralizing antibody titer at post-vaccination. The flu strain assessed was A/Vietnam/1194/2004 (A/VIET). This outcome presents results for subjects participating to Phase C of the study.
Time Frame: At Days 21 and 42
Population: as for outcome 69
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 38 | 15 | 42 | 13
Participants
  A/VIET, Day 21: number analyzed (Participants) | 36 | 15 | 29 | 8
  A/VIET, Day 21 | 29 | 7 | 23 | 3
  A/VIET, Day 42: number analyzed (Participants) | 38 | 14 | 42 | 13
  A/VIET, Day 42 | 37 | 6 | 42 | 5

72. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against 2 Strains of Influenza Disease
Description: Titers of serum neutralizing antibodies are presented as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off value of 1:28. The 2 influenza strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO) strains. Results presented are for subjects participating in Phase A of the study. Subjects participating to Phases B and C of the study were not analysed at these persistence time points for this outcome.
Time Frame: At Months 6, 12 and 24
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 49 | 14 | 40 | 14
Titer
  A/VIET, Month 6 | 781.2 [641.5 to 951.5] | 208.5 [108.6 to 400.3] | 756.1 [624.5 to 915.5] | 482.3 [313.4 to 742.3]
  A/VIET, Month 12: number analyzed (Participants) | 47 | 14 | 36 | 14
  A/VIET, Month 12 | 238.9 [186.1 to 306.6] | 35.4 [16.7 to 74.9] | 179.4 [126.1 to 255.3] | 27.6 [13.4 to 56.9]
  A/VIET, Month 24: number analyzed (Participants) | 47 | 13 | 38 | 11
  A/VIET, Month 24 | 302.5 [231.0 to 396.0] | 39.4 [16.3 to 95.5] | 234.5 [177.1 to 310.6] | 46.6 [18.4 to 118.3]
  A/INDO, Month 6: number analyzed (Participants) | 43 | 13 | 37 | 11
  A/INDO, Month 6 | 113.8 [87.2 to 148.6] | 17.0 [11.1 to 26.1] | 106.8 [82.6 to 138.0] | 16.9 [11.1 to 25.8]
  A/INDO, Month 12: number analyzed (Participants) | 47 | 14 | 36 | 14
  A/INDO, Month 12 | 170.8 [132.7 to 220.0] | 18.2 [11.4 to 29.1] | 139.7 [105.8 to 184.6] | 21.9 [12.2 to 39.2]
  A/INDO, Month 24: number analyzed (Participants) | 47 | 13 | 38 | 11
  A/INDO, Month 24 | 188.5 [144.6 to 245.7] | 31.8 [14.6 to 69.3] | 146.0 [111.7 to 190.8] | 20.5 [11.6 to 36.3]

73. Secondary Outcome: Number of Seroconverted Subjects Against 2 Strains of Influenza Disease as Regards to Neutralizing Antibody Response
Description: A seroconverted subject as regards to neutralizing antibody response was a subject with a minimum 4-fold increase in neutralizing antibody titer at post-vaccination. The 2 influenza strains assessed were A/Vietnam/1194/04 (A/VIET) and A/Indonesia/05/2005 (A/INDO) strains. Results presented are for subjects participating in Phase A of the study. Subjects participating to Phases B and C of the study were not analysed at these persistence time points for this outcome.
Time Frame: At Months 6, 12 and 24.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group
Number analyzed (Participants) | 47 | 13 | 40 | 14
Participants
  A/VIET, Month 6 | 41 | 9 | 38 | 13
  A/VIET, Month 12: number analyzed (Participants) | 45 | 13 | 34 | 14
  A/VIET, Month 12 | 37 | 3 | 23 | 3
  A/VIET, Month 24: number analyzed (Participants) | 45 | 12 | 36 | 14
  A/VIET, Month 24 | 36 | 3 | 23 | 4
  A/INDO, Month 6: number analyzed (Participants) | 39 | 12 | 35 | 11
  A/INDO, Month 6 | 34 | 0 | 31 | 1
  A/INDO, Month 12: number analyzed (Participants) | 43 | 13 | 34 | 14
  A/INDO, Month 12 | 37 | 1 | 31 | 2
  A/INDO, Month 24: number analyzed (Participants) | 43 | 12 | 36 | 11
  A/INDO, Month 24 | 40 | 3 | 33 | 2

74. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: AESIs are adverse events such as clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. AESIs assessed included neuroinflammatory disorders such as cranial nerve disorders, multiple sclerosis,transverse myelitis, Guillain-Barré syndromeor neuritis), musculoskeletal disorders (such as systemic lupus erythematosus, cutaneous lupus, polymyositis, rheumatoid arthritis, reactive arthritis, psoriatic arthropathy, or undifferentiated spondyloarthropathy), gastrointestinal disorders (such as Crohn's disease, ulcerative colitis, ulcerative proctitis, celiac disease), metabolic diseases (such as autoimmune thyroiditis, Addison's disease). skin disorders (such as psoriasis, vitiligo, Raynaud's phenomenon, or autoimmune bullous skin diseases), and other conditions as autoimmune hemolytic anemia, thrombocytopenias, antiphospholipid syndrome, vasculitis, autoimmune hepatitis, or sarcoidosis.
Time Frame: Throughout the entire study period, from Day 0 to Month 24
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A-A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Number analyzed (Participants) | 51 | 18 | 51 | 18 | 51 | 17 | 49 | 17 | 49 | 17 | 49 | 18
Participants | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): from Day 0 to Month 24. Unsolicited adverse events (AEs): during the 21-days period post Dose 1 on Day 0 or the 30-days period post Dose 2 on Day 42. Solicited local and general symptoms: within 7 days post any vaccination.
Arm/Group | GSK1562902A -A Lot 1 3-5Y Group | Fluarix-A 3-5Y Group | GSK1562902A-A Lot 1 6-9Y Group | Fluarix-A 6-9Y Group | GSK1562902A-B Lot 2 3-5Y Group | Fluarix-B 3-5Y Group | GSK1562902A-B Lot 2 6-9Y Group | Fluarix-B 6-9Y Group | GSK1562902A-C Lot 3 3-5Y Group | Fluarix-C 3-5Y Group | GSK1562902A-C Lot 3 6-9Y Group | Fluarix-C 6-9Y Group
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/18 | 0/51 | 0/18 | 1/51 | 1/17 | 0/49 | 0/17 | 2/49 | 0/17 | 1/49 | 0/18
Other Adverse Events (participants affected / at risk) | 42/51 | 17/18 | 48/51 | 14/18 | 42/51 | 11/17 | 41/49 | 13/17 | 43/49 | 13/17 | 46/49 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A -A Lot 1 3-5Y Group (N=51) | Fluarix-A 3-5Y Group (N=18) | GSK1562902A-A Lot 1 6-9Y Group (N=51) | Fluarix-A 6-9Y Group (N=18) | GSK1562902A-B Lot 2 3-5Y Group (N=51) | Fluarix-B 3-5Y Group (N=17) | GSK1562902A-B Lot 2 6-9Y Group (N=49) | Fluarix-B 6-9Y Group (N=17) | GSK1562902A-C Lot 3 3-5Y Group (N=49) | Fluarix-C 3-5Y Group (N=17) | GSK1562902A-C Lot 3 6-9Y Group (N=49) | Fluarix-C 6-9Y Group (N=18)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — This SAE was assessed as causally related to study vaccination
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — This SAE was assessed as causally related to study vaccination
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A -A Lot 1 3-5Y Group (N=51) | Fluarix-A 3-5Y Group (N=18) | GSK1562902A-A Lot 1 6-9Y Group (N=51) | Fluarix-A 6-9Y Group (N=18) | GSK1562902A-B Lot 2 3-5Y Group (N=51) | Fluarix-B 3-5Y Group (N=17) | GSK1562902A-B Lot 2 6-9Y Group (N=49) | Fluarix-B 6-9Y Group (N=17) | GSK1562902A-C Lot 3 3-5Y Group (N=49) | Fluarix-C 3-5Y Group (N=17) | GSK1562902A-C Lot 3 6-9Y Group (N=49) | Fluarix-C 6-9Y Group (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 0 | 0 | 2 | 6 | 2 | 3 | 0 | 3 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 3 | 2 | 1 | 4 | 1 | 3 | 0 | 10 | 2 | 6 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 1
Impetigo (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myringitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpangina (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 3 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 4 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (General disorders) | 9 | 3 | 3 | 2 | 4 | 0 | 4 | 1 | 4 | 0 | 0 | 2
Induration (General disorders) | 7 | 1 | 12 | 6 | 4 | 1 | 6 | 1 | 14 | 0 | 10 | 1
Pain (General disorders) | 31 | 7 | 44 | 12 | 27 | 3 | 36 | 9 | 37 | 7 | 44 | 15
Redness (General disorders) | 10 | 2 | 12 | 5 | 6 | 4 | 6 | 3 | 16 | 2 | 6 | 1
Swelling (General disorders) | 10 | 1 | 14 | 7 | 9 | 2 | 10 | 2 | 18 | 2 | 14 | 3
Drowsiness (General disorders) | 7 | 1 | 0 | 0 | 9 | 1 | 0 | 0 | 12 | 1 | 0 | 0 — Symptom assessed in subjects aged 3-5 years.
Fever (axillary temperature >=37.5°C) (General disorders) | 8 | 0 | 0 | 0 | 10 | 2 | 0 | 0 | 18 | 0 | 0 | 0 — Symptom assessed in subjects aged 3-5 years.
Irritability (General disorders) | 9 | 1 | 0 | 0 | 13 | 2 | 0 | 0 | 18 | 0 | 0 | 0 — Symptom assessed in subjects aged 3-5 years.
Loss of appetite (General disorders) | 12 | 1 | 0 | 0 | 8 | 1 | 0 | 0 | 15 | 1 | 0 | 0 — Symptom assessed in subjects aged 3-5 years.
Shivering (General disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 10 | 1 | 0 | 0 — Symptom assessed in subjects aged 3-5 years.
Sweating (General disorders) | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 — Symptom assessed in subjects aged 3-5 years
Vomiting (General disorders) | 7 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 6 | 1 | 0 | 0 — Symptom assessed in subjects aged 3-5 years
Arthralgia (General disorders) | 0 | 0 | 6 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 9 | 2 — Symptom assessed in subjects aged 6-9 years.
Fatigue (General disorders) | 0 | 0 | 7 | 1 | 0 | 0 | 6 | 1 | 0 | 0 | 11 | 2 — Symptom assessed in subjects aged 6-9 years.
Fever (axillary temperature >= 37.5°C) (General disorders) | 0 | 0 | 7 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 18 | 0 — Symptom assessed in subjects aged 6-9 years.
Gastrointestinal symptoms (General disorders) | 0 | 0 | 9 | 5 | 0 | 0 | 4 | 5 | 0 | 0 | 16 | 5 — Symptom assessed in subjects aged 6-9 years.
Headache (General disorders) | 0 | 0 | 20 | 5 | 0 | 0 | 11 | 2 | 0 | 0 | 25 | 3 — Symptom assessed in subjects aged 6-9 years.
Myalgia (General disorders) | 0 | 0 | 10 | 3 | 0 | 0 | 11 | 2 | 0 | 0 | 13 | 2 — Symptom assessed in subjects aged 6-9 years
Shivering (General disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 7 | 0 | 0 | 0 | 13 | 3 — Symptom assessed in subjects aged 6-9 years.
Sweating (General disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 3 | 2 | 0 | 0 | 6 | 1 — Symptom assessed in subjects aged 6-9 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.